# Emulation of the effects of oral semaglutide on cardiovascular outcomes in individuals with type 2 diabetes and established atherosclerotic cardiovascular disease and/or chronic kidney disease: SOUL trial

NCT06659718

23<sup>rd</sup> April 2025

# 1. Title Page

| Title | Emulation of the effects of oral semaglutide on cardiovascular outcomes in individuals with type 2 diabetes and established atherosclerotic cardiovascular disease and/or chronic kidney disease: SOUL trial (NCT03914326) |
|---|---|
| Research question & Objectives | The SOUL trial aims to evaluate the effect of oral semaglutide versus placebo on MACE outcomes (CV death, nonfatal MI or nonfatal stroke) among individuals with type 2 diabetes and established atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD). |
| Protocol version | Version 5 |
| Last update date | 23st April 2025 |
| Contributors | Primary investigator contact information: Dr. Shirley Wang Swang1@bwh.harvard.edu Contributor names: Shirley Wang, Sushama Kattinakere Sreedhara, Elyse DiCesare Sushama implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform. |
| Study registration | Site: <text> Identifier: <text></text></text> |
| Sponsor | Organization: Food and Drug Administration Contact: Dianne Paraoan dianne.paraoan@fda.hhs.gov |
| Conflict of interest | Dr. Wang has consulted for Veracity Healthcare Analytics, Exponent Inc, and MITRE and FFRDC for Centers for Medicare and Medicaid for unrelated work. |

# Table of contents

| 1. Title Page | |
|---|---|
| 2. Abstract | |
| 3. Amendments and updates | |
| 4. Rationale and background | 5 |
| 5. Research question and objectives | |
| Table 1 Primary and secondary research questions and objective | |
| 6. Research methods | |
| 6.1. Study design | |
| 6.2. Study design diagram | |
| 6.3. Setting | |
| 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population | |
| 6.3.2 Context and rationale for study inclusion criteria: | |
| 6.3.3 Context and rationale for study exclusion criteria | 9 |
| 6.4. Variables | |
| 6.4.1 Context and rationale for exposure(s) of interest | |
| 6.4.2 Context and rationale for outcome(s) of interest | |
| 6.4.3 Context and rationale for follow up | |
| Table 2. Operational Definitions of Follow Up | |
| 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications). | |
| 6.5. Data analysis | |
| 6.5.1 Context and rationale for analysis plan | |
| Table 4. Primary, secondary, and subgroup analysis specification | |
| Table 5. Sensitivity analyses – rationale, strengths and limitations | |
| 6.6.1 Context and rationale for data sources | |
| Table 6. Metadata about data sources and software | |
| 6.7. Data management | |
| 6.8. Quality control | |
| 6.9. Study size and feasibility | |
| 7. Limitation of the methods | |
| 8. Protection of human subjects | |
| 9. References | |
| 10. Appendices | |
| 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment | |
| 2 Code algorithms | |
| 3 Flowchart for cohort assembly | |
| 4 1st feasibility assessment | |
| 5 2nd feasibility assessment | |
| 6 Balance Assessment - PS Distribution and C-Statistic | |
| 7 Balance Assessment - Table 1 | |
| 8 Covariate – Algorithm | |

#### 2. Abstract

This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the SOUL trial described below. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The SOUL trial, which is a superiority trial to evaluate the effect of oral semaglutide versus placebo on MACE outcomes (CV death, nonfatal MI, or nonfatal stroke) among individuals with type 2 diabetes (T2DM) and established atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD).

The database study designed to emulate SOUL will be a new-user active comparative study, where we compare the effect of oral semaglutide versus sitagliptin on MACE outcome among patients with T2DM and with established ASCVD and/or CKD. Sitagliptin was selected to act as an active-comparator proxy for placebo. Sitagliptin and the class of dipeptidyl peptidase-4 (DPP-4) inhibitors have been demonstrated not to have an effect on MACE in a series of RCTs, and they are used in similar stages of disease/line of therapy as semaglutide, as well as being similarly costly.

The study will use three data sources: Optum Clinformatics, Merative Marketscan, and Medicare.

Optum: Study period between 20<sup>th</sup> Sept 2019 – 29<sup>th</sup> February 2024 Marketscan: Study period between 20<sup>th</sup> Sept 2019 - 31<sup>st</sup> Dec 2022 Medicare: Study period between 20<sup>th</sup> Sept 2019 – 31<sup>st</sup> Dec 2020

# 3. Amendments and updates

| Version date | Version number | Section of protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 19 <sup>th</sup> Aug 2024 | 2 | 6.4, 6.5, Table 2-4, appendices 5-8 | Inclusion Exclusion Criteria: Adding TIRZEPATIDE to the list of other GLP1, Stroke definition to include only Ischemic stroke Outcome: Stroke definition to include only Ischemic stroke | Better algorithms for exclusion criteria and outcome |

| | | | Added covariates for PS adjustment | To operationally define covariates and adjust for confounding |
|---|---|---|---|---|
| | | | Power and feasibility (balance checks) post PS matching added in appendices 5, 6 and Table 1 | Pre-planned data check |
| | | | Changed primary analysis from PS fine-stratification weights to 1:1 PS matching | The power calculation indicates that there will be sufficient power with 1:1 matching |
| | | | Added planned sensitivity analyses | To pre-specify sensitivity analyses |
| 7 <sup>th</sup> December<br>2024 | 3 | 6.4.3 | Added Nursing home admission as one of the censoring reason. | This censoring reason was left out of the protocol in error, and we are amending it to be consistent with our other protocols |
| 16 <sup>th</sup> December<br>2024 | 3.1 | Appendices | Added the FDA protocol review dates for the first and second feasibility | The protocol review dates by the FDA were not documented in the previous version. |
| 10 <sup>th</sup> March<br>2025 | 4 | Appendices | Covariate code algorithms for Pap smear, COPD, pneumonia, and diabetic nephropathy were corrected. | Errors in the implementation of covariate code algorithms for Pap smear, COPD, pneumonia, and diabetic nephropathy were identified. |
| 17 <sup>th</sup> April 2025 | 5 | Negative control outcomes | Added Hernia and Lumbar radiculopathy | Given the ongoing discussion around semaglutide and its potential association with non-arteritic anterior ischemic optic neuropathy (NAION) as a negative control outcome, we |

| wanted to include alternative |
|-------------------------------|
| negative control outcomes. |

# 4. Rationale and background

The purpose of this protocol is to specify the emulation of the SOUL trial (NCT03914326). Oral semaglutide became available on September 20<sup>th,</sup> 2019.¹ The trial enrolled 9,650 participants between June 17, 2019 – March 24, 2021. The trial design is event-driven with an expected 3.5 to 5 years follow-up period and an assumed outcome rate of 3.5% in the placebo arm. The trial uses 90% power with a 0.025 type 1 error rate to confirm superiority.².³

# 5. Research question and objectives

## Table 1 Primary and secondary research questions and objective

## A. Primary research question and objective

| Objective: | To evaluate the comparative safety effect of oral semaglutide versus sitagliptin (proxy for placebo) on MACE outcomes (CV death, nonfatal MI, or nonfatal stroke) in patients with diabetes and established CV or kidney disease |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will be superior to sitagliptin at preventing MACE |
| Population (mention key inclusion-exclusion criteria): | The study population included patients aged 50 years or older with type 2 diabetes (T2DM) and established atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD). |
| | Patients were excluded if they had recent MI, stroke, hospitalization for unstable angina or transient ischemic attack, class IV heart failure, prior treatment with GLP-1, history of multiple endocrine neoplasia type 2, medullary thyroid cancer, pancreatitis, bariatric surgery, current or recent pregnancy, history of non-melanoma skin cancer, dialysis of sever renal impairment, proliferative retinopathy or maculopathy requiring treatment, history of diabetic ketoacidosis. |
| Exposure: | Oral semaglutide |
| Comparator: | Sitagliptin |
| Outcome: | Major adverse cardiac event (MACE), including myocardial infarction, stroke, and all cause death |

| Time (when follow up begins and ends): | 1 days after cohort entry date until the first of outcome, disenrollment, end of study period, 365 days after cohort entry date, discontinuation (30 days grace and risk window), switch between the arms, start of any other GLP1 agonists (including injectable semaglutide) |
|---|---|
| Setting: | Patients may be treated in outpatient settings. The outcome will be measured from inpatient hospitalizations and/or death. |
| Main measure of effect: | Hazard ratio |

# B. Secondary research question 1 and objective

| Objective: | To evaluate the effect of oral semaglutide versus sitagliptin on negative control outcomes, including A. cataract surgery, B. hernia and C. lumbar radiculopathy |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will not have a different effect from sitagliptin. |
| Population (mention key inclusion-exclusion criteria): | The study population included patients aged 50 years or older with type 2 diabetes (T2DM) and established atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD). |
| | Patients were excluded if they had recent MI, stroke, hospitalization for unstable angina or transient ischemic attack, class IV heart failure, prior treatment with GLP-1, history of multiple endocrine neoplasia type 2, medullary thyroid cancer, pancreatitis, bariatric surgery, current or recent pregnancy, history of non-melanoma skin cancer, dialysis of sever renal impairment, proliferative retinopathy or maculopathy requiring treatment, history of diabetic ketoacidosis. In addition, patients were excluded for baseline hernia or lumbar radiculopathy when the negative outcome was hernia or lumbar radiculopathy respectively. |
| Exposure: | Oral semaglutide |
| Comparator: | Sitagliptin |
| Outcome: | Separate analyses were run for cataract surgery, hernia, and lumbar radiculopathy |
| Time (when follow up begins and ends): | 1 days after cohort entry date until the first of outcome, disenrollment, end of study period, death, 365 days after cohort entry date, discontinuation (30 days grace and risk window), switch between the arms, start of any other GLP1 agonists (including injectable semaglutide) |

| Setting: | Patients may be treated in outpatient settings. The outcome will be measured using procedure codes in an outpatient setting. |
|---|---|
| Main measure of effect: | Hazard ratio |

#### 6. Research methods

# 6.1. Study design

Research design (e.g. cohort, case-control, etc.): New user active comparator cohort study

Rationale for study design choice: The new user active comparator design is a powerful design that may be able to address confounding by indication. It accomplishes this, in large part, through judicious selection of an appropriate active-comparator group.<sup>4,5</sup> While selection of an appropriate comparator in the design phase is crucial, cohort studies often require additional adjustment of measurable confounders. A common method for adjusting for confounding is via a propensity score (PS).

#### 6.2. Study design diagram



Note: The CV disease inclusion may include acute MI codes but any acute MI in the 60 days is excluded. History of heart failure is an inclusion criterion, but heart failure class IV is excluded.

#### 6.3. Setting

#### 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population

Time 0 in the database study was defined to emulate randomization to oral semaglutide versus sitagliptin in the clinical trial design. See appendix tables 1 and 2a for operational definitions and detailed code algorithms.

#### 6.3.2 Context and rationale for study inclusion criteria:

Study inclusion criteria were defined to emulate the inclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. See appendix tables 1 and 2b for operational definitions and detailed code algorithms.

A flowchart of the study cohort assembly is provided in Appendix 3.

#### 6.3.3 Context and rationale for study exclusion criteria

Study exclusion criteria were defined to emulate the exclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. See appendix tables 1 and 2c for operational definitions and detailed code algorithms.

A flowchart of the study cohort assembly is provided in Appendix 3.

#### 6.4. Variables

#### 6.4.1 Context and rationale for exposure(s) of interest

The exposure and comparator were defined to emulate the agents compared for the trial, oral semaglutide versus sitagliptin. See appendix tables 1 and 2a for operational definitions and detailed code algorithms.

#### Algorithm to define duration of exposure effect:

Assuming the effect of the drug lasts for 30 days after the days' supply, we allow 30 days gap between the dispensation (grace period) and also add 30 days at the end of days' supply of dispensation (exposure risk window).

# 6.4.2 Context and rationale for outcome(s) of interest

The primary outcome for the database study was defined to emulate the primary outcome for the trial of MACE. In the trial, this was a combination of myocardial infarction, stroke, and cardiovascular death. In our emulation, due to inability to capture cause of death, our modified MACE outcome was measured as inpatient myocardial infarction, inpatient stroke, and all-cause mortality. See appendix tables 1 and 2d for operational definitions and detailed code algorithms. Optum includes death information from the inpatient discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. MarketScan includes information from the inpatient discharged dead

status, NDI cause of death, and social security death master file. The positive predictive value for the myocardial infarction outcome algorithm using ICD-9 codes was observed to be 88.4% and 94% in validation studies.<sup>6,7</sup> The PPV for the ischemic stroke outcome algorithm was 88% and 95% in validation studies using ICD9 codes.<sup>6,8</sup> The ICD9 code algorithms were mapped to ICD10 codes and reviewed by a clinician, but the performance of the mapped codes was not further validated.

Secondary outcomes from the trial that will be evaluated include components of the MACE outcome including:

- 1. Myocardial infarction
- 2. Stroke
- 3. All cause Death

Control outcomes of interest include:

- 1. Cataract surgery. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.
- 2. Hernia. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.
- 3. Lumbar radiculopathy. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.

#### 6.4.3 Context and rationale for follow up

Both on-treatment (OT) and intention-to-treat (ITT) analyses will be conducted. Adherence in clinical practice databases is expected to be much worse than in the trial, Therefore the OT analysis will be the primary analysis. The OT analysis targets the relative hazard of outcomes while on treatment and may more closely emulate the effect observed in highly adherent trial participants.

Table 2. Operational Definitions of Follow Up

| Follow up start | Day 1 | |
|---|---|---|
| Follow up end <sup>1</sup> | Select all that apply | Specify |
| Date of outcome | Yes | |
| Date of death | Yes | Part of the outcome |
| End of observation in data | Yes | Date of disenrollment |
| Day X following index date (specify day) | Yes | Day 365 |

| End of study period (specify date) | Yes |
|---|---|
| End of exposure (specify operational details, e.g. stockpiling algorithm, grace period) | Yes |
| Date of add to/switch from exposure (specify algorithm) | Yes |
| Other date (specify) | Yes |

| Different dates for each database (Optum: 29th Feb 2024, Marketscan Dec 31st 2022, Medicare Dec 31st 2020) |
|---|
| 30 days grace window and 30 days risk window |
| Date of augmentation or switching from an exposure to a |
| comparator and vice versa. |
| Nursing home admission, Censor upon starting any other |
| GLP1 agonists including injectable semaglutide. |

# 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications)

We identified a series of covariates that were likely confounders due to being strong risk factors for the primary outcome that were associated with choice of treatment. These include demographics, disease severity related variables, comorbid conditions, comedications, frailty, healthcare utilization and markers of health seeking behaviour.

Table 3. Operational Definitions of Covariates

| Characteristic | Conceptual<br>definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Age | Cohort entry year – year of birth, (last observed value in the baseline) | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Gender | Male, Female<br>(last observed value in<br>the baseline) | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Region | Northeast, Midwest/North central, South, West (last observed value in the baseline) | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Year of Cohort<br>Entry | 2019 (Sept-Dec),<br>2020 (Jan-March),<br>2020 (April-June),<br>2020 (July-Sept),<br>2020 (Oct-Dec), 2021<br>(Jan-Dec), 2022 (Jan-<br>Dec), 2023 (Jan-Dec),<br>2024 (Jan - Feb) | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |


| Characteristic | Conceptual definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Insulins | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Meglitinides | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| SU-2nd gen | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Metformin | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Thiazolidinedion es | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| SGLT-2i | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Alpha-<br>glucosidase<br>inhibitors | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| ACEs/ARBs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Thiazides | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Beta-blockers | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide | n/a | Investigator review of codes, |

| Characteristic | Conceptual<br>definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | sources in<br>Appendix 8 |
| Calcium<br>channel<br>blockers | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Loop diuretics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Other diuretics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Nitrates | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Hear failure<br>medications<br>(Digoxin +<br>Entresto +<br>Ivabradine) | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anti-arrhythmics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| COPD/asthma medications | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Statins | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Other lipid-<br>lowering drugs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Antiplatelet agents | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Oral<br>anticoagulants | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| NSAIDs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Oral corticosteroids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Bisphosphonate<br>s | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Opioids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anti-<br>depressants | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Gabapentinoids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Benzodiazepine<br>s | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anxiolytics/hypn otics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide | n/a | Investigator review of codes, |

| Characteristic | Conceptual<br>definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | sources in<br>Appendix 8 |
| Medications for dementia | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Combined comorbidity score | Comorbidity score ranging from -2 to 26 | Continuous | [-180, 0] | Any | ICD10-CM | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Gagne, Joshua J<br>et al. <sup>9,10</sup> |
| Frailty score | | Continuous | [-180, 0] | Any | ICD10-CM | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Kim et al. <sup>11</sup> |
| Unique generic medicines | | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Unique brand medicines | | Continuous | [-180, 0] | n/a | ICD10-CM | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Hospitalizations<br>[-90, 0] | | Binary | [-90, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | |
| Hospitalizations<br>[-180, 0] | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | |
| ED visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Office visits | | Continuous | [-180, 0] | OP | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Endocrinologist visit | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide | n/a | Investigator review of codes, |

| Characteristic | Conceptual<br>definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | sources in<br>Appendix 8 |
| Cardiologist visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Internal medicine/family medicine visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Electrocardiogra<br>ms | | Binary | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Echocardiogram<br>s | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| HbA1c tests received | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Glucose tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Lipid tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Creatinine tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Bone mineral density test | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual<br>definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Basic or<br>comprehensive<br>metabolic blood<br>chem test | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Mammogram | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Pap smear | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| PSA | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Flexible<br>Sigmoidoscopy<br>or colonoscopy<br>or CT virtual<br>colonoscopy | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Flu vaccine/<br>Pneumococcal<br>vaccine | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Telemedicine | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

 $<sup>^{1}</sup>$  IP = inpatient, OP = outpatient, ED = emergency department, OT = other,  $^{n}$ /a = not applicable  $^{2}$  See appendix for listing of clinical codes for each study parameter

<sup>&</sup>lt;sup>3</sup> Specify whether a diagnosis code is required to be in the primary position (main reason for encounter)

## 6.5. Data analysis

#### 6.5.1 Context and rationale for analysis plan

The study will use a propensity score (PS) 1:1 nearest neighbor matching with a caliper of 0.01 on the propensity score scale. The PS will be estimated as the probability of initiating oral semaglutide versus sitagliptin given the baseline patient characteristics using multivariable logistic regression models. As diagnostics for PS models, the study will evaluate covariate balance using standardized differences and c-statistics post-matching. The study will estimate the hazard ratio for oral semaglutide versus sitagliptin on MACE outcome in the matched population using a Cox proportional hazards model.

Table 4. Primary, secondary, and subgroup analysis specification

#### A. Primary analysis

| Hypothesis: | Oral semaglutide might decrease risk of MACE outcome compared to sitagliptin in those with diabetes and established CV |
|---|---|
| | disease |
| Exposure contrast: | Oral semaglutide vs sitagliptin |
| Outcome: | MACE |
| Analytic software: | Aetion, STATA 17, SAS 9.4, R.4.4.0 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | n/a |

# B. Secondary Analysis 1

| Hypothesis: | Oral semaglutide has no effect on risk of negative control outcomes compared to sitagliptin. Negative control outcomes |
|---|---|
| | include: A. cataract surgery, B. hernia, C. lumbar radiculopathy |
| Exposure contrast: | Oral semaglutide vs sitagliptin |
| Outcome: | Separate analyses were run for each negative control outcome, including cataract surgery, hernia and lumbar |
| | radiculopathy |

| Analytic software: | Aetion, STATA 17, SAS 9.4, R.4.4.0 |
|---|---|
| Model(s): | |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | n/a |

Table 5. Sensitivity analyses – rationale, strengths and limitations

| | What is being varied? How? | Why?<br>(What do you expect to<br>learn?) | Strengths of the sensitivity analysis compared to the primary | Limitations of the sensitivity analysis compared to the primary |
|---|---|---|---|---|
| Re-weighted population distribution | We will re-weight the population distribution of the pooled database study cohorts to reflect that of the RCT if that information is made public prior to publication of our results. | We will learn about potential effect modification due to different distributions of key characteristics such as age/sex in the RCT versus the database study. | The population distributions will be more aligned. | The measurement of these population characteristics may be measured differently in the RCT vs database study, with different levels of specificity and sensitivity. |
| Negative control<br>outcomes, including<br>cataract surgery,<br>hernia, lumbar<br>radiculopathy | We evaluate negative control outcomes of cataract surgery, hernia, and lumbar radiculopathy, where no causal effect is expected from semaglutide or sitagliptin | We will evaluate the potential impact of residual confounding on this outcome for which there is not expected to be a causal effect | The evaluates the robustness of<br>the interpretation of the primary<br>analysis by evaluating the<br>potential magnitude of<br>unmeasured confounding | This analysis assumes that the confounding structure is the same or similar for the negative control outcome as the outcome of interest |
| PS-adjustment<br>method | Instead of 1:1 PS matching, we will use PS fine stratification weights. The analytic cohort will be asymmetrically trimmed at 1% | Use of fine-stratification weights will have more power than 1:1 matching | More power to estimate ATT | More complex to understand than simple 1:1 match, potentially less closely balanced |

of the tails. The analytic cohort will be weighted to estimate the average effect in the treated (ATT).

Each exposed patient will be assigned a weight = 1.

Each comparator patient will be assigned a weight =

 $\frac{\binom{N exposed in strata i}{N_{total exposed}}}{\binom{N unexposed in strata i}{N_{total unexposed}}}$ 

Apply benchmark, expand, calibrate (BenchExCal) sensitivity and tipping point analysis We will use the observed difference in result from emulation of SUSTAIN6 to recalibrate the result from the database study emulation of PIONEER6. We will conduct a tipping point analysis with a range of plausible estimates of the expected difference.

We expect to learn about the performance of BenchExCal in an example where we emulate an RCT for an expanded indication and an RCT result for the expanded indication is available.

The analysis will calibrate the primary result based on expected differences due to bias and/or design emulation differences and propagate uncertainty regarding the impact of these factors into the frequentist primary result

The ability to appropriately calibrate the result depends on how "close" the clinical context is between the initial and expanded indication. The approach assumes that the net effect of bias and design emulation differences is the similar.

#### 6.6. Data sources

#### 6.6.1 Context and rationale for data sources

**Reason for selection:** The study will be conducted in 3 US health care claims databases: Optum Clinformatics (2019-Feb 2024), Merative Marketscan (2019-2022) and Medicare (a sample that includes all patients with diabetes or heart failure diagnosis, 2019-2020).

Strengths of data source(s): Each data source contains deidentified, longitudinal, date-stamped information on patient enrollment, demographics, inpatient/outpatient diagnosis and procedures, admission and discharge dates, and medication dispensation. The death data is captured in the Optum database from inpatient discharge status, social security death master file, and deaths scraped from obituaries or other sources. The death data in MarketScan is captured from the social security death master file and inpatient discharge status. It is recognized that the social security death master file has high specificity and positive predictive value for deaths. While this data resource has under captured deaths since 2011, the capture of deaths is not expected to be differential between compared exposure groups. The death data is captured in the Medicare database from inpatient discharge status, and social security death master file.

Limitations of data source(s): Patient healthcare encounters are only observable when they are enrolled in an insurance plan that contributes to the database. Patients may change insurance plans for multiple reasons. Both Optum Clinformatics and Merative MarketScan are primarily employer based insurance databases where patients may disenroll with job changes. Patients in Medicare may move in and out of fee-for-service plans. We are excluding person-time in health maintenance organization (HMO) plans due to concerns about the completeness of capture of diagnoses and procedures. This means that we require

patients to be enrolled in Medicare parts AB and D during the baseline assessment window and censor patients if they switch to part C. In claims data, dispensing data for inpatient medication is unavailable. Diagnoses reflect billing practices, therefore algorithms (preferably validated) are needed for accurate phenotyping of patient conditions. Services that are not covered by insurance do not appear in the data. The trial evaluated cardiovascular deaths, however we will evaluate all cause death in the emulation because most deaths in this cohort of patients at high cardiovascular risk will be related to cardiovascular reasons, the cause of death is not recorded for databases not linked to NDI, and the performance of NDI at identifying cardiovascular causes of death may be suboptimal.<sup>15</sup>

#### Data source provenance/curation:

Information about Optum Clinformatics and Merative MarketScan can be found in data dictionaries and user guides that are provided to clients. Information about Medicare data provenance and curation can be found on the ResDac website. 16

Table 6. Metadata about data sources and software

| | Data 1 | Data 2 | Data 3 |
|---|---|---|---|
| Data Source(s): | Optum Clinformatics | Merative Marketscan | Medicare |
| Study Period: | 20th Sept 2019-29th Feb 2024 | 20th Sept 2019-31st Dec 2022 | 20th Sept 2019-31st Dec 2020 |
| Eligible Cohort Entry Period: | 20th Sept 2019-29th Feb 2024 | 20th Sept 2019-31st Dec 2022 | 20th Sept 2019-31st Dec 2020 |
| Data Version (or date of last update): | April 2024 | Mortality Cut Set A<br>Received 2024-03-01 | DUA 59286_Received 2023-10-<br>17 |
| Data sampling/extraction criteria: | n/a | n/a | Patients with a diabetes or heart failure diagnosis |
| Type(s) of data: | Administrative healthcare claims | Administrative healthcare claims | Administrative healthcare claims |
| Data linkage: | n/a | n/a | Linkage to National Death Index |
| Conversion to CDM*: | n/a | n/a | n/a |
| Software for data management: | Aetion Evidence Platform® (2024) | Aetion Evidence Platform® (2024) | Aetion Evidence Platform® (2024) |

\*CDM = Common Data Model

# 6.7. Data management

<u>Tracking data:</u> The Data Use Agreement (DUA) Custodian (Principal Investigator) and the Division Operations Manager (Winta Tekle) are responsible for receiving and creating a record of new data associated with the given request. The Operations Manager is responsible for all indexing and archiving of documents and

electronic media related to data that the Division receives and will log data location, data contents, and associated DUA and Institutional Review Board (IRB) numbers in the Division's centralized tracking system.

<u>Handling and storage:</u> In-scope data will be stored utilizing Mass General Brigham approved information systems – i.e., Division servers and Mass General Brigham network storage.

<u>Archiving</u>: Data retention and any removal will be executed by the Division Operations Manager (Winta Tekle) and Data Manager (Todd MacGarvey). The Division follows Mass General Brigham enterprise record retention policies and follow the terms of the agreement through which the in-scope data was received.

Information security: The Division follows Mass General Brigham's Enterprise Information Security Program (EISP). The EISP helps by providing assurance that Mass General Brigham information and information systems are protected from unauthorized access, use, disclosure, duplication, modification, or destruction in order to maintain their confidentiality, integrity, and availability. To that end, the EISP policies, standards and procedures create an information security framework that is aligned with the recommendations of the International Organization for Standardization's (ISO) publication 27001 and the National Institute of Standards and Technology's (NIST) publication 800-53 Family of Controls and MGB regulatory and legal requirements (as a HIPAA covered entity).

Mass General Brigham workforce members are required to complete new workforce privacy and information security training upon hire and annually thereafter. Refresh training is provided as appropriate. Mass General Brigham workforce members are required to review and sign a Confidentiality Agreement upon hire and annually thereafter. Additionally, we follow Enterprise Information Security and Privacy policies, including Managing Workforce Members Information Security Responsibilities Policy, which was developed to help assure that Mass General Brigham workforce members are competent and eligible to support the information security responsibilities associated with their role. Mass General Brigham workforce, including Division staff, are required to comply with Enterprise Information Security and Privacy Policies.

<u>Facilities:</u> The research team uses a highly secure, state-of-the-art, computing facility housed at Mass General Brigham's Corporate Data Centers in Needham and Marlborough, Massachusetts as well as Amazon Web Services (AWS). We maintain redundant storage for maximal data integrity and high-speed data access.

The Division uses Mass General Brigham corporate provisioned servers to analyze and store data in connection with this project. There are strict access controls enforced by technical means to ensure that only study staff who have been approved to conduct data analyses and contracted data engineers are able to access data (e.g., Mass General Brigham Authentication (Active Directory) utilized; auditing, logging, and monitoring enabled; firewalls enabled; etc.). All Division servers used in this study are accessible to only authorized staff only through the MGB network and utilizing VPN as appropriate (i.e., users must be on the network and logged into VPN to access). Mass General Brigham has a network information security monitoring team and in-scope servers are enrolled in enterprise security tools (e.g., vulnerability scanning service, antivirus, etc.).

The Division also uses AWS. In-scope AWS services / resources have undergone review and assessment by Mass General Brigham's Information Security Risk Assessment Team/ InfoSec Risk Management Team as required and in alignment with NIST 800-30: Guide for Conducting Risk Assessments. In-scope AWS servers are for our exclusive use (reserved instances), are covered under our organization's Business Associate Agreement with AWS. In-scope servers are housed in anonymous facilities that are not branded as AWS facilities. Physical access is strictly controlled both at the perimeter and at building ingress points by professional security staff utilizing video surveillance, intrusion detection systems, and other electronic means.

Security attributes and controls for the Division's use of in-scope AWS in connection with this project include: encryption at rest and in transit (industry standard AES-256 encryption, SSL/TSL), anti-malware, latest OS updates and patches as well as anti-virus; multi-factor authentication (MFA), Identity and Access

Management, including SSO; auditing and logging; principle of least privilege, including for traffic and ports (e.g., deny all default configurations), use of VPC enabled Step functions, etc.; separation between environments; minimum necessary (out of the box AWS roles are not used as they can be overly permissive); all data would reside in the US domestic regions – use only US east HIPAA compliant region; performance monitoring enabled and reviewed as per internal processes; passwords compliant with enterprise password policy and, as appropriate, more protective password requirements; etc. Our Division's AWS use is also subject to ongoing evaluation and monitoring as well – e.g., vulnerability scanning and management, access review, etc.

A data file list will be maintained in Amazon S3 and tracked through Cloudtrail and Cloudwatch. Reporting of data file availability for any file stored in an S3 bucket will be controlled by MGB.

Amazon EC2, Amazon EBS, and Amazon VPC are integrated with AWS CloudTrail, a service that provides a record of actions taken by a user, role, or an AWS service in Amazon EC2, Amazon EBS, and Amazon VPC. CloudTrail captures all API calls for Amazon EC2, Amazon EBS, and Amazon VPC as events, including calls from the console and from code calls to the APIs. MGB IT/security staff have full access to CloudTrail to ensure that CloudTrail monitoring is available at all times. Amazon CloudWatch Events delivers a near-real-time stream of system events that describe changes in AWS resources. Amazon CloudTrail can log, continuously monitor, and retain account activity related to actions across the MGB AWS infrastructure. CloudTrail provides event history of MGB AWS account activity. This event history simplifies security analysis, resource change tracking, and troubleshooting and complies with requirements to ensure the data file inventory is controlled by MGB.

Backups: Backups are created using industry recognized Cryptographic mechanisms (e.g., 256-bit AES encryption) as appropriate and required. Data are backed up within the MGB network from the MGB Needham data center to the MGB Marlborough data center via replication/mirroring and volume-level snapshots.\_AWS Backup supports both instance-level backups as Amazon Machine Images (AMIs) and volume-level backups as separate snapshots based on the resource tags. AMIs allow MGB IT and security staff to create backups of all S3 and EC2 instances. This backup approach allows elimination of EC2 instances when access to CMS data files is no longer needed. Use of temporary instances will allow highest security control to be applied regarding for whom and when CMS data files are accessible.

In addition to the safeguards listed above, the Division follows enterprise privacy and information security policies and maintains internally procedures in connection with this project to safeguard the data in connection with this project as appropriate and required including: Physical Security and Environmental Controls for Electronic Information Policy; IT Access Control Standards for Users policy; Safeguarding Fax Copiers Printers Telephone Use and Pagers; Physical Removal and Transport of Protected Health Information and Personal Information policy, etc.

# 6.8. Quality control

Senior Programmers and Research Specialists perform QA/QC on raw or common data model converted data via SAS/R/Aetion software. The protocol will be iteratively developed and pre-specified data checks including feasibility counts and balance on baseline covariates will be conducted with outputs reviewed by both MGB and FDA team members. Team members will review code lists to ensure fidelity to intended algorithms.

#### 6.9. Study size and feasibility

First feasibility assessment: Details of power calculations after applying eligibility criteria and matching on ages, sex and comorbidity score are available in appendix 4.

Second feasibility assessment: Details of power calculations after matching or weighting on all predefined propensity score variables are available in appendix 5. Propensity score distribution plots with c-statistics are available in appendix 6. Table 1 showing prevalence of baseline characteristics and standardized differences in distribution are available in appendix 7.

#### 7. Limitation of the methods

As we are using secondary data and the data were not collected for research, some important variables may not be collected or will be measured imperfectly. We have selected validated algorithms when possible and we have created proxies for important variables that are not directly captured in the data to reduce confounding by unmeasured factors. One measurement difference is for the primary outcome, where for the RCT, MACE was defined as stroke, myocardial infarction, and cardiovascular death, whereas in our database study, it is defined as stroke, myocardial infarction, and all cause death.

When comparing results from an RCT to a database study that emulates the design, we assume that the findings from the single RCT are internally valid which is not guaranteed.

Although we plan to emulate the important features of each RCT as closely as possible in healthcare claims, there may be some elements of RCT design that are not emulable with a database study, which means that the RWE and RCT will address slightly different clinical questions. For example, in routine clinical care, adherence to treatment is typically not as high as it is in an RCT with strong measures in place to encourage adherence to the study protocol. This means that there is more discontinuation and short-term medication use in the patients identified in claims databases than trial participants.

Apparent agreement between RCT and database study results could occur if the effects of multiple factors (chance, emulation differences, bias) cancel each other out.

# 8. Protection of human subjects

This study has been approved by the Brigham and Women's Hospital Institutional Review Board.

# 9. References

- 1. Novo Nordisk Receives FDA Approval of OZEMPIC® (semaglutide) Injection For the Treatment of Adults with Type 2 Diabetes. <a href="https://www.prnewswire.com/news-releases/novo-nordisk-receives-fda-approval-of-ozempic-semaglutide-injection-for-the-treatment-of-adults-with-type-2-diabetes-300567052.html#:~:text=OZEMPIC%C2%AE%20(semaglutide)%20injection%200.5%20mg%20or%201%20mg%20was,adults%20with%20type%202%20diabetes. PR Newswire.
- 2. ClinicalTrials.gov. Trial to Evaluate Cardiovascular and Other Long-term Outcomes With Semaglutide in Subjects With Type 2 Diabetes (SUSTAIN™ 6). National Institutes of Health. Accessed April 30, 2024. <a href="https://www.clinicaltrials.gov/study/NCT01720446">https://www.clinicaltrials.gov/study/NCT01720446</a>

- 3. McGuire DK, Busui RP, Deanfield J, et al. Effects of oral semaglutide on cardiovascular outcomes in individuals with type 2 diabetes and established atherosclerotic cardiovascular disease and/or chronic kidney disease: Design and baseline characteristics of SOUL, a randomized trial. *Diabetes Obes Metab*. Jul 2023;25(7):1932-1941. doi:10.1111/dom.15058
- 4. Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. *Pharmacoepidemiol Drug Saf.* Aug 2010;19(8):858-68. doi:10.1002/pds.1926
- 5. Ray WA. Evaluating Medication Effects Outside of Clinical Trials: New-User Designs. *American journal of epidemiology*. November 1, 2003 2003;158(9):915-920. doi:10.1093/aje/kwg231
- 6. Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. *Pharmacoepidemiology and drug safety*. Jun 2010;19(6):596-603. doi:10.1002/pds.1924
- 7. Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. *Am Heart J*. Jul 2004;148(1):99-104. doi:10.1016/j.ahj.2004.02.013
- 8. Tirschwell DL, Longstreth WT, Jr. Validating administrative data in stroke research. *Stroke; a journal of cerebral circulation*. Oct 2002;33(10):2465-70. doi:10.1161/01.str.0000032240.28636.bd
- 9. Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. *J Clin Epidemiol*. Jul 2011;64(7):749-59. doi:10.1016/j.jclinepi.2010.10.004
- 10. Sun JW, Rogers JR, Her Q, et al. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. *Med Care*. Dec 2017;55(12):1046-1051. doi:10.1097/mlr.000000000000824
- 11. Kim D, Schneeweiss S, Glynn R, Lipsitz L, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. *Journals of Gerontology: Medical Sciences*. 2017;73:980-987. doi:10.1093/gerona/glx229
- 12. Desai RJ, Rothman KJ, Bateman BT, Hernandez-Diaz S, Huybrechts KF. A Propensity-score-based Fine Stratification Approach for Confounding Adjustment When Exposure Is Infrequent. *Epidemiology*. Mar 2017;28(2):249-257. doi:10.1097/ede.00000000000595
- 13. Jarosek S. Death Information in the Research Identifiable Medicare Data. Accessed June 17, 2024. <a href="https://resdac.org/articles/death-information-research-identifiable-medicare-data">https://resdac.org/articles/death-information-research-identifiable-medicare-data</a>
- 14. Hill ME, Rosenwaike I. The Social Security Administration's Death Master File: The Completeness of Death Reporting at Older Ages. *Social Security Bulletin*. 2002;64(1):45-51.
- 15. Olubowale OT, Safford MM, Brown TM, et al. Comparison of Expert Adjudicated Coronary Heart Disease and Cardiovascular Disease Mortality With the National Death Index: Results From the REasons for Geographic And Racial Differences in Stroke (REGARDS) Study. *Journal of the American Heart Association*. May 3 2017;6(5)doi:10.1161/jaha.116.004966
- 16. Research Data Assistance Center (ResDAC). https://resdac.org/. Centers for Medicare & Medicaid Services (CMS).

# 10. Appendices

See accompanying excel file.

1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment

#### 2 Code algorithms

- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome

- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate Algorithm

# **Appendices**

- 1 Target Trial Framework, Operational Definitions and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate algorithm sources

| | SOUL trial definitions | (OPTUM) | (CMS) | (MarketScan) | Notes/Questions | Color coding |
|---|---|---|---|---|---|---|
| ent assignment (time 0,<br>Index date) | Parallel, blinded randomization to treatment A vs B | criteria) | Non-randomized initiation of treatment A vs B<br>(first eligible entry to study population after applying inclusion-exclusion<br>criteria) | Non-randomized initiation of treatment A vs B<br>(first eligible entry to study population after applying inclusion-<br>exclusion criteria) | | |
| Exposure | Semaglutide: Increasing doses (3 mg/7 mg/14 mg) of semaglutide tablets to<br>be taken with water at the same time every morning in a fasting state | Washout window: [-180, -1] Inoldent with respect to: both exposure and reference Source of algorithm: N/A Messurement characteristics: n/a | Code type: NDC Generic Care setting: Drug Diagnosis position: 1/A Washort window: [-180, -1] Incidient with respect to: both exposure and reference Source of algorithm: 1/A Messurement chearcteristics: Oral only | Code type: NDC Generic Care setting: Drug Diegnoeis poetitor: N/A Washout window: [-180, -1] incident with respect to: both exposure and reference Source of algorithm: N/A Messurement characteristics: Oral only | We defined oral semaglutide using ndc codes and generic name with route of administration | Good proxy definition |
| Comparator | Placebo: Placebo tablets to be taken with water at the same time every morning in a fasting state | Code type: NDC Generic Care setting: Presciption Claims Diagnosis position: N/A Washout window: [-180,-1] Incident with respect to: both exposure and reference Source of algorithm: N/A Measurement characteristics: n/a | Code type: NDC Generic Care setting: Presiciption Claims Diagnosis position: N/A Washout window: [-180, -1] Incidient with respect to: both exposure and reference Source of algorithm: N/A Measurement characteristics: n/a | Code type: NDC Generic Care setting: Presciption Claims Diegnoeis poetiton: N/A Washout window: [-180, -1] Incident with respect to: both exposure and reference Source of algorithm: N/A Measurement characteristics: n/A | We used sitagliptin as an active comparator proxy for placebo. We allowed sitagliptin alone or in combination pills with metformin only. | Moderate proxy definition |
| Primary Outcome | Time to first occurrence of a major adverse cardiovascular event (MACE), a composite endpoint consisting of cardiovascular (CV)death/non-fatal myocardial infarction/non-fatal stroke (Time Frame: From randomisation (week 0) to end-of-trial (up to 61 months ormore) (trial is event driven) ] | Code type: DX Care setting: Inpatient Diagnosis position: Primary for Stroke, Any for MI Weshout Window: Source of algorithm: PROMISE team Messurement characteristics: PY for MI using ICD9 codes was 8.8.4% and 94% [https://pubmed.ncbi.nlm.nih.gov/20140892/ and nttps://pubmed.ncbi.nlm.nih.gov/15215788/] PY for ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.nlm.nih.gov/1234739/ and nttps://pubmed.ncbi.nlm.nih.gov/20140892/] Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | Code type: DX Care setting: Inpatient Diagnosis position: Primary for Stroke, Any for MI Weshout window: Source of algorithm: PROMISE team Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94% [Intps://pubmed.ncbi.nlm.nim.gov/2014.0932/ and https://pubmed.ncb.inm.nim.gov/1521.5798/] PPV for ischemic stroke using ICD9 codes was 88% and 95% [Intps://pubmed.ncb.inm.nim.gov/12364739/ and | Code type: DX Care setting: Inpatient Diagnosis position: Primary for Stroke, Any for MI Weshout window: Source of algorithm: PROMISE team Messurement characteristics: PPV for MI using ICDS codes was 88.4% and 94%: [https://pubmed.ncbi.nlm.nim.gov/20140982/ and https://pubmed.ncbi.nlm.nim.gov/20140982/ and https://pubmed.ncbi.nlm.nim.gov/20140982/ and https://pubmed.ncbi.nlm.nim.gov/20140982/ BBM and 45% [https://pubmed.ncbi.nlm.nim.gov/20140892/] BBM of the above ICDS codes were mapped to ICD10, but no validation study was performed. | Optum death includes information from the inpatient discharged dead status, social security death master file, and deaths straped from obtusines or other sources. MarketScan includes information from the inpatient descharged dead status up until 2016. Medicare includes information from the inpatient descharged dead status, NOT cause of death, and social security death master file. | Poorly measured in database but not critical for the analysis |
| Follow up start | t Randomization date | Date of initiation of treatment A vs B | Date of initiation of treatment A vs B | Date of initiation of treatment A vs B | | Poorly measured and important for the |
| | Up to 61 months | Earliest of: outcome, end of observation in data, end of study period, discontinuation, switch to opposite arm, switch to other glp1/injection semaglutide, or 365 days. | Earliest of: outcome, end of observation in data, end of study period, discontinuation, switch to opposite arm, switch to other glp1/injection semaglutide, or 365 days. | Earliest of: outcome, end of observation in data, end of study period, discontinuation, switch to opposite arm, switch to other glp1/injection semaglutide, or 365 days. | | aliarysis |
| Causal estimand<br>Effect estimation | | On-treatment | On-treatment | On-treatment | | 1 |
| Inclusion criteria | Cox proportional nazards model | Applied before/after selection of Index date: Before | + | Applied before/after selection of Index date: Before | | † |
| 1 | Diagnosed with Type 2 diabetes mellitus HDA1c between 6.5% and 10.0% (47 - 86 mmol/mol) reflected in the latest available lab | Assessment window: [Start of all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: n/a | Assessment window; [Start of all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: n/a | Assessment Window; [Start of all available data, 0] Code type; DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics; n/a | | |
| 2 | data that would not be more than 30 days old | Can't be measured in claims but not important for the analysis | Can't be measured in claims but not important for the analysis | Can't be measured in claims but not important for the analysis | | |
| 3 | Male or female, age equal to or above 50 years at the time of signing informed consent | Applied before/after selection of Index date: Before Assessment window: [0, 0] Code type: N/A Care settins: N/A | Applied before/after selection of Index date: Before Assessment window: [0, 0] Code type: N/A Care setting: N/A | Applied before/after selection of Index date: Before Assessment window: [0, 0] Code type: N/A | | |
| 4 | At least one of the following conditions: | Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A | Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A | Core setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A | | , |
| 4 | At least one of the following conditions: Coronary heart disease defined by at least one of the following criteria: I. Prior myocardial infarction II. Prior cronnary researchistation procedure II. 50% or above stenois in coronary artery documented by cardiac catheterization, computerized tomography coronary anglography IV. Coronary heart disease with schaemia documented by stress test with any imaging modality | Diagnosis position: N/A<br>Source of algorithm: N/A | Diagnosis position: N/A<br>Source of algorithm: N/A | Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A | We defined by old MI, acute MI, previous CABG/PTCA/Stent procedures, history of CABG/PTCA diagnoses, Stable angina, coronary atherosclerosis | |
| 4 | Coronary heart disease defined by at least one of the following criteria: L. Prior myocardial infarction II. Prior croonary revascularization procedure II. 95% or above stenosis in coronary artery documented by cardiac catheterization, computerized tomography coronary angiography N. Coronary heart disease with incidenation documented by stress test with any imaging | Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: [Start of all available data, 0] Code type: DX, PX Core setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, Investigator reviwed codes | Diagnosis position: IV/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: [Start of all available data, 0] Code type IX, FX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, investigator reviwed codes | Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [Start of all available data, 0] Code type: D/C Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, investigator reviwed codes | CABG/PTCA/Stent procedures, history of CABG/PTCA | |
| 4 | Coronary heart disease defined by at least one of the following criteria: I. Prior myocardial infarction II. Prior cromary revascularization procedure III. Prior cromary revascularization procedure III. Softs or above stenois in coronary artery documented by cardiac catheterization, computerized tomography coronary angiography V. Coronary heart disease with ischaemia documented by stress test with any imaging modality Cerebrovascular disease with inchaemia documented by stress test with any imaging modality Cerebrovascular disease defined by at least one of the following criteria: I. Prior stroke II. Prior carotida artery revascularization procedure III. Prior stroke III. Prior stroke III. Prior stroke | Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [Start of all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, Investigator reviwed codes Measurement characteristics: n/a Applied before/after selection of index date: Before Assessment window: [Start of all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Diagnosis position: IV/A Source of algorithm: IV/A Measurement characteristics; IV/A Applied before/after selection of Index date: Before Assessment window: [Start of all available data, 0] Code type: IV, EX Care settling: Any Source of algorithm: PROMISE team, Investigator reviwed codes Measurement characteristics: IV/A Applied before/after selection of Index date: Before Assessment window: [Start of all available data, 0] Code type: IV, EX Care settling: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team | Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Applied before/after selection of Index date: Before Assessment window: [Start of all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team, investigator reviewd codes Measurement characteristics: n/a Applied before/after selection of Index data: Before Assessment window: [Start of all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team | CABG/PTCA/Stent procedures, history of CABG/PTCA diagnoses, Stable angina, coronary atherosclerosis | |

| | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of Index date: Before | |
|---|---|---|---|---|
| | Assessment window: [-180, 0] | Assessment window: [-180, 0] | Assessment window: [-180, 0] | |
| | Code type: DX | Code type: DX | Code type: DX | |
| Chronic kidney disease defined as: i. eGFR below 60mL/min/1.73 m^2 (based on med records using latest available and no more than 6 months old assessment) | Diagnosis position: Any | Care setting: Any | Care setting: Any | We defined using CKD3/4 |
| records using latest available and no more than 6 months old assessment) | | Diagnosis position: Any | Diagnosis position: Any | - ' |
| | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| | Measurement characteristics: n/a | Measurement characteristics: n/a | Measurement characteristics: n/a | |
| eria | | | | |
| lia . | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | |
| | Assessment window: [-60, 0] | Assessment window: [-60, 0] | Assessment window: [-60, 0] | |
| Any of the following: myocardial infarction, stroke, hospitalisation for unstable angina | | Code type: DX | Code type: DX | |
| 1 pectoris or transient ischaemic attack within thevpast 60 days prior to the day of | Care setting: Inpatient | Care setting: Inpatient | Care setting: Inpatient | |
| screening | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any | |
| | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| | Messurement characteristics: n/a | Measurement characteristics: n/a | Measurement characteristics: n/a | |
| Planned coronary, carotid, or peripheral artery revascularization known on the day of | Can't be measured in claims | Can't be measured in claims | Can't be measured in claims | |
| screening | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | |
| | Assessment window:[-180.0] | Assessment window:[-180.0] | Assessment window:[-180, 0] | |
| | Code type: DX, PX | Code type: DX. PX | Code type: DX, PX | |
| | Care setting: DX Inpatient confinement only, PX - Any | Care setting: DX Inpatient confinement only, PX - Any | Care setting: DX Inpatient confinement only, PX - Any | We defined it by occurrence of heart failure in i |
| 3 Heart failure presently classified as being in New York Heart Association Class IV | Diagnosis position: Any | | Diagnosis position: Any | we defined it by occurrence of neart failure in i |
| | | Diagnosis position: Any | | setting with oxygen use |
| | Source of algorithm: Promise team, Frailty score<br>Measurement characteristics: n/a | Source of algorithm: Promise team, Frailty score<br>Measurement characteristics: n/a | Source of algorithm: Promise team, Frailty score Measurement characteristics: n/a | |
| | Measurement characteristics: n/a | Measurement characteristics: n/a | Measurement characteristics: n/a | |
| | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | |
| | Assessment window: [-180, 0] | Assessment window: [-180, 0] | Assessment window: [-180, 0] | |
| | Code type: RX | Code type: RX | Code type: RX | We used GLP1 agonists/DDP4/Pramlintide and |
| 4 Treatment with any glucagon-like peptide-1 receptor agonist within 30 days before | Care setting: N/A | Care setting: N/A | Care setting: N/A | using look back window of 180 days rather tha |
| screening | Diagnosis position: N/A | Diagnosis position: N/A | Diagnosis position: N/A | days |
| | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A | |
| | Measurement characteristics: n/a | Measurement characteristics: n/a | Measurement characteristics: n/a | |
| | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | |
| | Assessment window: [-180, -1] | Assessment window: [-180, -1] | Assessment window: [-180, -1] | |
| 0 4 1 | Code type: NDC | Code type: NDC | Code type: NDC | |
| 15 Semaglutide | Care setting: N/A | Care setting: N/A | Care setting: N/A | |
| | Diagnosis position: N/A | Diagnosis position: N/A | Diagnosis position: N/A | |
| | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A | |
| | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | Applied before/after selection of index date: Before | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | |
| | Assessment window: [-180, 0] | Assessment window: [-180, 0] | Assessment window: [-180, 0] | |
| | Code type: DX | Code type: DX | Code type: DX | |
| 5 History of MEN-2 or family history of medullary thyroid cancer | Care setting: Any | Care setting: Any | Care setting: Any | |
| | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any | |
| | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | Applied before/after selection of Index date: Before Assessment window: [-180, 0] | Applied before/after selection of Index date: Before Assessment window: [-180, 0] | Applied before/after selection of Index date: Before Assessment window: [-180, 0] | |
| | Code type: DX | | | |
| 8 m | | Code type: DX | Code type: DX | |
| 6 History of pancreatitis | Care setting: Any Diagnosis position: Any | Care setting: Any Diagnosis position: Any | Care setting: Any Diagnosis position: Any | |
| | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| | Measurement characteristics; N/A | Measurement characteristics; N/A | Measurement characteristics: N/A | |
| | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | |
| | Assessment window: [Start of all available data, 0] | Applied belong and delection of mack data. Select | | |
| | | Acceptant window: (Start of all available data (1) | Acceptant window: [Start of all available data 0] | |
| | | Assessment window: [Start of all available data, 0] | Assessment window: [Start of all available data, 0] | |
| History of or planning bariatric surgery, including banding procedures or | Code type: PX | Code type: PX | Code type: PX | Cannot canture planned surderies |
| 7 History of or planning bariatric surgery, including banding procedures or surgical gastric and/or intestinal bypass | Code type: PX<br>Care setting: Any | Code type: PX<br>Care setting: Any | Code type: PX<br>Care setting: Any | Cannot capture planned surgeries |
| | Code type: PX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis position: Any | Cannot capture planned surgeries |
| | Code type: PX<br>Care setting: Any<br>Diagnosis position: Any<br>Source of algorithm: PROMISE team | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Cannot capture planned surgeries |
| | Code type: PX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis position: Any | Cannot capture planned surgeries |
| | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: (1508) | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [130.0] | Code type: PX Care setting: Any Diagnosis poettion: Any Bource of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1:80, 0] | Cannot capture planned surgeries |
| surgical gastric and/or intestinal bypass | Code type: PX Care setting: Any Diagnosis poeition: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index data: Before Assessment window: [180, 0] Code type: DX, PX | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristica: N/A Applied before/after selection of Index data: Before Assessment window: [-180, 0] Code type: DX, PX | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [150, 0] Code type: DX, PX | Cannot capture planned surgeries |
| | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment windows (180.0) | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [130.0] | Code type: PX Care setting: Any Diagnosis poettion: Any Bource of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1:80, 0] | Cannot capture planned surgeries Cannot capture planned pregnancies |
| surgical gastric and/or intestinal bypass | Code type: PX Care setting: Any Diagnosis poetition: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis poetition: Any | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any | |
| surgical gastric and/or intestinal bypass | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IV/A Applied before/after selection of Index data: Before Assessment window: [1:50.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Prepancy team | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics. N/A Applied before/arter selection of Index date: Before Assessment window: [180, 0] Code type: DX, PY Care setting: Any Diagnosis position: Any Source of algorithm: Presenancy team | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of align/thm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: (150. 0) Code type: DX, PX Care setting: Any Diagnosis position: Any Source of selection: Prepagacy team | |
| surgical gastric and/or intestinal bypass | Code type: PX Care setting: Any Diagnosis poetition: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Code tyne: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/Arter selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Anny Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | |
| surgical gastric and/or intestinal bypass | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index data: Before Assessment window: [1.50.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Prepancy team Measurement characteristics: IVA Applied before/after selection of index data: Before | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Measurement characteristics: N/A Applied before; Arfair selection of Index data: Before Assessment window: 1:80. 0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before; Arfair selection of Index data: Before | Code type: PX Care setting: Any Diagnosis position: Any Source of sligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: 1:50. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before | |
| surgical gastric and/or intestinal bypass | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1826, 0] | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/arter selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/arter selection of Index date: Before Assessment window: [1825, 0] | Code type: PX Care setting: Any Diagnosis poetion: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: (136.0) Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: (1363.0) | |
| surgical gastric and/or intestinal bypass Plans for pregnancy during the course of the study for women of child-bearin potential | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window; [1:80.0] Gode type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: IV/A Applied before/after selection of Index date: Before Assessment window; [1:825, 0] Code type: CX | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before, After selection of Index date: Before Assessment window: [180, or] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825, o] Code type: DX | Code type: PX Care setting: Any Diagnosale position: Any Source of algorithm: PROMISE team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1-80.0] Code type: DX, PX Care setting: Any Diagnosale position: Any Source of algorithm: Pregnancy team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1-82.5.0] Code type: DX Code type: DX | |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: [1:80, 0] God type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: [1:825, 0] Code type: DX. Care setting: Any Care setting: Any Care setting: Any Care setting: Any | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825, 0] Code type: DX Care setting: Any | Code type: PX Care setting: Any Diagnosis poetton: Any Bource of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [158.0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825.0] Code type: DX Care setting: Any Care setting: Any | |
| Surgical gastric and/or intestinal bypass Plans for pregnancy during the course of the study for women of child-bearin potential | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/share selection of index date: Before Assessment window: [180.0] Gode type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/safers selection of index date: Before Assessment window: [1825, 0] Code type: DX UPPY Care setting: Any Diagnosis position: N/A Diagnosis position: N/A Diagnosis position: N/A Diagnosis position: N/A | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before, After selection of Index date: Before Assessment window: [180, or] Code type: DX, PX Care setting: Any Diagnosis position: Any Bource of algorithm: Pregnancy team Measurement characteristics: N/A Applied beforte/after selection of Index date: Before Assessment window: [1825, o] Code type: DX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosale position: Any Source of algorithm: PROMISE team Messurement characteristics: N/A Applied before/ after selection of Index date: Before Assessment window: [1-50, 0] Code type: DX, PX Care setting: Any Diagnosale position: Any Source of algorithm: Pregnancy team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1-825, 0] Code type: DX Care setting: Any Diagnosale position: Any | |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithms: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: [1:80, 0] Gode type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithms: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index data: Before Assessment window: [1:825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithms: PROMISE team | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics. N/A Applied before/arter selection of Index date: Before Assessment window: [180.0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/arter selection of Index date: Before Assessment window: [1825.0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Code type: PX Care setting: Any Diagnosis poettion: Any Source of align/thm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [150, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of align/thm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1525, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of align/thm: PROMISE team | |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/share selection of index data: Before Assessment window; [180.0] Gode type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/syster selection of index data: Before Assessment window; [1825, 0] Code type: DX Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before, After selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied beforter/after selection of Index date: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Code type: PX Care setting: Any Diagnosale position: Any Source of algorithm: PROMISE team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: 1-180. 0] Code type: DX, PX Care setting: Any Diagnosale position: Any Source of algorithm: Pregnancy team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: (-1825, 0] Code type: DX Care setting: Any Diagnosale position: Any Source of algorithm: PROMISE team Messurement characteristics: N/A | |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithms: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1:80.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithms: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1:825.0] Care setting: Any Diagnosis position: Any Source of algorithms: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Measurement characteristics: N/A Applied before/after selection of Index date: Before | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics. N/A Applied before/arter selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before | Code type: PX Care setting: Any Diagnosis poettion: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [150. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1525. 0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | |
| Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1825, 0] Code type: DX Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1825, 0] | Code type: PX Care setting: Any Diagnosis position: any Diagnosis position: any Source of algorithm: PPOMISE team Measurement ohereotestation: M/A Applied bofrey, fater selection of Index date: Before Assessment window: [1-80, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/afface selection of Index date: Before Assessment window: [1-82:5, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/afface selection of Index date: Before Assessment window: [1-80:0] | Code type: PX Care setting: Any Diagnosis position: Any Source of sigorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1-50, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of sigorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1-52, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1-50, 0] | Cannot capture planned pregnancies |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window: [1:80.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window: [1:825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window: [1:80, 0] Code type: DX Applied before/after selection of index date: Before Assessment window: [1:80, 0] Code type: DX. PX | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Code Sper DX Code Sper DX Code | Code type: PX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of aligorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-180, 0] Code type: DX, PX Code bype: DX, PX | Cannot capture planned pregnancies |
| Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825, 0] Code type: DX Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX Care setting: Any Code type: DX Code ty | Code type: PX Care setting: Any Diagnosis position: any Diagnosis position: any Source of algorithm: PPOMISE team Measurement characteristics: 1/2 Applied bofres/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Code type: DX, PX Care setting: Any | Code type: PX Care setting: Any Diagnosis position: Any Source of sigorithm: PROMISE team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of sigorithm: Pregnancy team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of sigorithm: PROMISE team Messurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX Care setting: Any Code type: DX Care setting: Any Code type: DX Care setting: Any Code type: DX Care setting: Any | Cannot capture planned pregnancies |
| Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window: [1:50.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Prepancy team Measurement characteristics: IVA Applied before/after selection of Index date: Before Assessment window: [1:52.5, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of Index date: Before Assessment window: [1:50.0] Code type: DX Care setting: Any Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis poeition: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of aligorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any | Cannot capture planned pregnancies We defined it based on CKDS, ESRD, Dialysis |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1:80, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1:8:25, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1:80, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement window: [1:80, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/arter selection of Index date: Before Assessment window: [130, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/arter selection of Index date: Before Assessment window: [130, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [130, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team | Code type: PX Care setting: Any Diagnosis poetton: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-150, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of aligorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Dource of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of aligorithm: PROMISE team | Cannot capture planned pregnancies We defined it based on CKDS, ESRD, Dialysis |
| Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index data: Before Assessment window: [±50.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Prepancy team Measurement characteristics: IVA Applied before/after selection of index data: Before Assessment window: [±52.0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index data: Before Assessment window: [±50.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Messurement characteristics: IVA | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before/Arier selection of Index data: Before Assessment window: 1:880.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: NA Applied before/Arier selection of Index data: Before Assessment window: [:825, 0] Code type: DX. Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before/Arier selection of Index data: Before Assessment window: [-180, 0] Code type: DX. PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Code type: PX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: 1:50. 0 Code type: DX, PX Care setting: Any Diagnosis position: Any Source of aligorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [:1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [:180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Source of aligorithm: PROMISE team Measurement characteristics: N/A | Cannot capture planned pregnancies We defined it based on CKDS, ESRD, Dialysis |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied befroy: After selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied befroy: After selection of Index date: Before Assessment window: [-1825, 0] Code type: DX Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied befrore/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/yefter selection of Index date: Before | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics. N/A Applied before/arter selection of Index date: Before Assessment window: [130. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1325. 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [130, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Measurement characteristics: N/A Applied before/after selection of Index date: Before | Code type: PX Care setting: Any Diagnosis poetton: Any Source of align/thm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [150, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of align/thm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1525, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of align/thm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [150, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of align/thm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Measurement characteristics: N/A Applied before/after selection of index date: Before | Cannot capture planned pregnancies We defined it based on CKDS, ESRD, Dialysis |
| B Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window; [±9.0.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: IVA Applied before/after selection of index date; Before Assessment window; [±825, 0] Code type: DX Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window; [±80, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date; Before Measurement characteristics: IVA Applied before/after selection of index date; Before Assessment window: 1500.01 | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before; Arfair selection of Index data: Before Assessment window: [180. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: NA Applied before; Arfair selection of Index data: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; Arfair selection of Index data: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; Affair selection of Index data: Before Assessment window: [180, 0] | Code type: PX Care setting: Any Diagnosis position: Any Source of signrithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: 1:50. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of signrithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: 1:825. 0] Code type: DX Care setting: Any Diagnosis position: Any Source of signrithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: 1:20. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of signrithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: 1:20. 0] Source of signrithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: 1:30. 0] | Cannot capture planned pregnancies We defined it based on CKDS, ESRD, Dialysis |
| Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal impairment (corresponding to eGFR <30 ml/min/1.73 m2) | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/arter selection of index date: Before Assessment window: [1:50.0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/arter selection of index date: Before Assessment window: [1:825.0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80,0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80,0] Code type: DX. PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:50,0] Code type: PX | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics. N/A Applied before/arter selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: DX PX Applied before/after selection of Index date: Before Assessment window: [180, 0] Code type: PX | Code type: PX Care setting: Any Diagnosis poetion: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:925. 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80, 0] Code type: DX Care setting: Any Diagnosis position: Any Bource of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80, 0] Code type: PX | Cannot capture planned pregnancies We defined it based on CKD5, ESRD, Dialysis transplant |
| Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window; [180.0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window; [1825, 0] Code type: DX Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window; [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [180, 0] Code type: PX Care setting: Any | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; Arfair selection of Index data: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before; Arfair selection of Index data: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; After selection of Index data: Before Assessment window: [180, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; After selection of Index data: Before Assessment window: [180, 0] Code type: PX Care setting: Any Care setting: Any Care setting: Any | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: PX Care setting: Any | Cannot capture planned pregnancies We defined it based on CKD5, ESRD, Dialysis of transplant |
| Plans for pregnancy during the course of the study for women of child-bearin potential Plistory of cancer, other than non-melanoma skin cancer, that required there in the S years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal impairment (corresponding to eGFR <30 ml/min/1.73 m2) | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IV.A Applied before/arter selection of index date: Before Assessment window: [180.0] Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: IV.A Applied before/after selection of Index date: Before Assessment window: [1828, 0] Code type: IV. Care setting: Any Diagnosis position: PROMISE team Measurement characteristics: IV.A Applied before/after selection of Index date: Before Assessment window: [180.0] Code type: IV. PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IV.A Applied before/after selection of Index date: Before Assessment window: [180.0] Code type: IV. PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IV.A Applied before/after selection of Index date: Before Assessment window: [180.0] Code type: IV. Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/arter selection of Index date: Before Assessment window: [-180, o] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-1825, o] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, o] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, o] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, o] Code type: PX Care setting: Any Diagnosis position: Any | Code type: PX Care setting: Any Diagnosis poeition: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [1:80. 0] Code type: DX, PX Care setting: Any Diagnosis poeition: Any Diagnosis poeition: Any Source of aligorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [1825. 0] Code type: DX, Care setting: Any Diagnosis poeition: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180. 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of aligorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [180. 0] Code type: PX Care setting: Any Diagnosis position: Any | Cannot capture planned pregnancies We defined it based on CKD5, ESRD, Dialysis of transplant |
| Plans for pregnancy during the course of the study for women of child-bearin potential History of cancer, other than non-melanoma skin cancer, that required there in the 5 years prior to randomization Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal impairment (corresponding to eGFR <30 ml/min/1.73 m2) | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window; [180.0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: IVA Applied before/after selection of index date: Before Assessment window; [1825, 0] Code type: DX Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window; [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [180, 0] Code type: PX Care setting: Any | Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; Arfair selection of Index data: Before Assessment window: [180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before; Arfair selection of Index data: Before Assessment window: [1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; After selection of Index data: Before Assessment window: [180, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before; After selection of Index data: Before Assessment window: [180, 0] Code type: PX Care setting: Any Care setting: Any Care setting: Any | Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-1825, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of Index date: Before Assessment window: [-180, 0] Code type: PX Care setting: Any | Cannot capture planned pregnancies We defined it based on CKD5, ESRD, Dialysis o |
| | | · | , | |
|---|---|---|---|---|
| | | Applied before/after selection of Index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of Index date: Before |
| | | Assessment window: [-180, 0] | Assessment window: [-180, 0] | Assessment window: [-180, 0] |
| | | Code type: DX, PX | Code type: DX, PX | Code type: DX, PX |
| 12 | History of diabetic ketoacidosis | Care setting: Any | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team |
| | | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of Index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of Index date: Before |
| | | Assessment window: [-180, 0] | Assessment window: [-180, 0] | Assessment window: [-180, 0] |
| | | Code type: Discharge Status Code, CPT/HCPCS Procedure Code, | Code type: Discharge Status Code, CPT/HCPCS Procedure Code, Provider | Code type: Discharge Status Code, CPT/HCPCS Procedure Code, |
| | | Provider Category Code | Category Code | Provider Category Code |
| 13 | Nursing home | Care setting: Any | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team |
| | | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A |
| I | | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before | Applied before/after selection of Index date: Before |
| | | Assessment window: [0, 0] | Assessment window: [0, 0] | Assessment window: [0, 0] |
| | | Code type: N/A | Code type: N/A | Code type: N/A |
| 14 | Age Gender missing<br>Excluded if last recorded value is missing | Care setting: N/A | Care setting: N/A | Care setting: N/A |
| | excluded it last recorded value is missing) | Diagnosis position: N/A | Diagnosis position: N/A | Diagnosis position: N/A |
| | | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A |
| | | | | Measurement characteristics: N/A |


| Contentional promotion 1971-16 P. | Cerebrovascular procedure | 037H0ZZ | PX | ICD-10 | DIJATION OF RIGHT COMMON CAROTID ARTERY, OPEN APPROACH | Cerebrovascular disease component |
|---|---|---|---|---|---|---|
| Continuous promotive | | | PX | ICD-10 | DILATION OF RIGHT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH | |
| Continuous Christian Continuous Cont | | | | | | |
| Cardiovariate provider | | | | ICD-10 | | |
| Communication Communicatio | Cerebrovascular procedure | 037H35Z | PX | ICD-10 | DILATION OF RIGHT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH | Cerebrovascular disease component |
| Continuous procedure | Cerebrovascular procedure | 037H366 | PX | ICD-10 | DILATION OF RIGHT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROA | Cerebrovascular disease component |
| Contentionating procedure Contentional pro | Cerebrovascular procedure | 037H36Z | PX | ICD-10 | | |
| Certificational promotion Certification | Cerebrovascular procedure | | | | | Cerebrovascular disease component |
| Certification production Company | | | | | | |
| Contemporation Cont | | | | | | · |
| Continuous products | · | | | | | · |
| Continuous Chipped P. C. D. D. D. D. D. D. D | | | | | , | |
| Certiferenous 1979-16 P. C. C. DATA/GOO BIOR COMMON (ACRID) ARTIFES HIS INTERNATIONAL PROPRIATE PRICE ARTIFICATION ASSIGNATION Certiferenous C. Certiferenous C. C. C. DATA/GOO BIOR COMMON (ACRID) ARTIFICATION PRICE PRI | | | | | | |
| Control Cont | | | | | | |
| Certamonical procedure CEPTING | | | | | | |
| Certificacional procedure O379-152 FX CO-10 Delando OF Reint COMMON (ARTIDID ARTITIC) FREICULATION, SPRINGART Certificacional procedure O379-162 FX CO-10 Delando OF Reint COMMON (ARTIDID ARTITIC) FREICULATION, SPRINGART Certificacional disease component Certificacional procedure O379-162 FX CO-10 Delando OF Reint COMMON (ARTIDID ARTITIC) FREIDULATION, SPRINGART CERTIFICACION (ARTIDID ARTITIC) FREIDULATION (ARTIDIO ARTITIC) FREIDULATION (ARTITIC) FREIDULATION ( | | | | | | |
| Cerebrosocular presented | | | | | · | |
| Certificacidar procedure | • | | | | | |
| Certiferoscolar procedure Certiferoscolar pr | | | | | · | |
| Cerebrosscalar procedure 971H45 PK CLD DILATION OF BROTH COMMON LABOTION ARTITLY, MININE AND DILAS, ALTITUM ROUTH MININES, PRECUTANCIUS BROCKED Cerebrosscalar disease component (Cerebrosscalar procedure 037H46 PK CLD DILATION OF BROTH COMMON LABOTION ARTITLY, MININES DILATION ARTITLA, MININES DILATION OF BROTH COMMON LABOTION ARTITLY, MININES DILATION ARTITLA, MININES DILATION OF BROTH COMMON LABOTION ARTITLY, MININES DILATION ARTITLA, MININES DILATION A | | | | | | |
| Cerebroscolar procedure 0,77452 PX CD-10 DUATHON OF RIGHT COMMON CARGITO ARTERY WITH TWO DRUG-ELUTING INTRALLMINAL DEVICES, PRECURATIONS ENDOSCOPE, APPROACH Cerebroscular disease component cerebroscoper in control of the process of the | | | | | | |
| Certificroscalar pricedure 0.371446 PX | · | | | | | |
| Cerebrosocation procedure | | | | | | |
| Cerebro-vascular procedure | | | | | | |
| Cerebrovascular procedure | | | | | | |
| Cerebrovascular procedure 0371466 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH HITRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular procedure 0371476 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH YOU PATRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular procedure 0371476 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH YOU PATRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular procedure 0371476 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH YOU PATRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular procedure 037146 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH YOU PATRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular procedure 0371477 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH ACTION, WITH THE REPORT COMMON CARDITO AFTER WITH THE DIR ON ARRIVE METABLUMINAL DEVICES, PERCURS AFTER COMMON CARDITO AFTER WITH THE DIR ON ARRIVE METABLUMINAL DEVICES, PERCURS AFTER COMMON CARDITO AFTER WITH THE DIR ON ARRIVE METABLUMINAL DEVICES, OPEN APPROACH Cerebrovascular procedure 0371602 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH THE DIR ON ARRIVE METABLUMINAL DEVICES, OPEN APPROACH Cerebrovascular procedure 0371602 PX (CD-10 DILATION OF RIGHT COMMON CARDITO AFTER WITH THE DIR ON ARRIVE METABLUMINAL DEVICES, OPEN APPROACH CEREBROVASCULAR DEV | | 037H47Z | PX | | DILATION OF RIGHT COMMON CAROTID ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC A | Cerebrovascular disease component |
| Cerebrosscular procedure 037H45 PX (C.)10 DILATION OR RIGHT COMMON CARDID ARTERY, BIFULCATION, WITH TWO INTRALLIMINAL EDVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H47 PX (C.)10 DILATION OR RIGHT COMMON CARDID ARTERY, BIFULCATION, WITH THEE BITTALLIMINAL EDVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H47 PX (C.)11 DILATION OR RIGHT COMMON CARDID ARTERY, BIFULCATION, WITH THEE BITTALLIMINAL EDVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H47 PX (C.)11 DILATION OR RIGHT COMMON CARDID ARTERY, BIFULCATION, WITH TOUR OR MORE INTRALLIMINAL EDVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)11 DILATION OR RIGHT COMMON CARDID ARTERY, BIFULCATION, WITH TOUR OR MORE INTRALLIMINAL EDVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)12 DILATION OR RIGHT COMMON CARDID ARTERY, BIFULCATION, WITH TOUR OR MORE INTRALLIMINAL EDVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)12 DILATION OR RIGHT COMMON CARDID ARTERY, BIFULTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)12 DILATION OR RIGHT COMMON CARDID ARTERY WITH TOUR OR MORE INTRALLIMINAL EDVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)12 DILATION OR RIGHT COMMON CARDID ARTERY WITH TOUR OR MORE INTRALLIMINAL EDVICES, OPEN APPROACH Cerebrosscular procedure 037H40 PX (C.)12 DILATION OR FIRST COMMON CARDID ARTERY WITH TOUR OR MORE INTRALLIMINAL EDVICES, OPEN APPROACH Cerebrosscular procedure 037H40 PX (C.)12 DILATION OF BIFT COMMON CARDID ARTERY WITH TOUR OR MORE BUILDING ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)13 DILATION OF BIFT COMMON CARDID ARTERY WITH TOUR OR MORE BUILDING ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)13 DILATION OF BIFT COMMON CARDID ARTERY WITH TOUR OR MORE BUILDING ENDOSCOPIC APPROACH Cerebrosscular procedure 037H40 PX (C.)13 DILATION OF BIFT COMMON CARDID ARTERY WITH TOUR OR BUILDING ENDOSCOPIC APPROACH Cerebrosscul | Cerebrovascular procedure | 037H4D6 | PX | ICD-10 | DILATION OF RIGHT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH | Cerebrovascular disease component |
| Cerebrovascular procedure 037H4Z PK CD-10 DIATION OF RIGHT COMMON CARDTO ARTEN WITH TWO NITRALLMANAL EPINCES, PRECUTANCIUS ENDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037H4Z PK CD-10 DIATION OF RIGHT COMMON CARDTO ARTEN WITH THE IRRALLMANIAL DEVICES, PRECUTANCIUS ENDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037H4Z PK CD-10 DIATION OF RIGHT COMMON CARDTO ARTEN WITH THE IRRALLMANIAL DEVICES, PRECUTANCIUS ENDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037H4Z PK CD-10 DIATION OF RIGHT COMMON CARDTO ARTEN WITH THE IRRALLMANIAL DEVICES, PRECUTANCIUS ENDOSCOPIC ACPROACH Cerebrovascular disease component cerebrovascular procedure 037H4Z PK CD-10 DIATION OF RIGHT COMMON CARDTO ARTEN, WITHOUT THE UNIVERSAL DEVICES, PRECUTANCIUS ENDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037H4Z PK CD-10 DIATION OF RIGHT COMMON CARDTO ARTEN, WITHOUT THE UNIVERSAL DEVICES, PRECUTANCIUS ENDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037H6Z PK CD-10 DIATION OF RIGHT COMMON CARDTO ARTEN, WITHOUT THE UNIVERSAL DEVICES, CPRIA APPROACH CEREBROVASCULAR disease component cerebrovascular procedure 037H6Z PK CD-10 DIATION OF LETT COMMON CARDTO ARTEN, WITH THE RIGHT SIN WITH THE RIG | Cerebrovascular procedure | 037H4DZ | PX | ICD-10 | DILATION OF RIGHT COMMON CAROTID ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH | Cerebrovascular disease component |
| Cerebrovascular procedure 037H6F PX CD-10 DILATION OF RIGHT COMMON CARDTO ARTER, REFURCATION, WITH FREE INTRALLIMINAL DEVICES, PERCUTANEOUS RIDDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037H66 PX CD-10 DILATION OF RIGHT COMMON CARDTO DATER, REFURCATION, WITH FOUR OR MORE RITARIALIMINAL DEVICES, PERCUTANEOUS RIDDOSCOPIC A Cerebrovascular disease component cerebrovascular procedure 037H65 PX CD-10 DILATION OF RIGHT COMMON CARDTO DATER, REFURCATION, WITH FOUR OR MORE RITARIALIMINAL DEVICES, PERCUTANEOUS RIDDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037H62 PX CD-10 DILATION OF RIGHT COMMON CARDTO DATER, REFURCATION, PERCUTANEOUS RIDDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF RIGHT COMMON CARDTO DATER, PERCUTANEOUS RIDDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF RESISTATION, PERCUTANEOUS RIDDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF LEFT COMMON CARDTO DATER, PERCUTANEOUS RIDDOSCOPIC APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF LEFT COMMON CARDTO DATER, WITH TOTAL DISMANLA EDVICES, OPEN APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF LEFT COMMON CARDTO DATER WITH TOTAL DISMANLA EDVICES, OPEN APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF LEFT COMMON CARDTO DATER WITH TOTAL DISMANLA EDVICES, OPEN APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF LEFT COMMON CARDTO DATER WITH TOTAL DISMANLA EDVICES, OPEN APPROACH Cerebrovascular disease component cerebrovascular procedure 037D02 PX CD-10 DILATION OF LEFT COMMON CARDTO DATER WITH TOTAL DISMANLA EDVICES, PERCUTAN | Cerebrovascular procedure | 037H4E6 | PX | ICD-10 | DILATION OF RIGHT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH | Cerebrovascular disease component |
| Cerebrovascular procedure G7714472 PX CD-10 DILATION OF RIGHT COMMON CAROTID AFTERY, BITHITE RITHRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure G771462 PX CD-10 DILATION OF RIGHT COMMON CAROTID AFTERY, BITHITE RITHRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure G771462 PX CD-10 DILATION OF RIGHT COMMON CAROTID AFTERY WITH FURD GR MODE INTRALLUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure G771462 PX CD-10 DILATION OF RIGHT COMMON CAROTID AFTERY, BITHICATION, WITH THOUGH COMMON CAROTID AFTERY WITH TWO DEVICES (PX PAPROACH Cerebrovascular disease component Cerebrovascular procedure G77162 PX CD-10 DILATION OF RIGHT COMMON CAROTID AFTERY WITH TWO DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure G77162 PX CD-10 DILATION OF LETT COMMON CAROTID AFTERY WITH TWO DEVICES (PX PAPROACH Cerebrovascular disease component Cerebrovascular procedure G77162 PX CD-10 DILATION OF LETT COMMON CAROTID AFTERY WITH TWO DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure G77162 PX CD-10 DILATION OF LETT COMMON CAROTID AFTERY WITH TWO DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure G77162 PX CD-10 DILATION OF LETT COMMON CAROTID AFTERY WITH THOUGH CAROTID AFTERY WITH THO | Cerebrovascular procedure | 037H4EZ | | ICD-10 | | |
| Cerebrossicular procedure G371462 PX CD-10 DILATION OF RIGHT COMMON CARDITO ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLIMINAL DEVICES, PERCUTAREOUS ENDOSCOPIC A PREPOACH Cerebrossicular procedure G371426 PX CD-10 DILATION OF RIGHT COMMON CARDITO ARTERY, BIFURCATION, PERCUTAREOUS ENDOSCOPIC, APPROACH Cerebrossicular disease component Cerebrossicular procedure G371062 PX CD-10 DILATION OF RIGHT COMMON CARDITO ARTERY, BIFURCATION, PERCUTAREOUS ENDOSCOPIC, APPROACH Cerebrossicular disease component Cerebrossicular procedure G371062 PX CD-10 DILATION OF RIGHT COMMON CARDITO ARTERY, BIFURCATION, PERCUTAREOUS ENDOSCOPIC, APPROACH Cerebrossicular disease component Cerebrossicular procedure G371062 PX CD-10 DILATION OF LEFT COMMON CARDITO ARTERY WITH THOUR GORD ELUTING INTRALLIMINAL DEVICES, OPEN APPROACH Cerebrossicular disease component Cerebrossicular procedure G371002 PX CD-10 DILATION OF LEFT COMMON CARDITO ARTERY WITH THOUR GORD EQUILITIES INTRALLIMINAL DEVICES, OPEN APPROACH Cerebrossicular disease component Cerebrossicular procedure G371002 PX CD-10 DILATION OF LEFT COMMON CARDITO ARTERY WITH THOUR GORD EDIG ELUTING INTRALLIMINAL DEVICES, OPEN APPROACH Cerebrossicular disease component Cerebrossicular procedure G371002 PX CD-10 DILATION OF LEFT COMMON CARDITO ARTERY WITH THOUR CARDITO ARTERY WITH THOUR ARTERY WITH THOU | | | | | | |
| Cerebrossacular procedure | | | | | | |
| Cerebroxiscular procedure 371442 Y 10-10 DILATTON OF RIGHT COMMON CARDITO ARTERY, REFULANDOS PROSCOPIC APPROACH Cerebroxiscular disease component | | | | | | |
| Cerebrovascular procedure 37104Z PX ICD-10 DILATION OF RIGHT COMMON CARDITO ARTERY, PERCUTANEQUIS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH TINDE CRUELLING INTRALLUMINAL DEVICE, SPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH THREE DEUG-ELIUTING INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH THREE DEUG-ELIUTING INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH THREE DEUG-ELIUTING INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH THREE DEUG-ELIUTING INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH THREE DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH THREE DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37106Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY WITH THREE DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37136Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY, WITH THREE DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 37136Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY, WITH TWO DIRECTURING INTRALLUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 37136Z PX ICD-10 DILATION OF LET COMMON CARDITO ARTERY, WITH TWO DIR | | | | | | |
| Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR DELECTIONS (INTRALLIMINAL DEVICE, OPEN APPROACH 1 Cerebrosscular disease component Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH TYD QUEUE-CLIUTINS (INTRALLIMINAL DEVICES, OPEN APPROACH 1 Cerebrosscular disease component Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR OR MORE DEBUGE. QUEIN NO REPORT CAROTIO ARTEN WITH FOUR PROACH 1 Cerebrosscular disease component Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR PROACH 1 Cerebrosscular disease component Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR PROACH 1 Cerebrosscular disease component Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR PROACH 1 Cerebrosscular disease component Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR PROACH 1 Cerebrosscular disease component Cerebrosscular procedure 03706Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR PROACH 1 Cerebrosscular disease component Cerebrosscular procedure 037136Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN WITH FOUR PROACH 1 Cerebrosscular procedure 037136Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN, BILLINGARD, ON ROME INTERNALIMINAL DEVICE, PERCUTANEOUS APPROACH 1 Cerebrosscular procedure 037136Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN, BILLINGARD, ON RANGE MITTANIAL DEVICE, PERCUTANEOUS APPROACH 1 Cerebrosscular procedure 037136Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN, BILLINGARD, ON WITH FOUR CELLUTING INTRALLIMINAL DEVICE, PERCUTANEOUS APPROACH 1 Cerebrosscular procedure 037136Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN, BILLINGARD, WITH THOSE QUELLUTING INTRALLIMINAL DEVICE, PERCUTANEOUS APPROACH 1 Cerebrosscular disease component 1 Cerebrosscular procedure 037136Z PK 10-10 OLIATON OF LETT COMMON CAROTIO ARTEN, BILLINGARD, WITH THOSE QUELLUTING INTRAL | | | | | | · |
| Cerebrovascular procedure 37/1052 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component | | | | | , | |
| Cerebrovascular procedure 037/062 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY WITH THEE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/062 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY WITH FOUR OR MORE GRUG-LUTING INTRALUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/062 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY WITH THREE INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/062 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY WITH THREE INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/062 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY WITH THREE INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/062 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY WITH FOUR OR MORE INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/1022 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY WITH FOUR OR MORE INTRALLUMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/1042 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY, BIFURCATION, WITH PRUG-ELUTING INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/1042 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY, BIFURCATION, WITH TWO DIRECE FLUTTING INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/1056 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY, BIFURCATION, WITH TWO DIRECE FLUTTING INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/1056 PX CD-10 DILATION OF LETT COMMON CARDITIO ARTERY, BIFURCATION, WITH THREE BIFURCATION, WITH THREE BIFURCATION, WITH THR | | | | | | |
| Cerebrovascular procedure 037107Z PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICE, SOPEN APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY WITH THIND INTRALUMINAL DEVICE, SOPEN APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY WITH THIND INTRALUMINAL DEVICES, OPEN APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY WITH THE INTRALLMINIAL DEVICES, OPEN APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY WITH THE INTRALLMINIAL DEVICES, OPEN APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY WITH FOUR OR MORE INTRALLMINIAL DEVICES, OPEN APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY WITH FOUR OR MORE INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY, BIFURCATION, WITH PINO PRUG-ELUTING INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY, BIFURCATION, WITH THYO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY, BIFURCATION, WITH THYO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY, BIFURCATION, WITH THYO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY, BIFURCATION, WITH THYO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY, BIFURCATION, WITH THYO DRUG ARMORE PARG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 03710FZ PX (CD-10 DILATION OF LEFT COMMON CARDIDI ARTERY, BIFURCATIO | • | | | | | · |
| Cerebrovascular procedure 037100Z PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY WITH INTRALLMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 03710FZ PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY WITH THE INTRALLMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037106Z PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY WITH THE INTRALLMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 037106Z PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY WITH THE INTRALLMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 0371346 PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY, OPEN APPROACH Cerebrovascular disease component Cerebrovascular procedure 0371345 PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALLMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 0371345 PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY, BIFURCATION, WITH THE DRUG-ELUTING INTRALLMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 0371365 PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY, BIFURCATION, WITH THE DRUG-ELUTING INTRALLMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 0371366 PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY, BIFURCATION, WITH THE DRUG-ELUTING INTRALLMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 0371367 PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY, BIFURCATION, WITH THE DRUG-ELUTING INTRALLMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 0371367 PX CD-10 DILATION OF LEFT COMMON CARDID ARTERY, BIFURCATION, WITH FINAL DIVINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component | | | | | · | |
| Cerebrovascular procedure 037/05Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH TWO INTRALLMINIAL DEVICES, OPEN APPROACH Cerebrovascular procedure 037/05Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH THOU INTRALLMINIAL DEVICES, OPEN APPROACH Cerebrovascular procedure 037/05Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH THOU ROR MORE INTRALLMINIAL DEVICES, OPEN APPROACH Cerebrovascular procedure 037/05Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THOU ROR LEVEL, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH THREE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH THREE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/14Z PX ICD-10 DIATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLMINIAL DEVICES, PERCUTANEOUS APPROAC | | | | | · | |
| Cerebrovascular procedure 037/06Z PX CD-10 DILATION OF LETF COMMON CAROTID ARTERY WITH THEE INTRALLMINAL DEVICES, OPEN APPROACH Cerebrovascular disease component | | | | | | |
| Cerebrovascular procedure Cerebrovascular pr | • | | | | | · |
| Cerebrovascular procedure O37/346 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, DEPA APPROACH Cerebrovascular procedure O37/342 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37/342 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37/355 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular drocedure O37/356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THEE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THEE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THEE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/3576 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/3577 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/3506 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/3516 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/3526 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37/3526 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH THE DRUG TRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular | · | | | | | |
| Cerebrovascular procedure O371346 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O371356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371357 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371366 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371367 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371377 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371377 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371377 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A Cerebrovascular disease component Cerebrovascular procedure O371377 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713786 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO BROWN DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713786 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713786 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713786 PX ICD-10 DILATION OF LEFT COMMON CAROTI | | | | | | |
| Cerebrovascular procedure O371342 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O371355 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371366 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371366 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371376 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371376 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS A Cerebrovascular disease component Cerebrovascular procedure O371376 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371370 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O371370 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O371370 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O371370 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLMINIAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O371370 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLMINIAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O371370 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THOR INTRALLMINIAL DEVICES, PERCU | | | | | · | |
| Cerebrovascular procedure O37135C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37136C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37137C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37137Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713D6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713D6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713D6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL | | | | | | · |
| Cerebrovascular procedure O37135C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37136C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37137C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37137Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713D6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713D6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713D6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O3713B6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL | | | | | DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH | |
| Cerebrovascular procedure 037136Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371376 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, WITH FOUR OR MORDE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A Cerebrovascular disease component Cerebrovascular procedure 0371376 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, WITH FOUR OR MORDE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371376 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371370 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371382 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371382 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure 0371386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular desease component Cerebrovascular procedure 0371386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular desease component Cerebrovascular procedure 0371386 PX IC | | | | | | |
| Cerebrovascular procedure O37;376 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLUMINAL DEVICES, PERCUTANEOUS A Cerebrovascular disease component Cerebrovascular procedure O37;375 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;375 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;385 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;385 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;385 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;385 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;385 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37;386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular desease component Cerebrovascular procedure O37;386 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37;386 PX ICD-10 DILATION OF LEFT COMMON CAR | Cerebrovascular procedure | | | | | |
| Cerebrovascular procedure O37/372 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/320 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/325 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH THO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/325 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/335 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/335 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/335 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/336 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/336 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/336 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/336 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular desease component Cerebrovascular procedure O37/346 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular desease component Cerebrovascular procedure O37/346 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular desease component Cerebrovascular procedure O37/346 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION | | | | | | |
| Cerebrovascular procedure 037/3D6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH INTRALLUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular disease component Oracer of the Common Carotid ARTERY WITH INTRALLUMINAL DEVICE, PERCUTANEOUS APPROACH Cerebrovascular disease component Oracer of the Common Carotid ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Oracer of the Common Carotid ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Oracer of the Common Carotid ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Oracer of the Common Carotid ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Oracer oracer orace | | | | | | |
| Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THEE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C Cerebrovascular procedure O37/35C Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/34C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/34C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular procedure O37/34C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure O37/34C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular proced | · | | | | · | · |
| Cerebrovascular procedure 037/356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/356 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/367 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/367 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/327 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/327 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/346 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH PRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/342 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular disease component Cerebrovascular disease component Cerebrovascular dis | | | | | | |
| Cerebrovascular procedure 037/35Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Orento O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, PERCUTANEOUS APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, PERCUTANEOUS APPROACH CEREbrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O37/35F PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC CEREBROACH | • | | | | | · |
| Cerebrovascular procedure 037.13F6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.13F2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.13G2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.13G2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.13Z2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.14G4 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.14G4 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.14G4 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure 037.14G4 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular disease component Cerebrovascular disease component Cerebrovascular procedure 037.14G6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular disease compon | | | | | | |
| Cerebrovascular procedure 037/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC Cerebrovascular disease component O17/35C PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUT | • | | | | | |
| Cerebrovascular procedure 037/3G6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Orerbrovascular procedure 037/3G2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Orerbrovascular procedure 037/3Z2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Orerbrovascular procedure 037/3Z2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Orerbrovascular procedure 037/4C2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Orerbrovascular procedure 037/4C2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Orerbrovascular procedure 037/4C2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Orerbrovascular disease compo | | | | | | |
| Cerebrovascular procedure 037/3GZ PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/3Z6 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/3Z2 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, PERCUTANEOUS APPROACH Cerebrovascular procedure PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/4Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Cerebrovascular procedure 037/4S PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH CEREBRO DRUG | | | | | | |
| Cerebrovascular procedure 037/326 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, PERCUTANEOUS APPROACH Cerebrovascular disease component Orebrovascular procedure 037/327 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, PERCUTANEOUS APPROACH Cerebrovascular DILATION OF LEFT COMMON CAROTID ARTERY, PERCUTANEOUS APPROACH PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Orebrovascular procedure 037/42 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component Orebrovascular disease Component Orebrovascular disease Component O | • | | | | | · |
| Cerebrovascular procedure 037/32Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, PERCUTANEOUS APPROACH Cerebrovascular procedure 037/446 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALLUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component 037/442 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALLUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component 037/45 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALLUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component 037/45 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALLUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH 04 DEVELOPMENT OF CARDINARY OF CAR | | | | | · | |
| Cerebrovascular procedure 0371446 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPR Cerebrovascular disease component Cerebrovascular procedure 037144Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O371456 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O371456 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O371456 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O371456 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component O371456 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH CEREBRO ARTERY DRUG-ELUTING INTRALU | | | | | | |
| Cerebrovascular procedure 037144Z PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH Cerebrovascular disease component 0371456 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC Cerebrovascular disease component | | | | | | |
| Cerebrovascular procedure 0371456 PX ICD-10 DILATION OF LEFT COMMON CAROTID ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIi Cerebrovascular disease component | | | | | | · |
| | | | | | · | · |
| | • | | | | • | · |


Cerebrovascular disease component

Symptomatic peripheral artery disease component


Symptomatic peripheral artery disease component


Symptomatic peripheral artery disease component

Symptomatic peripheral artery disease component


Symptomatic peripheral artery disease component

Symptomatic peripheral artery disease component


Symptomatic peripheral artery disease component REMI' Symptomatic peripheral artery disease component

Symptomatic peripheral artery disease component


Symptomatic peripheral artery disease component


Symptomatic peripheral artery disease component


OXYGEN ACCESSORY, DC POWER ADAPTER FOR PORTABLE CONCENTRATOR, ANY TYPE, REPLACEMENT ONLY, IMMERSION EXTERNAL HEATER FOR NEBULIZER NEBULIZER PORTABLE WITH SMALL COMPRESSOR, WITH LIMITED FLOW OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV, TO 244 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV. TO 488 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV. TO 732 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV. TO 976 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV, TO 1220 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV. TO 1464 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV. TO 1708 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM FOULV, TO 1952 CU. FT. OXYGEN CONCENTRATOR, HIGH HUMIDITY SYSTEM EQUIV, TO OVER 1952 CU. FT. OXYGEN CONCENTRATOR, SINGLE DELIVERY PORT, CAPABLE OF DELIVERING 85 PERCENT OR GREATER OXYGEN CONCENTRATION AT THE PRESCRIBED FLOW RATE OXYGEN CONCENTRATOR, DUAL DELIVERY PORT, CAPABLE OF DELIVERING 85 PERCENT OR GREATER OXYGEN CONCENTRATION AT THE PRESCRIBED FLOW RATE, EACH PORTABLE OXYGEN CONCENTRATOR, RENTAL

## DURABLE MEDICAL EQUIPMENT, MISCELLANEOUS

OXYGEN CONCENTRATOR, MANUFACTURER SPECIFIED MAXIMUM FLOW RATE DOES NOT EXCEED 2 LITERS PER MINUTE, AT 85 PERCENT OR GREATER CONCENTRATION.

OXYGEN CONCENTRATOR, MANUFACTURER SPECIFIED MAXIMUM FLOW RATE GREATER THAN 2 LITERS PER MINUTE, DOES NOT EXCEED 3 LITERS PER MINUTE, AT 85 PERCENT OR GREATER CONCENTRATION OXYGEN CONCENTRATOR, MANUFACTURER SPECIFIED MAXIMUM FLOW RATE GREATER THAN 3 LITERS PER MINUTE, DOES NOT EXCEED 4 LITERS PER MINUTE, AT 85 PERCENT OR GREATER CONCENTRATION OXYGEN CONCENTRATOR, MANUFACTURER SPECIFIED MAXIMUM FLOW RATE GREATER THAN 4 LITERS PER MINUTE, DOES NOT EXCEED 5 LITERS PER MINUTE, AT 85 PERCENT OR GREATER CONCENTRATION OXYGEN CONCENTRATOR, MANUFACTURER SPECIFIED MAXIMUM FLOW RATE GREATER THAN 5 LITERS PER MINUTE, AT 85 PERCENT OR GREATER CONCENTRATION OXYGEN AND WATER VAPOR ENRICHING SYSTEM WITH HEATED DELIVERY

OXYGEN AND WATER VAPOR ENRICHING SYSTEM WITHOUT HEATED DELIVERY E1388 - not matched

MULTIPLE ENDOCRINE NEOPLASIA [MEN] TYPE IIA MULTIPLE ENDOCRINE NEOPLASIA [MEN] TYPE IIB CYTOMEGALOVIRAL PANCREATITIS IDIOPATHIC ACUTE PANCREATITIS

BILIARY ACUTE PANCREATITIS

DRUG INDUCED ACUTE PANCREATITIS

OTHER ACLITE PANCREATITIS

IDIOPATHIC ACUTE PANCREATITIS WITHOUT NECROSIS OR INFECTION IDIOPATHIC ACUTE PANCREATITIS WITH UNINFECTED NECROSIS IDIOPATHIC ACUTE PANCREATITIS WITH INFECTED NECROSIS

BILIARY ACUTE PANCREATITIS WITHOUT NECROSIS OR INFECTION BILIARY ACUTE PANCREATITIS WITH UNINFECTED NECROSIS BILIARY ACUTE PANCREATITIS WITH INFECTED NECROSIS ALCOHOL INDUCED ACUTE PANCREATITIS

ALCOHOL INDUCED ACUTE PANCREATITIS WITHOUT NECROSIS OR INFECTION ALCOHOL INDUCED ACUTE PANCREATITIS WITH UNINFECTED NECROSIS ALCOHOL INDUCED ACUTE PANCREATITIS WITH INFECTED NECROSIS

DRUG INDUCED ACUTE PANCREATITIS WITHOUT NECROSIS OR INFECTION DRUG INDUCED ACUTE PANCREATITIS WITH UNINFECTED NECROSIS DRUG INDUCED ACUTE PANCREATITIS WITH INFECTED NECROSIS

OTHER ACUTE PANCREATITIS WITHOUT NECROSIS OR INFECTION OTHER ACUTE PANCREATITIS WITH UNINFECTED NECROSIS OTHER ACUTE PANCREATITIS WITH INFECTED NECROSIS ACUTE PANCREATITIS, UNSPECIFIED

ACUTE PANCREATITIS WITHOUT NECROSIS OR INFECTION, UNSPECIFIED ACUTE PANCREATITIS WITH UNINFECTED NECROSIS, UNSPECIFIED ACUTE PANCREATITIS WITH INFECTED NECROSIS, UNSPECIFIED ALCOHOL-INDUCED CHRONIC PANCREATITIS OTHER CHRONIC PANCREATITIS

BYPASS STOMACH TO DUODENUM WITH AUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH BYPASS STOMACH TO JEJUNUM WITH AUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH BYPASS STOMACH TO ILEUM WITH AUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH

Heart failure class IV component overlap with oxygen use component

Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component

Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component

Heart failure class IV component overlap with oxygen use component

Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component Heart failure class IV component overlap with oxygen use component GLP1-RA

GLP1-RA GLP1-RA GLP1-RA

GLP1-RA GIP1-RA

GLP1-RA DPP4-is DPP4-is DPP4-is

DPP4-is DPP4-is

DPP4-is DPP4-is DPP4-is

DPP4-is DPP4-is Pramlintide


GASTRIC RESTRICTIVE PROCEDURE, WITH GASTRIC BYPASS FOR MORBID OBESITY; WITH SHORT LIMB (150 CM OR


CONTINUING PREGNANCY AFTER SPONTANEOUS ABORTION OF ONE FETUS OR MORE, FIRST TRIMESTER, NOT


PRETERM PREMATURE RUPTURE OF MEMBRANES, ONSET OF LABOR WITHIN 24 HOURS OF RUPTURE,


HUMAN IMMUNODEFICIENCY VIRUS [HIV] DISEASE COMPLICATING PREGNANCY, CHILDBIRTH AND THE


MATERNAL MALIGNANT NEOPLASMS, TRAUMATIC INJURIES AND ABUSE CLASSIFIABLE ELSEWHERE BUT


DX ICD-10

MALIGNANT NEOPLASM OF RIGHT CHOROID

C69.31

Cancer


# Flowchart for Cohort Assembly

<u>Link to Aetion reports:</u>
Date conducted:

CMS

https://bwh-dope.aetion.com/project/2153/cohort/57260/116334/comparative/basics 8/2/24

OPTUM

https://bwh-dope.aetion.com/project/1701/cohort/57259/116336/comparative/basics 8/2/24

MarketScan

https://bwh-dope.aetion.com/project/2152/cohort/57257/116333/comparative/basics 8/2/24

| | · · | Optum<br>(Sep 19, 2019 and Feb 29, 2024) | | Marketscan<br>(Sep 20, 2019 and Dec 31, 2022) | | S<br>and Dec 31,<br>D) |
|---|---|---|---|---|---|---|
| | Less Excluded Patients | Remaining<br>Patients | Less Excluded Patients | Remaining<br>Patients | Less Excluded Patients | Remaining<br>Patients |
| Patients in dataset | | 93,159,383 | | 119,592,975 | | 28,874,258 |
| Patients meeting cohort entry criteria | | | | | | |
| (Exposure: Oral Semaglutide, Reference: Sitagliptin) | | 430,611 | | 338,596 | | 598,543 |
| Excluded due to insufficient enrollment [30 days gap allowed] | | | | | | |
| (-180, 0) | -63,127 (15%) | 367,484 | -33,585 (10%) | 305,011 | -132,300 (22%) | 466,243 |
| Excluded due to prior use of referent (-180, 0) | -200,671 (55%) | 166,813 | -206,126 (68%) | 98,885 | -384,027 (82%) | 82,216 |
| Excluded due to prior use of exposure (-180, 0) | -53,951 (32%) | 112,862 | -37,763 (38%) | 61,122 | -3,606 (4%) | 78,610 |
| Excluded because patient qualified in >1 exposure category | -24 (<1%) | 112,838 | -8 (<1%) | 61,114 | -4 (<1%) | 78,606 |
| Inclusion 1- Age >=50 (0, 0) | -4,206 (4%) | 108,632 | -11,468 (19%) | 49,646 | -0 (<1%) | 78,606 |
| Inclusion 2- DM Type 2 (all available data, 0) | -2,186 (2%) | 106,446 | -1,697 (3%) | 47,949 | -280 (<1%) | 78,326 |
| Inclusion 3: Cardiac/Cerebral/PVD/Stable angina/Atherosclerosis/CKD | | | | | | |
| (all available data, 0 except for CKD -180, 0) | -23,704 (22%) | 82,742 | -17,903 (37%) | 30,046 | -13,938 (18%) | 64,388 |
| Exclusion 1: MI/Stroke/Unstable angina/TIA [inpatient] | | | | | | |
| (-60, 0) | -812 (<1%) | 81,930 | -398 (1%) | 29,648 | -993 (2%) | 63,395 |
| Exclusion 2: Heart failure class IV (-180, 0) | -185 (<1%) | | -26 (<1%) | 29,622 | -0 (<1%) | 63,395 |
| Exclusion 3: GLP1 agonists/DDP4/Pramlintide (-180, 0) | -3,422 (4%) | 78,323 | -1,234 (4%) | 28,388 | -2,630 (4%) | 60,765 |
| Exclusion 4: Semaglutide (-180, -1) | -1,721 (2%) | 76,602 | -470 (2%) | 27,918 | -352 (<1%) | 60,413 |
| Exclusion 5: History of MEN-2 (-180, 0) | -0 (<1%) | 76,602 | -0 (<1%) | 27,918 | -0 (<1%) | 60,413 |
| Exclusion 5: History of pancreatitis (-180, 0) | -182 (<1%) | 76,420 | -41 (<1%) | 27,877 | -125 (<1%) | 60,288 |
| Exclusion 6: Bariatric surgery (all available data, 0) | -196 (<1%) | | -100 (<1%) | 27,777 | -281 (<1%) | 60,007 |
| Exclusion 7: Pregnancy (-180, 0) | -3 (<1%) | | -3 (<1%) | 27,774 | -2 (<1%) | 60,005 |
| Exclusion 8: Cancer (-1825, 0) | -4,470 (6%) | | -1,461 (5%) | 26,313 | -5,721 (10%) | 54,284 |
| Exclusion 9: CKD stage 5, End-stage renal disease, dialysis or renal transplant (-180, 0) | -540 (<1%) | | -135 (<1%) | 26,178 | -530 (<1%) | 53,754 |
| Exclusion 10: Proliferative retinopathy or maculopathy (-180, 0) | -559 (<1%) | | -157 (<1%) | 26,021 | -571 (1%) | 53,183 |
| Exclusion 11: Diabetic ketoacidosis (-180, 0) | -112 (<1%) | | -36 (<1%) | 25,985 | -89 (<1%) | 53,094 |
| Exclusion 12: Nursing home (-180, 0) | -1,181 (2%) | | -65 (<1%) | 25,920 | -1,010 (2%) | 52,084 |
| Excluded based on Age missing | -0 (<1%) | | -0 (<1%) | 25,920 | -0 (<1%) | 52,084 |
| Excluded based on Gender missing | -0 (<1%) | | -0 (<1%) | 25,920 | -0 (<1%) | 52,084 |
| Patients in Exposure Group | | 17,311 | | 5,209 | | 1,745 |
| Patients in Referent Group | | 52,048 | | 20,711 | | 50,339 |
| Total Patients | | 69,359 | | 25,920 | | 52,084 |

#### Appendix 4. 1st Feasibility Assessment

#### Table of Contents

- A. Patient characteristics by treatment group
- B. Summary Parameters of Study Population
- C. Median Follow up Time in Overall Study Population
- D. Reasons for Censoring in Overall Study Population
- E. Initial Power Assessment
- F. Aetion Report Links
- G. Review by Principal Investigator and FDA

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a 1:1 PS-matched comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Phoward at (2001).

Optum: Study period between 20<sup>th</sup> Sept 2019 - 29<sup>th</sup> February 2024 Marketscan: Study period between 20<sup>th</sup> Sept 2019 - 31<sup>st</sup> Dec 2022 Medicare: Study period between 20<sup>th</sup> Sept 2019 - 31<sup>st</sup> Dec 2020

#### A. Patient characteristics by treatment group (we start 1 days after CED, so we drop few patients and hence table 1 number of patients are little different than the attrition table)

| UNMATCHED | | Optum | | Marketscan | | | Medicare | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | | Exposure - Semagiutide<br>oral | Difference | Reference- Sitagliptin | Exposure - Semaglutide<br>oral | Difference | Reference- Sitagliptin | Exposure - Semaglutide<br>oral | Difference |
| Number of patients | 51,947 | 17,273 | - (-, -) | 20,669 | 5,203 | - (-, -) | 50,218 | 1,740 | - (-, -) |
| Age | | | | | | | | | |
| mean (sd) | 73.39 (7.96) | 69.02 (8.24) | 4.37 (4.23, 4.51) | 67.24 (10.47) | 61.93 (8.13) | 5.31 (5.05, 5.58) | 76.10 (6.87) | 73.60 (5.82) | 2.51 (2.23, 2.79) |
| median [IQR] | 73.00 [68.00, 79.00] | 69.00 [64.00, 75.00] | - (-, -) | 65.00 [59.00, 75.00] | 61.00 [56.00, 65.00] | - (-, -) | 75.00 [71.00, 81.00] | 73.00 [69.00, 77.00] | - (-, -) |
| Gender without unknown | | | | | | | | | |
| Male; n (%) | 24,695 (47.5%) | 8,619 (49.9%) | -2.4% (-3.2%, -1.5%) | 11,625 (56.2%) | 2,956 (56.8%) | -0.6% (-2.1%, 0.9%) | 23,883 (47.6%) | 874 (50.2%) | -2.7% (-5.1%, -0.3%) |
| Female; n (%) | 27,251 (52.5%) | 8,652 (50.1%) | 2.4% (1.5%, 3.2%) | 9,044 (43.8%) | 2,247 (43.2%) | 0.6% (-0.9%, 2.1%) | 26,335 (52.4%) | 866 (49.8%) | 2.7% (0.3%, 5.1%) |
| Uknown; n (%) | 1 (0.0%) | 2 (0.0%) | -0.0% (-0.0%, 0.0%) | | | | | | |
| CCI (180 days)- ICD9 and<br>ICD10 | | | | | | | | | |
| mean (sd) | 2.24 (2.37) | 1.75 (2.05) | 0.49 (0.45, 0.52) | 1.49 (2.09) | 1.04 (1.68) | 0.45 (0.40, 0.51) | 1.82 (2.16) | 1.66 (1.92) | 0.16 (0.06, 0.25) |
| median [IQR] | 2.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |

#### B. Summary Parameters of Overall Study Population (Step 1)

| UNMATCHED | Optum | Marketscan | Medicare |
|---|---|---|---|
| Variable | Value | Value | Value |
| Number of patients in<br>full cohort | 69,359 | 25,920 | 52,084 |
| Number of patients<br>dropped as incomplete<br>cases | 0 | 0 | 0 |
| Number of patients that did not begin follow-up | 139 | 48 | 126 |
| Number of patients in<br>analytic cohort | 69,220 | 25,872 | 51,958 |
| Number of events | 1,781 | 441 | 1520 |
| Number of person-<br>years | 32,140.18 | 11,971.28 | 21,016.00 |
| Number of patients in<br>group: Sitagliptin | 51,947 | 20,669 | 50,218 |
| Number of patients in<br>group: Semaglutide -<br>oral | 17,273 | 5,203 | 1,740 |
| Risk per 1,000 patients | 25.73 | 17.05 | 29.25 |
| Rate per 1,000 person-<br>years | 55.41 | 36.84 | 72.33 |

# C. Median Follow up Time in Overall Study Population (Step 1)

| UNMATCHED | Optum | Marketscan | Medicare |
|---|---|---|---|
| Patient Group | | | Median Follow-Up<br>Time (Days) [IQR] |
| Overall Patient Population | 118 [59, 263] | 118 [58, 279] | 118 [58, 210] |

#### D. Reasons for Censoring in Overall Study Population (Step 1)

| UNMATCHED | Optum | Marketscan | Medicare |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 1,781 (2.6%) | 441 (1.7%) | 1,520 (2.9%) |
| Start of an additional<br>exposure | 528 (0.8%) | 229 (0.9%) | 101 (0.2%) |
| End of index exposure (30 days risk, grace windows) | 37,256 (53.8%) | 12,296 (47.5%) | 20,691 (39.8%) |
| Maximum follow-up time<br>(365 days) | 11,410 (16.5%) | 4,538 (17.5%) | 3,304 (6.4%) |

| Specified date reached | 7,850 (11.3%) | 3,579 (13.8%) | 22,377 (43.1%) |
|---|---|---|---|
| End of patient enrollment | 5,067 (7.3%) | 3,507 (13.6%) | 1,398 (2.7%) |
| Nursing home<br>admission/Other GLP1<br>(including inj.Semaglutide) | 5,328 (7.7%) | 1,282 (5.0%) | 2,567 (4.9%) |

| Fine stratification | Optum | Marketscan | Medicare |
|---------------------|--------|------------|----------|
| Exposure | 17,273 | 5,203 | 1,740 |
| Reference | 46,752 | 18,602 | 45,196 |

| Matched number | Optum | Marketscan | Medicare |
|----------------|--------|------------|----------|
| Exposure | 16,277 | 5,203 | 1,740 |
| Reference | 16,277 | 5,203 | 1,740 |

#### E. Initial Power Assessment

Based on 1:1 randomization and assuming an annulized placebo MACE rate of 3.5%, a true HR of 0.83, it was determinded that total

| Superiority Analys | is (fine strati) |
|---------------------------|------------------|
| Number of patients | |
| matched | |
| Reference | 110,551 |
| Exposed | 24,216 |
| Risk per 1,000 patients | 25.45 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 3429.4 |
| Power | 1.0 |

| Superiority | Analysis (1:1) |
|------------------------------|----------------|
| Number of patients | 1 |
| matched | |
| Reference | 23,220 |
| Exposed | 23,220 |
| Risk per 1,000<br>patients | 25.45 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events<br>expected | 1181.8 |
| Power | 0.9 |

#### F. Aetion Report Links

### Aetion report link:

For Semaglutide vs Sitagliptin cohort

Optum
Step 1: https://bwh-dope.aetion.com/project/1701/rwrs/123631 Step 2: https://bwh-dope.aetion.com/project/1701/rwrs/123632

Marketscan
Step 1: https://bwh-dope.aetion.com/project/2152/rwrs/123617
Step 2: https://bwh-dope.aetion.com/project/2152/rwrs/123618

Medicare
Step 1: https://bwh-dope.aetion.com/project/2153/rwrs/123624 Step 2: https://bwh-dope.aetion.com/project/2153/rwrs/123625

#### G. Review by principal investigator and FDA

Stop analyses until feasibility and power are reviewed by primary investigators and FDA.

| First review by FDA | Date reviewed: | 30th Sept 2024 |
|-----------------------|----------------|------------------|
| Final review and | | |
| approval by FDA after | Date reviewed: | 3rd October 2024 |
| comments were | Date reviewed. | 310 October 2024 |
| addressed | | |

# Appendix 5. 2nd Feasibility Assessment

# **Table of Contents**

- A. Median Follow up Time by Treatment Group
- B. Reasons for Censoring by Treatment Group
- C. Final Power Assessment
- D. Aetion report Links
- E. Review by Principal Investigator and FDA

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a 1:1 PS-matched comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the formulas from Chow et al. (2008).

# A. Median Follow Up Time by Treatment Group (Step 1)

| UNMATCHED | Optum | Marketscan | Medicare |
|---|---|---|---|
| Patient Group | | Median Follow-Up | Median Follow-<br>Up Time (Days)<br>[IQR] |
| Overall Patient<br>Population | 118 [59, 263] | 118 [58, 279] | 118 [58, 210] |

# B. Summary Parameters of Overall Study Population (Step 1)

| UNMATCHED Optum | | Marketscan | Medicare |
|---|---|---|---|
| Variable | Value | Value | Value |
| Number of patients in full cohort | 69,359 | 25,920 | 52,084 |
| Number of patients dropped as incomplete cases | 0 | 0 | 0 |
| Number of patients<br>that did not begin<br>follow-up | 139 | 48 | 126 |
| Number of patients in analytic cohort | 69,220 | 25,872 | 51,958 |
| Number of events | 2,031 | 441 | 1520 |
| Number of person-<br>years | 32,944.78 | 11,971.28 | 21,016.00 |
| Number of patients in group:<br>Sitagliptin | 51,947 | 20,669 | 50,218 |
| Number of patients<br>in group:<br>Semaglutide - oral | 17,273 | 5,203 | 1,740 |
| Risk per 1,000 patients | 29.34 | 17.05 | 29.25 |
| Rate per 1,000 person-years | 61.65 | 36.84 | 72.33 |

C. Reasons for Censoring in Overall Study Population (Step 1)

| UNMATCHED | Optum | Marketscan | Medicare |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 1,781 (2.6%) | 441 (1.7%) | 1,520 (2.9%) |
| Start of an additional exposure | 528 (0.8%) | 229 (0.9%) | 101 (0.2%) |
| End of index exposure<br>(30 days risk, grace<br>windows) | 37,256 (53.8%) | 12,296 (47.5%) | 20,691<br>(39.8%) |
| Maximum follow-up time (365 days) | 11,410 (16.5%) | 4,538 (17.5%) | 3,304 (6.4%) |
| Specified date<br>reached | 7,850 (11.3%) | 3,579 (13.8%) | 22,377<br>(43.1%) |
| End of patient enrollment | 5,067 (7.3%) | 3,507 (13.6%) | 1,398 (2.7%) |
| Nursing home<br>admission/Other<br>GLP1 (including<br>inj.Semaglutide) | 5,328 (7.7%) | 1,282 (5.0%) | 2,567 (4.9%) |

# D. Final Power Assessment (Step 3)

Based on 1:1 randomization and assuming an annulized placebo MACE rate of 3.5%, a true HR of 0.83, it was determinded that total of 1225 first MACEs are required to confirm superiority with primary outcome of 90% power using a 1 sided type 1 error rate of 0.025

calculate\_ess <- function(weights) {
 sum(weights)^2 / sum(weights^2)}
ess\_treatment\_1 <- calculate\_ess(soul\_fs\$psweight[soul\_fs\$Treatment == 1])
ess\_treatment\_0 <- calculate\_ess(soul\_fs\$psweight[soul\_fs\$Treatment == 0])</pre>

#### <u>OPTUM</u>

ESS for Reference: 18,708.86 ESS for Exposure: 17,239

# MARKETSCAN-

ESS for Reference: 8,452.76 ESS for Exposure: 5,189

Numbers below are based on the PS assessed based on all the covariates given in the Balance - Table 1 sheet

118262

24165

| Superiority Analysis (fine strati) | |
|------------------------------------|---------|
| Number of patients | |
| matched | |
| Reference | 118,262 |
| Exposed | 24,165 |
| Risk per 1,000 patients | 27.15 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events<br>expected | 3866.5 |
| Power | 1.0 |

| Superiority | Superiority Analysis (1:1) |
|---------------------|----------------------------|
| Number of patients | |
| matched | |
| Reference | 21,902 |
| Exposed | 21,902 |
| Risk per 1,000 | |
| patients | 27.15 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events | 1189.2 |
| expected | 1100.2 |
| Power | 0.9 |

21902 21902

### E. Aetion Report Links

# Aetion report link:

· For Semaglutide vs Sitagliptin cohort

# <u>Optum</u>

Step 1: https://bwh-dope.aetion.com/project/1701/rwrs/116788

Step 3: https://bwh-dope.aetion.com/project/1701/rwrs/123633

#### Marketscan

Step 1: https://bwh-dope.aetion.com/project/2152/rwrs/123617

Step 3: https://bwh-dope.aetion.com/project/2152/rwrs/123619

# <u>Medicare</u>

Step 1: https://bwh-dope.aetion.com/project/2153/rwrs/123624

Step 3: https://bwh-dope.aetion.com/project/2153/rwrs/123626

# F. Review by Principal Investigator and FDA

Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| First review by FDA | Date reviewed: | 30th Sept 2024 |
|---|---|---|
| Final review and<br>approval by FDA<br>after comments<br>were addressed | Date reviewed: | 3rd October 2024 |
| Reason for stopping (if required): | | |

# OPTUM MARKETSCAN MEDICARE unadjusted cstats, Optum: 0.79899 unadjusted cstats, Marketscan: 0.79016 unadjusted cstats, Medicare: 0.85518 PS distribution: Unadjusted Cohort PS distribution: Unadjusted Cohort 1:1 matching cstats, Optum: 0.49949 1:1 matching cstats, Marketscan: 0.49974

0.4 Propensity Score



Exposure

Stagistin (networks)

Semaglishis Onli (orpicum)

# fine-stratified cstats, Optum: 0.50022







| Summary, PS distribution, Unadjusted cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN | MARKETSCAN Minimum Maximum Mean Median 25th pct 75th pct | | | | | |
| Reference | 2.58E-05 | 0.848 | 0.166 | 0.12 | 0.0477 | 0.245 |
| Exposure | 0.00532 | 0.895 | 0.341 | 0.325 | 0.205 | 0.463 |

| Summary, PS distribution, 1:1 matched cohort | | | | | | |
|---|---|---|---|---|---|---|
| OPTUM | OPTUM Minimum Maximum Mean Median 25th pct 75th pct | | | | | |
| Reference | 0.00111 | 0.91 | 0.371 | 0.365 | 0.239 | 0.489 |
| Exposure | 0.00111 | 0.912 | 0.371 | 0.365 | 0.239 | 0.49 |

OPTUM Minimum Maximum Mean Median 25th pct 75th pct

0.154 0.0569 0.296 0.397 0.256 0.549

 Reference
 2.44E-05
 0.964
 0.196

 Exposure
 0.00111
 0.95
 0.409

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| OPTUM | Minimum Maximum Mean Median 25th pct 75th pct | | | | | |
| Reference | 0.0785 | 11.7 | 1 | 0.609 | 0.0785 | 1.36 |
| Exposure | 1 | 1 | 1 | 1 | 1 | 1 |

| Summary, PS distribution, 1:1 matched cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN Minimum Maximum Mean Median 25th pct 75th pct | | | | | | |
| Reference | 0.00531 | 0.848 | 0.326 | 0.314 | 0.198 | 0.44 |
| Exposure | 0.00532 | 0.848 | 0.326 | 0.314 | 0.198 | 0.44 |
| | • | • | • | • | • | |

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN Minimum Maximum Mean Median 25th pct 75th pc | | | | | | |
| Reference | 0.0737 | 7.82 | 1 | 0.547 | 0.0737 | 1.43 |
| Exposure | 1 | 1 | 1 | 1 | 1 | 1 |

# fine-stratified cstats, Medicare: 0.5



| Summary, PS distribution, Unadjusted cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE | MEDICARE Minimum Maximum Mean Median 25th pct 75th pct | | | | | |
| Reference | 2.72E-05 | 0.76 | 0.0306 | 0.01 | 0.00274 | 0.0376 |
| Exposure | 0.000506 | 0.713 | 0.119 | 0.0906 | 0.0481 | 0.162 |

| Summary, PS distribution, 1:1 matched cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE Minimum Maximum Mean Median 25th pct 75th pct | | | | | | |
| Reference | 0.000506 | 0.477 | 0.11 | 0.0885 | 0.0469 | 0.156 |
| Exposure 0.000506 0.477 0.11 0.0885 0.0469 0.15 | | | | | | |

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.0545 | 17.9 | 1 | 0.357 | 0.0545 | 1.1 |
| Exposure | 1 | 1 | 1 | 1 | 1 | 1 |

| Variable | Octu<br>Sitagliptin - reference | m: Unadusted cohort semagluide - sapoure Sid diff 17,260 60.01 (8,24) 60.01 (8,01) 60.01 (8,01) 60.01 (8,01) 60.01 (8,01) 60.01 (8,01) | Os<br>Sitagliptin - refer | stem 14 matched cobort secs Semiglatife - seporum Sid dill 15,184 68.86 (7.80) 0.051 773.180.8 0.001 1409 (9.5) 0.001 | Octum: Fin<br>Situgliptin - reference | e stratification cohert Semaglatide - exposure 57,239 10.01 (8.24) 10.035 1633.0 (50.1) 10.005 | Markets Stagliptin - reference | an: Unadjusted cohort Semaglutide - exposure | Sed diff | Marketscan-1:1 matched cohert Sitagliptin - reference Semaglatide - exposure Std delf | Markets<br>Stagliptin - refere | can: Fine stratification cohort<br>nce Semaglutide - exposure Std dff | Medicare: Unadiusted cohort Sitsgliptin - reference Semaglutide - exposure 1 | isd diff | Medicare: 1:1 matched cohort Sitagliptin - reference Semaglutide - exposure Std diff | Medicare: Fine stratification cohort Stagliptin - reference Semaglatide - exposure Std dfff |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of patients Age mean (sd) | 73.39 (7.96) | 17,240<br>69.01 (E.24) 0.54 | 70.12 (7.55) | 15,184<br>69.98 (7.90) 0.017 | 49,959<br>69.30 (7.82) | 17,239<br>59.01 (8.24) 0.035 | 20,612<br>67.27 (10.46) | at: Unadvated cohort Semaglutide - exposure 5,197 51.94 (8.13) 2244 (43.2) 821 (15.8) | 0.569 | 4951 4951<br>62.22 (8.44) 62.19 (8.17) 0.004 | 20,279<br>61.96 (8.38) | Cart: Pire systemiciation context nece Semaglutide - exposure Std diff 5,189 61.94 (8.12) 0.001 2228.0 (4.11) 0.001 | Medicare Unablashed cohort Stagiljetin - reference Samaglatide - exposure 1 20,007 28,30 (6.87) 72,00 (5.82) 20224 (52.4) 806 (40.8) 20224 (52.4) 2 | 0.294 | 73.53 (6.02) 73.69 (5.83) 0.028 | 73.60 (5.93) 73.60 (5.82) 0.001 |
| Female; n (%) Region | 27227 (52.5) | 8634 (50.1) 0.048<br>0.122 | 7723 (50.9) | 7713 (50.8) 0.001<br>0.01 | 25347.8 (50.7) | 8633.0 (50.1) 0.013<br>0.005 | 9015 (41.7) | 2244 (43.2) | 0.011 | 2166 (43.7) 2110 (43.0) 0.015<br>0.019 | 8738.8 (43.1) | 2238.0 (43.1) 0.001<br>0.019 | 26224 (52.4) 866 (49.8) | 0.052 | 845 (50.1) 845 (50.0) 0.001<br>0.022 | 23999.1 (50.0) 865.0 (49.8) 0.003<br>0.011 |
| Midwest n (%) West n (%) West n (%) | 7588 (14.6)<br>28416 (54.8)<br>9280 (17.9) | 2004 (16.0)<br>2024 (16.0)<br>2021 (57.0)<br>2924 (16.9) | 2481 (16.3)<br>8562 (56.4)<br>2659 (17.5) | 2499 (16.4)<br>2499 (16.4)<br>8593 (56.6)<br>2693 (17.1) | 4681.7 (9.4)<br>8300.7 (16.6)<br>28463.4 (57.0)<br>8513.2 (17.0) | 1984.0 (16.9)<br>19820.0 (57.0)<br>2914.0 (16.9) | 8407 (31.1)<br>8443 (41.0) | 1107 (21.3)<br>2836 (54.6) | | 1118 (22.6) 1091 (22.0)<br>2649 (53.5) 2650 (53.5)<br>380 (7.7) | 4421.9 (21.8)<br>10947.1 (54.0)<br>1624.5 (8.0) | 1107.0(21.3)<br>2128.0(54.5)<br>433.0(8.3) | 10654 (21.3) 320 (18.4)<br>9418 (18.8) 276 (15.9)<br>21076 (42.3) 767 (44.1)<br>8909 (17.8) 376 (21.6) | | 261 (25.6) 273 (56.2)<br>760 (43.8) 746 (44.3)<br>369 (21.8) 363 (21.5) | 7704.8 (16.0) 276.0 (15.9)<br>21089.8 (43.9) 767.0 (44.2)<br>10510.3 (21.5) 374.0 (23.5) |
| Year of cohort entry 2019 (Sept-Dec); n (%) 2020 (Inp.March); n (%) | 3771 (7.3) | 1001 (0.4)<br>2094 (16.8)<br>9821 (57.0)<br>2014 (16.9)<br>0.809<br>6 (0.0)<br>120 (0.7)<br>243 (1.4) | 7 (0.0) | 6 (0.0)<br>170 (0.0) | 144.3 (0.3) | 0.07<br>5.0 (0.0) | 2678 (13.0) | 71 (1.4) | 0.709 | 380 (7.7) 401 (8.1) 0.041<br>61 (1.2) 71 (1.4) 0.041 | 238.5 (1.2) | 71.0(1.4) | 11976 (23.9) 20 (1.2)<br>11387 (22.7) 102 (6.2) | 1.244 | 14 (0.8) 20 (1.2)<br>103 (5.1) 107 (6.3) | 610.5 (1.3) 19.0 (1.1)<br>2699.4 (5.6) 107.0 (6.2) |
| 2020 (April-June); n (%)<br>2020 (April-June); n (%)<br>2020 (April-June); n (%) | 3331 (6.4)<br>3387 (6.5) | 243 (1.4)<br>403 (2.3)<br>616 (3.6) | 223 (1.5)<br>364 (2.4)<br>598 (1.6) | 241 (1.6)<br>296 (2.6)<br>555 (1.9) | 144.3 (0.3)<br>395.4 (0.8)<br>599.1 (1.2)<br>1045.9 (2.1)<br>1720.9 (3.4)<br>8072.6 (19.8)<br>13254.0 (26.5) | 243.0 (1.4)<br>43.0 (2.3)<br>516.0 (2.6) | 1670 (8.1)<br>1969 (9.6)<br>1869 (9.1) | 203 (3.9)<br>300 (5.8)<br>417 (8.0) | | 285 (3.7) 203 (4.1)<br>298 (6.0) 298 (6.0)<br>439 (6.0) 414 (8.4) | 756.6 (3.7)<br>1141.5 (5.6)<br>1635.0 (8.1) | 166.0 (1.2)<br>201.0 (1.9)<br>300.0 (5.8) | 8729 (17.4) 127 (7.3)<br>9468 (18.9) 606 (34.8)<br>8697 (17.0) 879 (50.5) | | 117 (6.9) 127 (7.5)<br>604 (35.7) 592 (35.0)<br>872 (30.4) 844 (49.9) | 3388.9 (7.1) 127.0 (7.3)<br>16994.6 (15.4) 606.0 (34.9)<br>24340.6 (50.7) 878.0 (50.5) |
| 2021 (Jan-Dec); n (%)<br>2022 (Jan-Dec); n (%)<br>2023 (Jan-Dec); n (%) | 12357 (23.8)<br>10103 (19.5)<br>9763 (18.8) | 3417 (19.9)<br>4585 (26.6)<br>6664 (38.7) | 3236 (21.3)<br>4142 (27.3)<br>5483 (36.1) | 3261 (21.5)<br>4083 (26.9)<br>5479 (36.1) | 9872.6 (19.8)<br>13254.0 (26.5)<br>19518 5 (30.1) | 1437.0 (19.9)<br>1685.0 (26.6) | 5836 (28.3)<br>4536 (22.0) | 1875 (36.1)<br>2164 (41.6) | | 1873 (37.8) 1815 (36.7)<br>1938 (39.1) 1983 (40.1) | 7564.7 (37.3)<br>8335.4 (41.1) | 417.0 (8.0)<br>1874.0 (36.1)<br>2158.0 (41.6) | | | 33,133,1 | |
| 2024 (Jan - Feb); n (%) Drug Jahuse or dependence; n (%) Minobal share or dependence: n (%) | 1967 (3.8)<br>1178 (2.3)<br>654 (1.3) | 1166 (6.8)<br>392 (2.3) 0.001 | 1023 (6.7)<br>336 (2.2)<br>179 (1.2) | 505 (3.9) | 19518.5 (19.1)<br>2408.4 (6.8)<br>1115.2 (2.2)<br>583.1 (1.7) | 1166.0 (6.8)<br>192.0 (2.3)<br>192.0 (2.3)<br>194.0 (1.1)<br>1048.0 (2.0)<br>105.0 (1.3) | 219 (1.1) | 41 (D.E)<br>36 (D.7) | 6.00<br>6.000<br>6.0000<br>6.000<br>6.0000<br>6.00 | 41 (0.9) 41 (0.8) 0.004<br>30 (0.8) 35 (0.7) 0.009 | 160.4 (0.8) | 41.0 (0.8) 0.001 | 414 (0.8) 18 (1.0)<br>218 (0.6) 7.02 41 | 0.022 | 18 (1.1) 16 (0.9) 0.012<br>10 (0.6) 7 (0.4) 0.025 | 501.8(1.0) 18.0(1.0) 0.000<br>198.5(0.4) 7.0(0.4) 0.002 |
| Underweight or normal weight; n (%) Overweight; n (%) Obese: n (%) | 2196 (4.2)<br>5303 (10.2)<br>7184 (13.8) | 348 (2.0) 0.127<br>1601 (9.3) 0.031<br>3301 (19.1) 0.143 | 359 (2.4)<br>1465 (9.6)<br>2692 (17.7) | 343 (2.3) 0.007<br>3453 (9.6) 0.003<br>2720 (37.9) 0.005 | 1057.0 (2.1)<br>4712.7 (9.4)<br>9626.6 (19.1) | 148.0 (2.0) 0.007<br>1601.0 (9.3) 0.005<br>1301.0 (19.1) 0.003 | 469 (2.3)<br>1537 (7.5)<br>1812 (8.8) | 47 (0.9)<br>318 (6.1)<br>595 (11.4) | 0.11<br>0.053<br>0.088 | 43 (0.9) 46 (0.9) 0.006<br>302 (6.1) 308 (6.2) 0.005<br>543 (31.0) 553 (31.2) 0.006 | 189.5 (0.9)<br>1263.1 (6.2)<br>2310.5 (11.4) | 36.0(0.7) 0.001<br>47.0(0.9) 0.001<br>318.0 (6.1) 0.004<br>592.0 (11.4) 0.001<br>865.0 (16.7) 0.02<br>999.0 (18.1) 0.012 | 21E (0.6) 7 (0.4)<br>2155 (4.4) 29 (1.7)<br>5643 (11.3) 171 (9.8)<br>7574 (15.1) 325 (1E.7) | 0.159<br>0.047<br>0.095 | 19 (1.1) 29 (1.7) 0.05<br>166 (9.1) 166 (9.8) 0.001<br>314 (18.6) 317 (18.8) 0.005<br>251 (14.9) 259 (15.3) 0.013 | 798.5 (1.7) 28.0 (1.6) 0.001<br>4695.1 (9.8) 170.0 (9.8) 0.001<br>8874.2 (18.5) 325.0 (18.7) 0.006 |
| Severe obess; n (%) Unspecified obesity; n (%) Smokins: n (%) | 5049 (9.7)<br>5557 (10.7)<br>8852 (17.1) | 3324 (19.3) 0.274<br>3018 (17.5) 0.166<br>2948 (17.1) 0.001 | 2429 (16.0)<br>2290 (15.1)<br>2598 (17.1) | 2504 (16.5) 0.001<br>2336 (15.4) 0.008<br>2595 (17.1) 0.001 | 9422.7 (18.9)<br>8614.1 (17.2)<br>8738.6 (17.5) | 1324.0 (19.3) 0.011<br>3018.0 (17.5) 0.007<br>2947.0 (17.1) 0.01 | 2021 (9.8)<br>2484 (12.1)<br>1800 (8.7) | 868 (16.7)<br>942 (18.1)<br>398 (7.7) | 0.204<br>0.17<br>0.039 | 764 (15.4) 785 (15.9) 0.012<br>874 (17.7) 865 (17.5) 0.005<br>382 (7.7) 350 (7.9) 0.006 | 3229.5 (15.9)<br>3579.2 (17.7)<br>1582.7 (7.8) | 865.0 (16.7) 0.02<br>939.0 (18.1) 0.012<br>397.0 (7.7) 0.006 | 4235 (8.5) 274 (15.8)<br>8797 (13.6) 354 (20.4)<br>7216 (14.4) 230 (13.2) | 0.047<br>0.095<br>0.225<br>0.181<br>0.034 | 251 (14.9) 259 (15.3) 0.011<br>341 (20.2) 319 (20.1) 0.001<br>219 (13.0) 227 (13.4) 0.014 | 7401.5 (15.4) 273.0 (15.7) 0.008<br>8649.8 (20.1) 353.0 (20.3) 0.006<br>6368.7 (13.3) 230.0 (13.2) 0.001 |
| Diabetic retinopathy; n (%) Diabetic neuropathy; n (%) Diabetic nechropathy; n (%) | 4533 (8.7)<br>14389 (27.7)<br>14389 (27.7) | 1371 (8.0) 0.038<br>4388 (25.5) 0.051<br>4388 (25.5) 0.051 | 1298 (8.5)<br>4030 (26.5)<br>4030 (26.5) | 1230 (8.1) 0.016<br>3950 (26.0) 0.02<br>3950 (26.0) 0.02 | 4131.0 (8.3)<br>13246.4 (26.5)<br>13246.4 (26.5) | 1371.0 (8.0) 0.012<br>4388.0 (25.5) 0.024<br>4388.0 (25.5) 0.024<br>1452.0 (20.0) 0.003<br>523.0 (3.6) 0.005 | 1296 (6.3)<br>4214 (20.4)<br>4215 (20.4) | 232 (4.5)<br>871 (16.8)<br>871 (16.8) | 0.081 | 228 (4.5) 224 (4.5) 0.004<br>869 (17.6) 833 (16.8) 0.019<br>869 (17.6) 833 (16.8) 0.019 | 928.4 (4.6)<br>3439.3 (17.0)<br>3439.3 (17.0) | 212.0 (4.5) 0.005<br>867.0 (16.7) 0.007<br>867.0 (16.7) 0.007 | 3366 (6.8) 108 (6.2)<br>9918 (19.8) 369 (21.2)<br>9918 (19.8) 369 (21.2) | 0.023<br>0.035<br>0.035 | 104 (6.2) 108 (6.4) 0.01<br>153 (20.9) 357 (21.1) 0.006<br>153 (20.9) 357 (21.1) 0.006 | 2993.9 (6.2) 108.0 (6.2) 0.001<br>10116.8 (21.1) 368.0 (21.2) 0.003<br>10116.8 (21.1) 368.0 (21.2) 0.003 |
| Diabetes with unspecified complications; n (%) Diabetes with other ophthalmic complications; n (%) Diabetes with peripheral circulatory disorders; n (%) | 2284 (4.4)<br>9029 (17.4) | 4388 (25.5) 0.051<br>4388 (25.5) 0.051<br>3453 (20.0) 0.007<br>623 (3.6) 0.04<br>3621 (15.2) 0.059 | 3057 (20.2)<br>621 (4.1)<br>2417 (15.9) | 1220 (E.1) 0.016<br>3950 (26.0) 0.012<br>3950 (26.0) 0.012<br>3055 (19.9) 0.007<br>578 (1.8) 0.015<br>2254 (15.5) 0.011 | 10064.4 (20.1)<br>1856.1 (3.7)<br>7739.2 (15.5) | 4388.0 (25.5) 0.024<br>1452.0 (20.0) 0.003<br>523.0 (3.6) 0.005<br>2620.0 (35.2) 0.008 | 2283 (11.1)<br>303 (1.5)<br>2026 (9.8) | 689 (13.3)<br>69 (1.3)<br>451 (8.7) | 0.067<br>0.012<br>0.04 | 869 (17.6) 833 (16.8) 0.039<br>633 (17.8) 645 (13.0) 0.007<br>51 (10) 63 (1.3) 0.023<br>405 (8.2) 427 (8.6) 0.016 | 2652.6 (13.1)<br>248.3 (1.2)<br>1707.4 (8.4) | 232.0 (4.5) 0.005<br>867.0 (16.7) 0.007<br>867.0 (16.7) 0.007<br>689.0 (13.3) 0.005<br>69.0 (13.3) 0.009<br>450.0 (8.7) 0.009 | 4061 (8.1) 160 (9.2)<br>893 (1.4) 28 (1.6)<br>4637 (9.3) 156 (9.0) | 0.019 | 255 (26.5) 257 (26.5) 0.023<br>25 (2.5) 27 (1.6) 0.01<br>164 (9.7) 353 (9.1) 0.022 | 4404.0 (9.2) 160.0 (9.2) 0.000<br>780.5 (1.6) 28.0 (1.6) 0.000<br>4112.0 (9.0) 156.0 (9.0) 0.000 |
| Diabetic foot + Lower extremity amputation; n (%) Skin infections; n (%) Exectle dysfunction; n (%) | 1257 (2.4)<br>2844 (5.5)<br>1235 (2.4) | 340 (2.0) 0.031<br>997 (5.8) 0.013<br>611 (3.5) 0.069 | 291 (1.9)<br>812 (5.3)<br>467 (3.1) | 301 (2.0) 0.005<br>841 (5.6) 0.009<br>440 (1.2) 0.005<br>2976 (19.6) 0.008<br>6591 (43.4) 0.001<br>11009 (8.7) 0.005<br>11957 (78.7) 0.005 | 1019.2 (2.0)<br>2907.2 (5.8)<br>1658.3 (3.3) | 339.0 (2.0) 0.005<br>997.0 (5.8) 0.002<br>511.0 (3.5) 0.012 | 298 (1.9)<br>1180 (5.7)<br>482 (2.3) | 85 (1.6)<br>282 (5.4)<br>150 (2.9) | 0.022<br>0.013<br>0.034 | 87 (1.8) 84 (1.7) 0.005<br>262 (5.3) 264 (5.3) 0.002 | 364.4 (1.8)<br>1084.7 (5.3)<br>580.2 (2.9) | 85.0 (1.6) 0.012 | 873 (1.7) 32 (1.8) | 0.007<br>0.035<br>0.054 | 27 (2.6) 32 (1.9) 0.023<br>107 (6.3) 110 (6.5) 0.007 | 876.7(1.8) 32.0(1.8) 0.001<br>3148.1(6.6) 112.0(6.5) 0.002<br>599.3(1.2) 23.0(1.3) 0.007 |
| Hypoglycemia; n (%)<br>Hyperglycemia, DKA, HONK; n (%)<br>Hypertension; n (%) | 10304 (19.9)<br>20986 (40.4)<br>44364 (85.5) | 3377 (19.6) 0.007<br>7589 (44.0) 0.073<br>14780 (85.7) 0.007 | 3022 (19.9)<br>6600 (43.5)<br>13087 (86.2) | 2976 (19.6) 0.008<br>6591 (43.4) 0.001<br>12009 (85.7) 0.015 | 1658.3 (3.3)<br>1658.3 (3.3)<br>9848.9 (39.7)<br>22372.1 (44.8)<br>43007.3 (86.1) | 511.0(3.5) 0.012<br>1376.0 (19.4) 0.003<br>7588.0 (44.0) 0.015<br>14779.0 (85.7) 0.01 | 2289 (11.1)<br>7872 (38.2)<br>16513 (80.1) | 675 (13.0)<br>2262 (43.5)<br>4161 (80.1) | 0.058<br>0.109<br>0.001 | 142 (2.9) 142 (2.9) 0.001<br>614 (12.4) 636 (12.8) 0.013<br>2167 (43.8) 2116 (43.1) 0.013<br>3949 (79.8) 3961 (80.0) 0.006 | 2613.1 (12.9)<br>8896.7 (43.9)<br>16246.6 (80.1) | 282.0 (5.4) 0.004<br>150.0 (2.9) 0.002<br>675.0 (13.0) 0.004<br>2255.0 (43.5) 0.008<br>4154.0 (80.1) 0.002<br>2946.0 (76.1) 0.001 | 4261 (8.5) 24 (8.5)<br>16880 (33.7) 722 (41.5)<br>25300 (70.5) 1231 (70.8) | 0.054<br>0.001<br>0.161<br>0.006<br>0.015 | 139 (E.2) 145 (E.6) 0.032<br>648 (18.3) 688 (40.7) 0.048<br>1199 (70.9) 1200 (71.0) 0.001 | 4084.6 (8.5) 148.0 (8.5) 0.000<br>19708.0 (41.0) 720.0 (41.5) 0.008<br>34042.6 (70.9) 1230.0 (70.8) 0.002 |
| Hyperlipidemia; n (%) Atrial fibrillation; n (%) Acute MI; n (%) | 39569 (75.4)<br>6369 (12.3)<br>895 (1.7) | 13663 (79.3) 0.068<br>1735 (10.1) 0.07<br>319 (1.9) 0.01 | 11993 (79.0)<br>1587 (10.5)<br>271 (1.8) | 11957 (78.7) 0.006<br>1575 (10.4) 0.003<br>258 (1.7) 0.007 | 19613.5 (79.3)<br>5101.9 (10.2)<br>506.9 (1.8) | 13662.0 (79.3) 0.002<br>1735.0 (10.1) 0.005<br>119.0 (1.9) 0.003 | 15076 (73.1)<br>2011 (9.8)<br>423 (2.1) | 3954 (76.1)<br>370 (7.1)<br>112 (2.2) | 0.068<br>0.095<br>0.007 | 3758 (75.9) 3752 (75.8) 0.003<br>361 (7.3) 353 (7.1) 0.006<br>90 (1.8) 106 (2.1) 0.023 | 15431.0 (76.1)<br>1416.3 (7.0)<br>423.6 (2.1) | 2948.0 (76.1) 0.001<br>370.0 (7.1) 0.006<br>111.0 (2.1) 0.003 | 20951 (53.8) 949 (54.6)<br>2006 (14.0) 227 (13.1)<br>204 (1.4) 25 (1.4) | 0.015<br>0.028<br>0.003 | 910 (53.8) 920 (54.4) 0.012<br>225 (13.3) 224 (13.3) 0.002<br>22 (1.3) 25 (1.5) 0.015 | 26258.8 (54.7) 948.0 (54.6) 0.002<br>6327.9 (13.2) 227.0 (13.1) 0.003<br>709.1 (1.5) 25.0 (1.4) 0.003 |
| Old MI; n (%) Cononary atherosclerosis; n (%) History of CABG(FTCA; n (%) | 2500 (4.8)<br>15675 (30.2)<br>4881 (9.4) | 10012.5 1001 | 715 (4.7)<br>4661 (30.7)<br>1395 (9.2) | 13927 (PLF) 0.000 1377 (PLF) 0.000 | 2327.5 (4.7)<br>15617.7 (31.3)<br>4654.6 (9.3)<br>612.3 (1.2) | 780.0 (4.5) 0.006<br>5365.0 (31.1) 0.003<br>1586.0 (9.2) 0.004<br>206.0 (1.2) 0.002<br>13.0 (0.1) 0.002 | 555 (2.7)<br>5976 (29.0)<br>876 (4.2) | 137 (2.6)<br>1478 (28.4)<br>214 (4.1) | 0.068<br>0.095<br>0.007<br>0.004<br>0.012<br>0.001<br>0.011<br>0.061<br>0.061<br>0.001<br>0.074<br>0.074<br>0.09 | 135 (2.7) 131 (2.6) 0.005<br>1415 (28.6) 1408 (28.4) 0.003<br>211 (4.3) 209 (4.2) 0.002 | 519.0 (2.6)<br>5743.5 (28.3)<br>880.9 (4.3) | 136.0 (2.6) 0.004<br>3476.0 (28.4) 0.003<br>214.0 (4.1) 0.011<br>68.0 (1.3) 0.01<br>2.0 (0.0) 0.004 | 2120 (4.3) 67 (2.9)<br>24126 (29.6) 536 (30.2)<br>4346 (8.7) 147 (8.5)<br>635 (1.3) 28 (1.6) | 0.02<br>0.023<br>0.008<br>0.029<br>0.001 | 74 [4.4] 55 (3.9) 0.024<br>537 [31.8] 510 (30.2) 0.035<br>130 (7.7) 145 (8.6) 0.032<br>25 [1.5] 28 (1.7) 0.014 | 1885.9 (3.9) 67.0 (3.9) 0.004<br>14422.2 (30.00) 555.0 (30.2) 0.004<br>4055.2 (8.4) 147.0 (8.5) 0.002<br>788.0 (1.5) 28.0 (1.6) 0.006 |
| Previous cardiac procedure; n (%) Cerebrovascular procedure; n (%) Ischemic stroke; n (%) | 571 (1.1)<br>45 (0.1)<br>5398 (10.4) | 208 (1.2) 0.01<br>13 (0.1) 0.004<br>1607 (9.3) 0.016 | 167 (1.1)<br>14 (0.1)<br>1478 (9.7) | 174(1.1) 0.004<br>12 (0.1) 0.005<br>1444 (9.5) 0.008 | 612.3 (1.2)<br>41.1 (0.1)<br>4804.8 (9.6) | 208.0 (1.2) 0.002<br>13.0 (0.1) 0.002<br>1607.0 (9.3) 0.01 | 295 (1.4)<br>26 (0.1)<br>1793 (8.7) | 68 (1.3)<br>2 (0.0)<br>340 (6.5) | 0.011<br>0.016<br>0.081 | 125 (2.7) 131 (2.6) 0.005<br>1415 (2.6) 1406 (2.4) 0.000<br>211 (4.3) 200 (4.2) 0.000<br>63 (1.3) 67 (1.4) 0.007<br>3 (0.1) 2 (0.0) 0.000<br>218 (6.4) 33 (6.7) 0.011 | 289.5 (1.4)<br>6.5 (0.0)<br>1364.1 (6.6) | 136.0 (2.6) 0.004<br>1476.0 (28.4) 0.003<br>214.0 (4.1) 0.011<br>68.0 (1.3) 0.01<br>2.0 (0.0) 0.004<br>139.0 (6.5) 0.004<br>139.0 (7.5) 0.005 | 635 (1.3) 28 (1.6)<br>57 (0.1) 2 (0.1)<br>4593 (8.2) 152 (8.7) | 0.029<br>0.001<br>0.015 | 25 (1.5) 28 (1.7) 0.014<br>2 (0.1) 2 (0.1) 0.001<br>152 (9.0) 151 (8.9) 0.002 | 738.0 (1.5) 28.0 (1.6) 0.006<br>60.1 (0.1) 2.0 (0.1) 0.003<br>4146.7 (8.6) 152.0 (8.8) 0.004 |
| PVD diagnosis or surgery; n (%) CXD Stage 3-4; n (%) Other cardiac dysrhythmia; n (%) | 8041 (15.5)<br>15765 (20.4)<br>8640 (16.6) | | 2153 (14.2)<br>4237 (27.9)<br>2344 (15.4) | 2112 (13.9) 0.008<br>4165 (27.4) 0.011<br>2357 (15.5) 0.002 | 6862.2 (13.7)<br>13646.9 (27.3)<br>7924.1 (15.9)<br>2721.4 (5.4) | 2326.0 (13.5) 0.007<br>4584.0 (26.6) 0.016<br>2676.0 (15.5) 0.009 | 2160 (10.5)<br>3434 (16.7)<br>2961 (14.4) | 393 (7.6)<br>674 (13.0)<br>616 (11.9) | 0.102<br>0.104<br>0.074 | 642 (3.0) 642 (3.0) 0.001<br>594 (3.0) 588 (3.9) 0.004 | 1562 8 (7.7)<br>2671 3 (13.2)<br>2475 2 (12.2) | 474 O (13 O) 0 00F | 5028 (10.0) 161 (9.3)<br>9968 (19.9) 347 (20.0)<br>7560 (15.1) 231 (13.3) | 0.027<br>0.001<br>0.052 | 161 (9.6) 160 (9.5) 0.006<br>338 (20.0) 339 (20.1) 0.001 | 4473.7 (9.3) 161.0 (9.3) 0.002<br>9658.8 (20.1) 347.0 (20.0) 0.003<br>6312.1 (13.1) 229.0 (13.2) 0.001 |
| Cardiomyopathy; n (%) Valve disorders; n (%) COPD; n (%) | 3067 (5.9)<br>1330 (2.6)<br>8674 (16.7) | 4584 (26.6) 0.084<br>2676 (15.5) 0.031<br>924 (5.4) 0.024<br>258 (2.1) 0.032<br>254 (14.9) 0.05<br>1179 (68) 0.039 | 821 (5.4)<br>360 (2.4)<br>2341 (15.4) | 807 (5.3) 0.004<br>330 (2.2) 0.013<br>2314 (15.2) 0.005 | 2721.4 (5.4)<br>1095.0 (2.2)<br>7888.2 (15.8) | 4584.0 (26.6) 0.016<br>(2676.0 (15.5) 0.000<br>124.0 (5.4) 0.004<br>158.0 (2.1) 0.008<br>158.0 (24.9) 0.025 | 2024 (5.0)<br>270 (1.8)<br>2186 (10.6) | 265 (4.7)<br>54 (1.2)<br>416 (8.0) | 0.013<br>0.046<br>0.09 | 229 (4.8) 229 (4.6) 0.01<br>61 (1.2) 56 (1.1) 0.009<br>429 (8.7) 397 (8.0) 0.023 | 951.8 (4.7)<br>241.7 (1.2)<br>1581.8 (7.8) | 514.0 (1.18) 0.031<br>246.0 (4.7) 0.002<br>54.0 (1.2) 0.004<br>416.0 (6.0) 0.008<br>274.0 (5.3) 0.001 | 9968 (19.9) 347 (20.0)<br>7560 (15.1) 221 (12.3)<br>2421 (4.8) 84 (4.8)<br>1289 (2.8) 43 (2.5)<br>6381 (12.7) 218 (12.5) | 0.001<br>0.052<br>0.001<br>0.019<br>0.006<br>0.001 | 82 (24.9) 0.014<br>82 (4.9) 0.014<br>80 (2.4) 41 (2.4) 0.004<br>215 (12.7) 214 (12.7) 0.002 | 2248.4 (4.7) 84.0 (4.8) 0.007<br>1162.7 (2.4) 41.0 (2.5) 0.004<br>5993.4 (12.5) 218.0 (12.6) 0.002 |
| Asthma; n (%) Obstructive sleep apnea; n (%) Pneumonia; n (%) | 3179 (6.1)<br>6663 (12.8)<br>2086 (4.0) | 1179 (6.8) 0.029<br>3412 (19.8) 0.189<br>468 (2.7) 0.072 | 990 (E.S)<br>2723 (17.9)<br>422 (2.8) | 1021 (6.7) 0.008<br>2754 (18.1) 0.005<br>430 (2.8) 0.001 | 3482.7 (7.0)<br>9843.6 (19.7)<br>1471.6 (2.9) | 1179.0 (6.8) 0.005<br>1412.0 (19.8) 0.002 | 994 (4.8)<br>3206 (15.6)<br>785 (3.8) | 274 (5.3)<br>1132 (21.8)<br>141 (2.7) | 0.021<br>0.16<br>0.062 | 250 (5.0) 260 (5.3) 0.009<br>1039 (21.0) 1039 (21.0) 0.001<br>126 (2.5) 132 (2.7) 0.008 | 1067.1 (5.3)<br>4327.9 (21.3)<br>530.0 (2.6) | 1128.0 (21.7) 0.01<br>140.0 (2.7) 0.005 | 2494 (5.0) 87 (5.0)<br>4662 (9.3) 238 (13.7)<br>1993 (4.0) 46 (2.6) | 0.001<br>0.137<br>0.075 | 88 (5.2) 86 (5.1) 0.005<br>248 (14.7) 229 (13.6) 0.032<br>44 (2.6) 46 (2.7) 0.007 | 2401.2 (5.0) 87.0 (5.0) 0.001<br>6460.0 (13.5) 237.0 (13.6) 0.006<br>1291.5 (2.7) 46.0 (2.6) 0.003 |
| CKD Stage 1-2; n (S) Acute renal disease (AO); n (S) Nephrotic syndrome; n (S) | 3092 (6.0)<br>3299 (6.4)<br>42 (0.1) | 888 (5.2) 0.035<br>698 (4.0) 0.104<br>6 (0.0) 0.019<br>2737 (15.9) 0.074 | 831 (5.5)<br>675 (4.4)<br>6 (0.0) | 2754 (18.1) 0.005<br>430 (2.8) 0.003<br>803 (5.3) 0.003<br>639 (4.2) 0.012<br>6 (0.0) 0.001<br>2483 (16.4) 0.002<br>8814 (58.0) 0.011 | 2621.1 (5.2)<br>2102.8 (4.2)<br>17.4 (0.0)<br>8125.2 (16.3) | 188.0(5.2) 0.004<br>198.0(5.2) 0.005<br>198.0(4.0) 0.005<br>5.0(0.0) 0.001<br>2727.0(15.9) 0.011<br>1980.0(57.9) 0.025 | 470 (2.3)<br>1075 (5.2)<br>17 (0.1) | 108 (2.1)<br>140 (2.7)<br>4 (0.1) | 0.16<br>0.062<br>0.014<br>0.13<br>0.002<br>0.098<br>0.029 | 89 (1.8) 105 (2.1) 0.023<br>130 (2.4) 137 (2.8) 0.009<br>5 (0.1) 4 (0.1) 0.007 | 426.8 (2.1)<br>567.3 (2.8)<br>16.0 (0.1) | 108.0 (2.1) 0.002<br>340.0 (2.7) 0.005<br>4.0 (0.1) 0.001<br>383.0 (7.4) 0.001<br>2599.0 (50.1) 0.014 | 1085 (2.2) 38 (2.2)<br>3187 (6.4) 66 (3.8)<br>33 (0.1) 1 (0.1) | 0.001<br>0.117<br>0.003 | 36 (2.1) 38 (2.2) 0.008<br>65 (3.8) 65 (3.8) 0.001<br>1 (0.1) 1 (0.1) 0.001 | 1053.8 (2.2) 38.0 (2.2) 0.001<br>1792.2 (3.7) 66.0 (3.8) 0.004<br>29.1 (0.1) 1.0 (0.1) 0.001 |
| Hypertensive nephropathy; n (%) Other renal conditions; n (%) Liver disease; n (%) | 9693 (18.7)<br>29991 (57.8)<br>5500 (10.6) | 2737 (15.9) 0.074<br>9981 (57.9) 0.002<br>1953 (11.3) 0.023 | 2473 (16.3)<br>8897 (58.6)<br>1677 (11.0) | 2483 (16.4) 0.002<br>8814 (58.0) 0.011<br>1680 (11.1) 0.001 | 8125.2 (16.3)<br>29539.3 (59.1)<br>5675.6 (11.4) | 2737.0 (15.9) 0.011<br>9980.0 (57.9) 0.025<br>1953.0 (11.3) 0.001 | 2092 (10.1)<br>10046 (48.7)<br>1829 (8.9) | 383 (7.4)<br>2607 (50.2)<br>437 (8.4) | 0.098<br>0.029<br>0.017 | 357 (7.2) 360 (7.3) 0.002<br>2516 (50.8) 2463 (49.7) 0.021<br>423 (8.5) 418 (8.4) 0.004 | 1491.8 (7.4)<br>10297.6 (50.8)<br>1794.1 (8.8) | 2599.0 (50.1) 0.001<br>2599.0 (50.1) 0.014<br>437.0 (8.4) 0.015 | 6378 (12.7) 196 (11.3)<br>23107 (46.2) 906 (52.1)<br>2815 (5.6) 97 (5.6) | 0.003<br>0.045<br>0.119<br>0.002 | 186 (11.0) 190 (11.2) 0.008<br>839 (49.6) 870 (51.5) 0.037<br>86 (5.1) 93 (5.5) 0.018 | 5395.2 (11.2) 196.0 (11.3) 0.001<br>24917.7 (51.9) 905.0 (52.1) 0.004<br>2627.1 (5.5) 96.0 (5.5) 0.002 |
| Hypothyroidsm; n (%) Outcoarthrist; n (%) Fractures; n (%) Factures; n (%) | 9435 (18.2)<br>10887 (21.0)<br>847 (1.6) | 1053 (11.3) 0.003<br>1053 (11.3) 0.003<br>1054 (17.5) 0.008<br>1056 (20.9) 0.001<br>225 (1.3) 0.002<br>245 (1.3) 0.05<br>1054 (4.0) 0.05<br>1054 (4.1) 0.05<br>1054 (4.1) 0.05<br>1054 (4.1) 0.05<br>1054 (4.1) 0.05 | 2681 (17.7)<br>3093 (20.4)<br>191 (1.3) | BB14(16.0] | 8825.1 (17.7)<br>10740.4 (21.5)<br>659.5 (1.3) | 2014.0 (17.5) 0.005<br>1605.0 (20.9) 0.014<br>215.0 (1.2) 0.006 | March Marc | 725 (14.0)<br>755 (14.5)<br>45 (0.9) | 0.029 0.017 0.024 0.02 0.055 0.086 0.05 0.090 0.001 | 688 (13.9) 697 (14.1) 0.005<br>736 (14.9) 731 (14.4) 0.014<br>34 (0.7) 45 (0.9) 0.035<br>64 (1.3) 69 (1.4) 0.009 | 2848.1 (14.0)<br>2901.9 (14.1)<br>165.5 (0.8) | 726.0 (14.0) 0.002<br>756.0 (14.6) 0.007<br>46.0 (0.9) 0.008<br>71.0 (1.4) 0.003<br>76.0 (1.5) 0.006 | 7622 (15.2) 280 (16.1)<br>9028 (18.0) 314 (18.1)<br>788 (1.6) 25 (1.4) | 0.024<br>0.001<br>0.013 | 267 (15.8) 270 (16.0) 0.005<br>286 (16.9) 304 (18.0) 0.028<br>27 (1.6) 23 (1.4) 0.02 | 7747.6 (16.1) 280.0 (16.1) 0.001<br>8688.3 (18.1) 314.0 (18.1) 0.001<br>647.1 (1.3) 25.0 (1.4) 0.008 |
| Past; n (%) Osteoporosis; n (%) Asystem n (%) Asystem n (%) | 2675 (5.2)<br>7593 (14.6) | 411 (2.4) 0.06<br>695 (4.0) 0.053<br>2434 (14.1) 0.015 | 683 (4.5)<br>2146 (14.1)<br>1822 (12.0) | 853 (4.3) 0.01<br>253 (4.1) 0.02<br>2134 (14.1) 0.002 | 2084.3 (4.2)<br>7102.8 (14.2)<br>6368.6 (12.7) | 1605.0 (20.9) 0.014<br>215.0 (1.2) 0.006<br>413.0 (2.4) 0.009<br>196.0 (4.0) 0.007<br>2434.0 (34.1) 0.003<br>2142.0 (22.4) 0.05 | 437 (2.1)<br>2082 (10.1)<br>1969 (9.6) | 75 (1.5)<br>495 (9.5)<br>511 (9.8) | 0.05 | 65 (1.3) 75 (1.5) 0.017<br>479 (9.7) 465 (9.4) 0.017<br>519 (10.5) 485 (9.4) 0.025 | 312.6 (1.5)<br>1911.8 (9.4)<br>2019.2 (10.0) | 756.0 (14.6) 0.007<br>45.0 (0.5) 0.008<br>71.0 (1.4) 0.003<br>76.0 (1.5) 0.006<br>495.0 (9.5) 0.004<br>500.0 (9.8) 0.004 | 9028 (18.0) 314 (18.1)<br>798 (1.6) 25 (2.4)<br>155 (0.3) 1 (0.1)<br>2421 (4.8) 77 (4.4)<br>4528 (9.0) 167 (9.6)<br>3556 (7.1) 117 (6.2) | 0.001<br>0.013<br>0.059<br>0.019<br>0.019 | 1(0.1) 1(0.1) 0.001<br>68 (4.0) 72 (4.3) 0.012<br>169 (10.0) 161 (9.5) 0.016<br>115 (6.8) 113 (6.7) 0.005 | 27.7 (0.1) 1.0 (0.1) 0.001<br>2098.2 (4.4) 77.0 (4.4) 0.003<br>4566.2 (9.5) 167.0 (9.6) 0.004<br>222.3 (6.7) 117.0 (6.7) 0.004 |
| Skep disorder; n (%) Dementia; n (%) Delinium; n (%) | 11831 (22.8)<br>3921 (7.6)<br>886 (1.7) | 4031(23.4) 0.014<br>500(1.2) 0.191<br>105 (0.6) 0.103<br>870(5.0) 0.032<br>1.21 (0.92) 0.002<br>2989 (17.3) 0.018 | 3459 (22.8)<br>561 (3.7)<br>99 (0.7) | 3514 (23.1) 0.009<br>544 (3.6) 0.006<br>303 (0.7) 0.003 | 11961.8 (23.9)<br>1656.2 (3.3)<br>315.6 (0.6) | | 3303 (16.0)<br>937 (4.5)<br>337 (1.6) | 826 (15.9)<br>56 (1.1)<br>22 (0.4) | 0.004<br>0.211<br>0.12 | 802 (16.2) 787 (15.9) 0.008<br>54 (1.1) 56 (1.1) 0.004<br>18 (0.4) 22 (0.4) 0.013 | 3303.4 (16.3)<br>209.5 (1.0)<br>84.6 (0.4) | 823.0 (15.9) 0.012<br>55.0 (1.1) 0.003<br>21.0 (0.4) 0.002 | 8542 (27.1) 279 (16.0)<br>2897 (5.8) 50 (2.9)<br>860 (1.7) 24 (1.4)<br>480 (1.0) 33 (1.9) | 0.028<br>0.141<br>0.027 | 257 (15.2) 273 (16.2) 0.026<br>59 (3.5) 50 (3.0) 0.03<br>17 (1.0) 23 (1.4) 0.033 | 7628.0 (15.9) 277.0 (15.9) 0.002<br>1380.8 (2.9) 49.0 (2.8) 0.003<br>631.6 (1.3) 24.0 (1.4) 0.006 |
| COVID; n (%) Number of antidabetic drugs on CED mean (sd) | 2252 (4.3) | 870 (5.0) 0.033 | 745 (4.9)<br>1.22 (0.89) | 763 (5.0) 0.005<br>1.22 (0.91) 0.003 | 1656.2 (3.3)<br>315.6 (0.6)<br>2484.7 (5.0)<br>1.22 (0.90) | 560.0(3.2) 0.004<br>105.0(0.6) 0.003<br>170.0(5.0) 0.003<br>1.21(0.92) 0.013<br>2989.0(17.3) 0.013 | 871 (4.2)<br>1.16 (0.86) | 1.22 (0.92) | 0.071 | 275 [5.6] 279 [5.6] 0.004<br>1.22 (0.90) 1.22 (0.92) 0.001 | 12113 (6.0) | 55.0(1.1) 0.003<br>21.0(0.4) 0.002<br>300.0(5.8) 0.008<br>1.22(0.92) 0.001<br>875.0(16.9) 0.016 | 489 (1.0) 33 (1.9)<br>1.18 (0.84) 1.21 (0.90) | 0.027<br>0.027<br>0.077<br>0.119<br>0.182 | 38 (2.2) 31 (1.8) 0.029<br>1.28 (0.91) 1.29 (0.89) 0.009 | 908.3 (1.9) 33.0 (1.9) 0.001<br>1.30 (0.90) 1.30 (0.90) 0.006 |
| Insulatin; n (%) Migitalides; n (%) SU-2nd een: n (%) | 8657 (16.7)<br>570 (1.1)<br>17351 (33.4) | 2989 (17.3) 0.018<br>154 (0.9) 0.021<br>5359 (31.0) 0.051 | 2656 (17.6)<br>134 (0.9)<br>4874 (32.1) | 2617 (17.2) 0.009<br>140 (0.9) 0.004<br>4845 (31.9) 0.004 | 1.22 (0.90)<br>9287.3 (18.6)<br>451.0 (0.9)<br>16957.1 (32.1) | 2989.0 (17.3) 0.033<br>154.0 (0.9) 0.001<br>5349.0 (31.0) 0.024 | 3052 (14.8)<br>237 (1.1)<br>5824 (28.3) | 880 (16.9)<br>42 (0.8)<br>1347 (25.9) | 0.058<br>0.035<br>0.053 | #18 (16.5) #29 (16.7) 0.006<br>47 (0.9) 42 (0.8) 0.011<br>1307 (26.4) 1291 (26.1) 0.007 | 3542.9 (17.5)<br>163.5 (0.8)<br>5332.4 (26.3) | 875.0 (16.9) 0.016<br>42.0 (0.8) 0.001<br>1345.0 (25.9) 0.009 | 8547 (17.1) 425 (24.4)<br>865 (1.7) 32 (1.8)<br>17558 (15.1) 596 (14.3) | 0.182<br>0.008<br>0.017 | 386 (22.8) 406 (24.0) 0.028<br>29 (1.7) 31 (1.8) 0.009<br>604 (35.7) 575 (34.0) 0.036 | 11760.1(24.5) 424.0(24.4) 0.002<br>868.2(1.8) 32.0(1.8) 0.003<br>16607.7(14.6) 596.0(14.3) 0.006 |
| Metformin; n (%) Thiazoldinedones; n (%) SGLT-2i: n (%) | 25735 (49.6)<br>3534 (6.8)<br>6700 (12.9) | 154 (0.9) 0.021<br>5350 (21.0) 0.051<br>10165 (00.1) 0.233<br>1098 (0.1) 0.049<br>4457 (25.9) 0.332<br>69 (0.4) 0.003<br>12166 (70.6) 0.022 | 8958 (59.0)<br>1257 (8.3)<br>3574 (23.5) | 340 (9.9) 0.004 4845 (31.9) 0.004 4845 (31.9) 0.004 3802 (58.6) 0.007 3201 (7.9) 0.014 3575 (23.5) 0.001 46 (9.4) 0.004 30712 (70.5) 0.003 | 10316.0 (60.7)<br>4288.1 (8.6)<br>13559.0 (27.1) | 154.0 (0.9) 0.001<br>5149.0 (31.0) 0.024<br>10165.0 (60.1) 0.011<br>1298.0 (8.1) 0.017<br>4457.0 (25.9) 0.029<br>159.0 (0.4) 0.011 | 10567 (51.3)<br>995 (4.8)<br>3111 (15.1) | 3392 (65.3)<br>314 (6.0)<br>1643 (31.6) | 0.015<br>0.053<br>0.287<br>0.054<br>0.398<br>0.006 | 2195 (64.5) 2196 (64.6) 0.001<br>293 (5.9) 284 (5.7) 0.008<br>3458 (29.4) 1467 (29.6) 0.004<br>17(0.3) 19 (0.4) 0.007 | 13293.5 (65.6)<br>1206.3 (5.9)<br>6292.2 (31.0) | 42.0 (0.1) 0.001<br>1345.0 (25.9) 0.009<br>1346.0 (65.1) 0.005<br>311.0 (6.0) 0.004<br>1616.0 (31.5) 0.011<br>19.0 (64.0) 0.001<br>3607.0 (69.5) 0.005 | 25148 (50.2) 1103 (63.4)<br>3003 (6.0) 126 (7.2)<br>4102 (8.2) 418 (24.0) | 0.008<br>0.017<br>0.269<br>0.05<br>0.441<br>0.04<br>0.043 | 1014 (E0.0) 1004 (E3.0) 0.061<br>124 (7.3) 119 (7.0) 0.011<br>159 (20.7) 373 (22.1) 0.033 | 30549.2 (63.6) \$101.0 (63.4) 0.095<br>3427.9 (7.1) \$26.0 (7.3) 0.094<br>\$10975.2 (22.9) 417.0 (24.0) 0.027 |
| Alpha-glucosidase inhibitors; n (%)<br>ACE + ARBs; n (%)<br>Thiazides; n (%) | 217 (0.4)<br>36114 (69.6)<br>14066 (27.1) | 69 (0.4) 0.003<br>12166 (70.6) 0.022<br>5172 (30.0) 0.064 | 68 (0.4)<br>10731 (70.7)<br>4552 (30.0) | 64 (0.4) 0.004<br>10712 (70.5) 0.003<br>4507 (29.7) 0.006 | 235.3 (0.5)<br>35361.2 (70.8)<br>14931.7 (29.9) | 59.0 (0.4) 0.011<br>12165.0 (70.6) 0.005<br>5172.0 (30.0) 0.002 | 68 (0.3)<br>13924 (67.6)<br>5562 (27.0) | 19 (0.4)<br>3612 (69.5)<br>1546 (30.1) | 0.006<br>0.042<br>0.07 | 17(0.3) 19(0.4) 0.007<br>3438 (69.4) 3441 (69.5) 0.001<br>1458 (29.4) 1485 (30.0) 0.012 | 74.4 (0.4)<br>14053.9 (69.3)<br>6068.8 (29.9) | 19.0 (0.4) 0.001<br>3607.0 (69.5) 0.005<br>1564.0 (30.1) 0.005 | 221 (0.4) 13 (0.7)<br>34509 (68.9) 1233 (70.9)<br>13133 (26.2) 491 (28.2) | 0.04<br>0.043<br>0.045 | 15 (0.9) 9 (0.5) 0.042<br>1223 (72.4) 1197 (70.8) 0.034<br>482 (28.5) 473 (28.0) 0.012 | 342.1(0.7) 13.0(0.7) 0.054<br>34138.8(71.1) 1231.0(70.9) 0.055<br>13592.5(28.3) 460.0(28.2) 0.052 |
| Beta blockers; n (%) Calcium channel blockers; n (%) Loop diuretics; n (%) | 26462 (51.0)<br>18766 (36.2)<br>9543 (18.4) | 8714 (50.5) 0.009<br>5992 (34.6) 0.033<br>3057 (17.7) 0.017<br>1349 (7.8) 0.043<br>1644 (8.4) 0.01 | 7755 (51.1)<br>5342 (35.2)<br>2717 (17.9) | 7672 (50.5) 0.011<br>5325 (35.1) 0.002<br>2696 (17.8) 0.004 | 25472.8 (51.0)<br>17526.8 (35.1)<br>9125.6 (18.1) | 8714.0 (50.5) 0.009<br>5961.0 (34.6) 0.011<br>8057.0 (17.7) 0.014 | 10357 (50.2)<br>6929 (33.6)<br>3095 (15.0) | 2454 (47.4)<br>1552 (29.9)<br>673 (12.9) | 0.057<br>0.061<br>0.06 | 2370 (47.9) 2354 (47.5) 0.006<br>1462 (29.5) 1489 (30.1) 0.012<br>621 (12.5) 629 (12.7) 0.005 | 9661.1 (47.6)<br>6150.4 (30.3)<br>2575.4 (12.7) | 2462.0 (47.4) 0.004<br>1551.0 (29.9) 0.01<br>672.0 (13.0) 0.007 | 28335 (56.6) 1015 (58.4)<br>18472 (36.9) 610 (35.1)<br>11152 (22.3) 419 (24.1) | 0.036<br>0.038<br>0.043 | 1005 (59.5) 981 (58.0) 0.029<br>623 (36.9) 602 (35.6) 0.026<br>376 (22.2) 405 (24.0) 0.041 | 27936.5 (58.2) 1015.0 (58.4) 0.005<br>17038.1 (35.5) 610.0 (35.1) 0.008<br>11563.1 (24.1) 419.0 (24.1) 0.001 |
| Other diaretics; n (%) Nitrates; n (%) HF drugs (Digoxin + Entresto + Ivabadrine); n (%) | 3478 (6.7)<br>4200 (8.1)<br>1383 (2.7) | 1349 (7.8) 0.043<br>1444 (8.4) 0.01<br>457 (2.7) 0.001 | 1140 (7.5)<br>1278 (8.4)<br>385 (2.5) | 1162 (7.7) 0.005<br>1248 (8.2) 0.007<br>400 (2.6) 0.006 | 9125.6 (18.3)<br>1951.0 (7.9)<br>4228.5 (8.5)<br>1338.2 (2.7) | 5961.0 (34.6) 0.011<br>1057.0 (17.7) 0.014<br>1349.0 (7.8) 0.003<br>1443.0 (8.4) 0.003<br>457.0 (2.7) 0.002 | 1457 (7.1)<br>1682 (8.2)<br>525 (2.5) | 376 (7.2)<br>404 (7.8)<br>131 (2.5) | 0.006<br>0.014<br>0.002 | 353 (7.1) 344 (6.9) 0.007<br>373 (7.5) 383 (7.7) 0.006<br>127 (2.4) 120 (2.4) 0.009 | 1434.6 (7.1)<br>1620.4 (8.0)<br>510.5 (2.5) | 1564.0 (30.1) 0.005<br>2462.0 (47.4) 0.004<br>1551.0 (29.9) 0.01<br>672.0 (13.0) 0.007<br>175.0 (7.2) 0.005<br>402.0 (7.7) 0.009<br>111.0 (2.5) 0.001<br>90.0 (1.7) 0.004 | 3753 (7.5) 172 (9.9)<br>4940 (9.9) 181 (10.4)<br>1688 (1.4) 55 (3.2) | 0.038<br>0.043<br>0.085<br>0.018<br>0.012 | 139 (8.2) 162 (9.6) 0.048<br>180 (10.7) 172 (10.2) 0.015<br>54 (3.2) 53 (3.1) 0.001 | 4611.8 (9.6) 172.0 (9.9) 0.01<br>4977.8 (10.4) 181.0 (10.4) 0.002<br>1517.9 (3.2) 55.0 (3.2) 0.001 |
| Anti-arrhythmics; n (%) COPD/asthma meds; n (%) Statins; n (%) | 1175 (2.3)<br>12374 (23.8)<br>40924 (78.9) | 309 (1.8) 0.033<br>4478 (26.0) 0.049<br>13901 (80.6) 0.044 | 269 (1.8)<br>3953 (26.0)<br>12317 (81.1) | 281 (1.9) 0.006<br>2924 (25.8) 0.004<br>12231 (80.6) 0.014 | 886.2 (1.8)<br>13387.6 (26.8)<br>40500.7 (81.1) | | 455 (2.2)<br>4401 (21.4)<br>15340 (74.4) | 90 (1.7)<br>1176 (22.6)<br>4025 (77.4) | 0.034<br>0.031<br>0.071 | 88 (1.8) 83 (1.7) 0.006<br>1102 (22.3) 1119 (22.6) 0.006<br>3835 (77.5) 3823 (77.2) 0.006 | 341.2 (1.7)<br>4570.9 (22.5)<br>15730.4 (77.6) | 90.0 (1.7) 0.004<br>1175.0 (22.6) 0.002<br>4018.0 (77.4) 0.003 | 1607 (3.2) 47 (2.7)<br>12026 (24.0) 423 (24.3)<br>38758 (77.4) 1396 (80.3) | 0.007 | 49 (2.9) 45 (2.7) 0.014<br>412 (24.4) 410 (24.3) 0.001<br>1353 (80.1) 1356 (80.2) 0.004 | 1289.9 (2.7) 47.0 (2.7) 0.001<br>11703.5 (24.4) 423.0 (24.4) 0.001<br>38527.4 (80.2) 1395.0 (80.3) 0.002 |
| Other lipid-lowering drugs; n (%) Antiplatelet agents; n (%) Oral anticoagulants; n (%) | 5544 (10.7)<br>7998 (15.4)<br>6163 (11.9) | \$377(20.0) | 1874 (12.3)<br>2317 (15.3)<br>1598 (10.5) | 18711/0519 0.0001 18711/0519 0.0001 18711/0519 0.0001 18711/0519 0.0001 18711/0519 0.0001 18711/1519 0.0001 | 40500.7 (B1.1)<br>6333.8 (12.7)<br>7574.8 (15.2)<br>5281.8 (30.6)<br>10518.1 (21.1) | 1478.0 (26.0) 0.029<br>12900.0 (80.6) 0.011<br>2161.0 (22.5) 0.004<br>2617.0 (15.2) 0.005<br>1796.0 (30.4) 0.005<br>1516.0 (20.5) 0.011 | 2634 (12.8)<br>3794 (18.4)<br>2385 (11.6) | 726 (14.0)<br>901 (17.3)<br>480 (9.2) | 0.042<br>0.07<br>0.057<br>0.081<br>0.06<br>0.006<br>0.004<br>0.002<br>0.004<br>0.003<br>0.071<br>0.071<br>0.071<br>0.071<br>0.071<br>0.071 | 600 (13.9) 600 (13.9) 0.001<br>862 (17.4) 862 (17.4) 0.001<br>476 (9.6) 464 (9.4) 0.005<br>988 (20.0) 992 (20.0) 0.002 | 2871.3 (14.2)<br>2573.0 (17.6)<br>1891.1 (9.3)<br>4108.6 (20.3) | 1175.0(22.6) 0.002<br>4018.0(77.4) 0.003<br>726.0 (14.0) 0.005<br>899.0 (17.3) 0.003<br>480.0 (0.3) 0.003<br>1056.0 (0.04) 0.002<br>715.0 (13.8) 0.008 | 12006 (24.9) 42 (24.1)<br>38758 (77.4) 1396 (90.3)<br>5958 (11.9) 565 (15.2)<br>880 (17.6) 385 (15.2)<br>286 (15.7) 277 (11.6)<br>3908 (18.2) 355 (20.4)<br>5000 (18.2) 355 (20.4) | 0.098<br>0.048<br>0.002 | 412 (24.4) 410 (24.3) 0.003<br>1351 (80.3) 1356 (80.2) 0.004<br>257 (15.2) 250 (44.8) 0.012<br>331 (19.7) 331 (19.6) 0.003<br>252 (14.8) 262 (15.5) 0.006<br>252 (14.8) 262 (15.5) 0.016<br>351 (20.6) 342 (20.3) 0.015 | 7241.4 (15.1) 263.0 (15.1) 0.002<br>9279.7 (19.3) 338.0 (19.5) 0.003<br>7421.4 (15.5) 272.0 (15.7) 0.006 |
| NSAIDs; n (%) Oral conticesteroids; n (%) Bisphosphonates; n (%) | 9436 (18.2)<br>6217 (12.0)<br>1722 (1.3) | 2536 (20.5) 0.059<br>2293 (13.3) 0.04<br>415 (2.4) 0.055 | 3088 (20.3)<br>1973 (13.0)<br>386 (2.5) | 3080 (20.3) 0.001<br>1993 (13.1) 0.004<br>393 (2.6) 0.003 | 10518.1 (21.1)<br>6746.1 (13.5)<br>1222.0 (2.4) | | 2726 (13.2)<br>2726 (13.2)<br>302 (1.5) | 1059 (20.4)<br>716 (13.8)<br>47 (0.9) | 0.057<br>0.016<br>0.052 | 988 (20.0) 992 (20.0) 0.002<br>866 (23.5) 669 (23.5) 0.002<br>45 (0.9) 47 (0.9) 0.004 | 4108.6 (20.1)<br>2852.1 (14.1)<br>191.8 (0.9) | 47.0(0.9) 0.004 | | 0.008 | 253 (20.9) 343 (20.3) 0.015<br>174 (10.3) 192 (11.4) 0.034<br>47 (2.8) 50 (3.0) 0.011 | 9739.6 (20.3) 355.0 (20.4) 0.004<br>5438.2 (11.3) 196.0 (11.3) 0.001<br>1399.2 (2.9) 51.0 (2.9) 0.001 |
| Opiolds; n (%) Anti-depressants; n (%) Gabapentinoids; n (%) | 10372 (20.0)<br>14756 (28.4)<br>11098 (21.4) | 3576 (20.7) 0.019<br>5304 (30.8) 0.051<br>3803 (22.1) 0.016 | 3173 (20.9)<br>4689 (30.9)<br>3382 (22.3) | 3140 (30.7) 0.005<br>4644 (30.6) 0.006<br>3379 (22.3) 0.001 | 10761.9 (21.5)<br>15947.4 (31.9)<br>11559.1 (23.1) | 415.0 (2.4) 0.003<br>1575.0 (20.7) 0.02<br>1304.0 (20.8) 0.025<br>1801.0 (22.1) 0.036<br>1573.0 (9.1) 0.006<br>1291.0 (8.1) 0.012 | 3712 (18.0)<br>5137 (24.9)<br>3143 (15.2) | 863 (16.6)<br>1333 (25.6)<br>795 (15.3) | 0.017<br>0.001 | 801 (16.2) 816 (16.5) 0.006<br>1392 (26.3) 1274 (25.7) 0.008<br>749 (15.1) 750 (15.1) 0.001<br>424 (8.6) 350 (7.9) 0.025<br>331 (5.7) 337 (6.8) 0.005 | 5299.5 (26.1)<br>5125.1 (15.4) | 47.0 (0.9) 0.004<br>863.0 (16.6) 0.008<br>1332.0 (25.7) 0.011<br>794.0 (15.3) 0.001<br>420.0 (8.1) 0.009<br>364.0 (7.0) 0.001<br>29.0 (0.3) 0.001 | 10062 (20.1) 191 (22.5)<br>14056 (28.1) 554 (31.9)<br>9377 (18.7) 381 (21.9) | 0.058<br>0.063<br>0.079<br>0.044<br>0.065<br>0.114 | 358 (21.2) 381 (22.5) 0.033<br>526 (31.1) 537 (31.8) 0.014<br>354 (20.9) 367 (21.7) 0.019 | 10870.1(22.6) 391.0(22.5) 0.003<br>15229.2(31.7) 553.0(31.8) 0.003<br>10489.4(21.8) 380.0(21.9) 0.001 |
| Anxiolytics/hypnotics; n (%) Demotis meds; n (%) Composition meds; n (%) | 3428 (6.6)<br>2432 (4.7) | 415 (2-4) 0.055<br>2676 (20.7) 0.019<br>5104 (20.8) 0.051<br>2003 (22.1) 0.016<br>1573 (0.1) 0.001<br>1191 (0.1) 0.055<br>258 (2.1) 0.145 | 1392 (8.2)<br>1203 (7.9)<br>354 (2.3) | 1991 11.1 0.004 | 4645.4 (9.1)<br>4197.7 (8.4)<br>1066.5 (2.1) | | ## 164.28 ## 165.24 ## 165.2 | 365 (7.0)<br>39 (0.8) | 0.052<br>0.037<br>0.017<br>0.001<br>0.002<br>0.002<br>0.042 | 36 (0.7) 39 (0.8) 0.007 | 1420.8 (7.0)<br>146.7 (0.7) | 29.0 (0.8) 0.002 | 201 (11.6)<br>2056 (6.1)<br>2820 (5.6)<br>2820 (5.6)<br>2820 (5.6) | 0.065 | 123 (7.3) 128 (7.6) 0.01<br>56 (3.3) 56 (3.3) 0.001 | 201.0(11.0) 0.002<br>2675.3(7.7) 134.0(7.7) 0.002<br>1557.5(3.2) 56.0(3.2) 0.001 |
| mean (sel) Fraily score many (sel) | 2.24 (2.37) | 1.75 (2.05) 0.219 | 1.82 (2.07)<br>0.16 (0.05) | 1.80 (2.06) 0.01 | 1.80 (2.06)<br>0.16 (0.04) | 1.75 (2.05) 0.023<br>2.16 (0.04) 0.033<br>11.81 (5.18) 0.05 | 1.49 (2.09)<br>0.16 (0.05) | 1.04 (1.68)<br>0.15 (0.03) | 0.239 | 1.05 (1.69) 1.04 (1.68) 0.006<br>0.15 (0.04) 0.15 (0.03) 0.002 | 0.15 (0.04) | 1.04 (1.68) 0.007<br>0.15 (0.03) 0.009 | 1.82 (2.16) 1.66 (1.93)<br>0.19 (0.06) 0.19 (0.05)<br>10.94 (4.76) 11.84 (4.89) | 0.078 | 1.71(2.02) 1.67(1.93) 0.019<br>0.19(0.05) 0.19(0.05) 0.014 | 1.66 (1.97) 1.66 (1.93) 0.001<br>0.19 (0.05) 0.19 (0.05) 0.001 |
| Unique generic medicines mean (sd) Unique brand medicines | 11/41 (5.14) | 11.81 (5.18) 0.072 | 11.84 (5.19) | 11.76 (5.13) 0.015 | 12.07 (5.30) | 11.81 (5.18) 0.05 | 0.16 (0.05)<br>10.47 (4.86) | 10.79 (4.77) | 0.066 | 10.71 (4.86) 10.72 (4.74) 0.002 | 10.87 (4.90) | 20.79 (4.77) 0.016 | | 0.187 | 11.72 (4.90) 11.77 (4.85) 0.01 | 11.82 (5.00) 11.84 (4.90) 0.005 |
| mean (sd) Hospitalizations [-90, 0]; n (%) Hospitalizations [-100, 0]; n (%) | 11.54 (5.25)<br>3282 (6.3)<br>4657 (9.5) | 11.92 (5.29) 0.073<br>494 (2.9) 0.166<br>987 (5.7) 0.144<br>3180 (18.4) 0.138 | 11.96 (5.29)<br>457 (3.0)<br>916 (6.0) | 11.88 (5.23) 0.015<br>472 (3.1) 0.006<br>905 (6.0) 0.003 | 12.19 (5.41)<br>1487.1 (3.0)<br>2943.0 (5.9)<br>9804.2 (19.6) | | 10.58 (4.96)<br>1300 (6.3)<br>2102 (10.2)<br>4956 (24.0) | 10.90 (4.86)<br>159 (3.1)<br>108 (5.9) | 0.065<br>0.154<br>0.157 | 10.81 (4.95) 10.83 (4.82) 0.004<br>152 (3.1) 155 (3.1) 0.003<br>202 (5.9) 296 (5.0) 0.005<br>857 (17.3) 894 (18.1) 0.02 | 10.98 (5.03)<br>641.2 (1.2)<br>1237.0 (5.1) | 10.90 (4.85) 0.017<br>159.0 (3.1) 0.005<br>308.0 (5.9) 0.007<br>930.0 (17.9) 0.011 | 11.04 (4.85) 11.98 (4.99)<br>4159 (8.3) 88 (4.3)<br>6322 (12.6) 152 (8.7)<br>12743 (25.5) 252 (20.2) | 0.189<br>0.141<br>0.127 | 11.84 (4.98) 11.90 (4.95) 0.012<br>80 (4.7) 84 (5.0) 0.011<br>142 (8.7) 150 (8.9) 0.006 | 11.95 (5.10) 11.97 (4.99) 0.004<br>2331.1 (4.9) 84.0 (4.8) 0.005<br>4228.7 (8.8) 152.0 (8.8) 0.002<br>9664.9 (20.1) 351.0 (20.2) 0.002 |
| ED visits; n (%) Office visits mean (sd) | 12492 (24.1)<br>4.91 (4.11) | 3180(18.4) 0.318<br>5.37(1.96) 0.31 <sup>3</sup> | 2997 (19.7)<br>5.33 (4.29) | 472 (3.1) 0.006<br>905 (6.0) 0.003<br>2914 (19.2) 0.014<br>5.29 (3.84) 0.009 | 9804.2 (19.6)<br>5.51 (4.76) | | 4956 (24.0)<br>4.74 (3.850 | 932 (17.9)<br>4.99 (1.91) | 0.15 | 857 (27.3) 894 (18.1) 0.02<br>4.96 (4.09) 4.94 (3.72) 0.003 | 3718.9 (18.3)<br>5.05 (4.21) | 930.0 (17.9) 0.011<br>4.99 (3.91) 0.015<br>698.0 (13.5) 0.006 | 4159 (8.3) 84 (4.8)<br>6322 (12.6) 152 (8.7)<br>12743 (25.5) 352 (20.2)<br>654 (7.51) 6.76 (8.72)<br>6607 (12.2) 289 (16.6) | 0.124 | 336 (19.9) 343 (20.3) 0.01<br>6.85 (19.71) 6.66 (8.41) 0.02<br>754 (15.3) 274 (16.7) 0.024 | 9664.9 (20.1) 351.0 (20.2) 0.002<br>6.67 (9.90) 6.75 (8.72) 0.008 |
| Endocrinologist visit; n (%) Cardiologist visit; n (%) Internal medicine/family medicine visits; n (%) | 4849 (9.3)<br>19351 (37.3)<br>45381 (87.4) | 1.75(2.25) 1.15(2.25) | 1639 (10.8)<br>5489 (36.1)<br>13358 (88.0) | 5.79(1.84) 0.000 1509(11.1) 0.011 1509(11.8) 0.011 1509(18.6) 0.000 1519(18.6) 0.000 1519(18.6) 0.000 1519(18.6) 0.000 1519(18.6) 0.000 1517(0.44) 0.000 1517(0.44) 0.000 1517(0.44) 0.000 1517(0.44) 0.000 1517(0.45) 0.000 | 5.51 (4.76)<br>5784.4 (11.6)<br>18494.5 (27.0)<br>44184.3 (88.4) | 1370 0 (37 0) 0.000 | 4.74 (3.89)<br>2155 (30.5)<br>7562 (36.7)<br>17018 (82.6) | 702 (13.5)<br>1829 (35.2)<br>4182 (80.5) | 0.000 0.114 0.117 0.000 0.000 0.001 0.0110 0.001 0.0110 0.001 0.0110 0.001 0.0110 0.001 0.001 0.001 0.001 0.001 0.000 | 646 (13.0) 654 (13.2) 0.005<br>1727 (34.9) 1755 (35.4) 0.012<br>1981 (80.4) 3992 (80.6) 0.006 | 2767.6 (13.6)<br>7222.5 (35.6)<br>16339.0 (80.6) | 698.0 (13.5) 0.005<br>1826.0 (35.2) 0.009<br>4175.0 (80.5) 0.003 | | | 259 [15.3] 274 [16.2] 0.024<br>704 [41.7] 678 [40.1] 0.031<br>1338 [79.2] 1336 [79.1] 0.003 | 7934.4 (16.5) 288.0 (16.6) 0.002<br>19132.4 (39.8) 686.0 (40.1) 0.005<br>18080.5 (79.3) 1375.0 (79.2) 0.003 |
| Electrocardiograms mean (sd) Echocardio | 0.62 (1.42) | 0.56(1.05) 0.051 | 0.56 (1.09) | 0.56 (1.05) 0.001 | 0.57 (1.13) | 0.56 (1.05) 0.011 | 1.08 (3.22) | 0.76 (2.09) | 0.118 | 0.75 (1.90) 0.76 (2.12) 0.009 | 0.77 (1.90) | 0.76 (2.09) 0.009 | 0.85 (2.32) 0.74 (1.87) | 0.02<br>0.056<br>0.015 | 0.76 (1.45) 0.74 (1.89) 0.011 | 0.73 (1.49) 0.74 (1.87) 0.004 |
| mean (sd) HbA1c tests received mean (sd) | 0.18 (0.47) | 0.17 (0.45) 0.026<br>1.42 (0.89) 0.158 | 0.17 (0.45) | 0.17 (0.44) 0.005<br>1.39 (0.82) 0.004 | 0.17 (0.45) | | 0.45 (2.26) | 0.30 (1.36) | 0.081 | 0.29(1.37) 0.30(1.37) 0.009<br>1.30(1.15) 1.30(0.91) 0.002 | 0.30 (1.36) | 0.30(1.36) 0.007 | 0.26 (0.79) 0.27 (1.23)<br>1.37 (1.35) 1.55 (1.12) | 0.015 | 0.28 (0.80) 0.27 (1.24) 0.007<br>1.48 (1.25) 1.54 (1.12) 0.044 | 0.26 (0.97) 0.27 (1.23) 0.013<br>1.54 (2.23) 1.55 (1.12) 0.094 |
| Glucose tests ordered<br>mean (sd)<br>Lipid tests ordered | 0.44 (2.16) | 0.38(1.14) 0.024 | 0.38(0.05) | 0.27(1.14) 0.005 | 1.42 (0.87)<br>0.39 (1.08)<br>0.99 (0.80) | 0.38 (1.14) 0.012 | 2.11 (2.02)<br>0.41 (2.02)<br>0.79 (0.91) | 0.37/1.52) | 0.021 | 0.36(1.36) 0.36(1.56) 0.001 | 0.38(1.24) | 0.37 (1.54) 0.012 | 051(2.86) 055(4.63) | 0.01 | 0.60 (4.58) 0.56 (4.69) 0.009 | 0.54 (3.24) 0.55 (4.63) 0.002 |
| mean (sd) Creatinine tests ordered mean (sd) | 0.89 (0.79) | 0.99 (0.79) 0.127 | 0.97 (0.81) | 0.97 (0.78) 0.001<br>0.03 (0.22) 0.006 | 0.99 (0.80) | | 0.79 (0.91)<br>0.01 (0.28)<br>429 (2.1) | 0.96 (0.85) | 0.198 | 0.95 (0.99) | 0.97 (1.02) | 0.0510.450 0.001<br>0.0510.460 0.001<br>14467.232 0.000<br>4186.0100.77 0.000<br>4186.0100.71 0.000<br>100.0111.8 0.000<br>107.0111.8 0.000<br>107.0111.8 0.000<br>107.0111.9 0.000<br>108.017.9 0.001<br>108.017.9 0.001<br>108.017.9 0.000 | 0.95 (1.08) 1.10 (0.94)<br>0.04 (0.39) 0.04 (0.32) | 0.001<br>0.128<br>0.006<br>0.028<br>0.16<br>0.069<br>0.071<br>0.129<br>0.016 | 1.10 (1.40) 1.09 (0.92) 0.007<br>0.04 (0.44) 0.04 (0.23) 0.006<br>68 (4.0) 59 (4.1) 0.001 | 1.09 (1.80) 1.00 (0.94) 0.008<br>0.04 (0.49) 0.04 (0.32) 0.002 |
| Some mineral density test: $n$ (%)<br>Basic or comprehensive metabolic blood chem test; $n$ (%) | 2143 (4.1)<br>42439 (81.8) | 795 (4.6) 0.024<br>14720 (85.4) 0.098 | 723 (4.8)<br>12899 (85.0) | 707 (4.7) 0.005<br>12885 (84.9) 0.003 | 2362.6 (4.7)<br>42687.0 (85.4) | 0.021 (0.21) 0.002; 178 (0.14 th) 0.0024; 147 (1.0 (18.4) 0.0024; 147 (1.0 (18.4) 0.0024; 147 (1.0 (18.4) 0.0024; 147 (1.0 (18.4) 0.0024; 147 (1.0 (18.4) 0.0024; 148 (18.4) 0.0024; 148 (18.4) 0.0024; 1 | 429 (2.1)<br>14887 (72.2) | 117 (2.3)<br>4193 (80.7) | 0.012 | 107 (2.2) 110 (2.2) 0.004<br>1961 (80.0) 2975 (80.3) 0.006 | 443.5 (2.2)<br>16402.5 (80.9) | 114.0 (2.2) 0.001<br>4186.0 (80.7) 0.005 | 1855 (1.7) 74 (4.2)<br>42664 (85.2) 1573 (90.5) | 0.028 | 68 (4.0) 69 (4.1) 0.003 | 2005.5 (4.2) 74.0 (4.3) 0.004<br>43546.5 (90.7) 1571.0 (90.4) 0.008 |
| Mammoeram: n (%) Pap amear: n (%) PSA: n (%) | 5955 (11.5)<br>5060 (9.7)<br>7083 (13.6) | 2529 (14.7) 0.095<br>2158 (12.5) 0.088<br>2946 (17.1) 0.096<br>802 (4.7) 0.021 | 2182 (14.4)<br>1846 (12.2)<br>2468 (16.3)<br>710 (4.7) | 2180 (14.4) 0.001<br>1851 (12.2) 0.001<br>2484 (16.4) 0.003 | 7354.9 (14.7)<br>6282.3 (12.6)<br>8365.4 (16.7)<br>2376.9 (4.8) | 2529.0 (14.7) 0.001<br>2158.0 (12.5) 0.002<br>2946.0 (17.1) 0.009 | 1798 (8.7)<br>1674 (8.1)<br>3297 (16.0) | 611 (11.8)<br>572 (11.0)<br>1014 (10.9)<br>268 (5.2) | 0.1<br>0.098<br>0.102 | 587 (31.9) 582 (31.8) 0.003<br>542 (30.9) 542 (30.9) 0.003<br>974 (30.7) 986 (39.9) 0.006 | 2433.6 (12.0)<br>2251.7 (13.1)<br>4042.9 (19.9) | 4186.0 (80.7) 0.005<br>630.0 (11.8) 0.008<br>571.0 (11.0) 0.001<br>1024.0 (12.9) 0.001<br>258.0 (5.2) 0.001 | 42664 (85.2) 1572 (90.5)<br>429 (88) 188 (10.8)<br>4447 (8.3) 188 (10.4)<br>4789 (13.6) 318 (18.3)<br>312 (14.3) 72 (4.3) | 0.059 | 187 (11.1) 183 (10.8) 0.008<br>184 (10.9) 175 (10.4) 0.017<br>329 (19.5) 304 (18.0) 0.018 | 5277.1(10.0) 187.0(10.0) 0.001<br>5007.8(10.4) 180.0(10.4) 0.002<br>875.9(18.7) 197.0(18.2) 0.002<br>1981.7(4.1) 71.0(4.1) 0.002 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual<br>colonoscopy: n (%) Flu vaccine/Pneumococcal vaccine: n (%) | 2189 (4.2)<br>11536 (22.2) | 802 (4.7) 0.021<br>3658 (21.2) 0.024 | 710 (4.7)<br>3237 (21.3) | 691 (4.6) 0.006<br>3233 (21.3) 0.001 | 2375.9 (4.8)<br>10812.2 (21.6) | 2158.0 (12.5) 0.002<br>2946.0 (17.1) 0.009<br>802.0 (4.7) 0.005<br>9658.0 (22.2) 0.01<br>2884.0 (35.7) 0.007 | 14887 (72.2)<br>1298 (8.7)<br>1674 (8.1)<br>1297 (16.0)<br>965 (4.7)<br>4244 (20.4)<br>4652 (19.7) | 268 (5.2)<br>909 (17.5) | 0.022 | 246 (5.0) 253 (5.1) 0.006<br>868 (17.5) 872 (17.6) 0.002<br>1126 (22.7) 1134 (22.9) 0.004 | 1053.6 (5.2)<br>3570.6 (17.6)<br>4672.0 (23.0) | 268.0 (5.2) 0.001<br>909.0 (17.5) 0.002<br>1181.0 (22.8) 0.006 | 1912 (3.8) 72 (4.1)<br>23315 (42.4) 820 (47.2)<br>9227 (38.4) 592 (34.0) | 0.016 | \$22 (16.5) \$2.50 ( | 1983.7 (4.1) 71.0 (4.1) 0.002<br>22520.1 (46.9) 819.0 (47.2) 0.005 |
| Telemedicine: n (%)<br>Stable Aneira: n (%)<br>Race | 8332 (16.3)<br>3847 (7.4) | 2884 (16.7) 0.018<br>1364 (7.9) 0.019 | 2544 (16.8)<br>1159 (7.6) | 2515 (16.6) 0.005<br>1180 (7.8) 0.005 | 8235.7 (16.5)<br>1976.1 (8.0) | 2884.0 (16.7) 0.007<br>1364.0 (7.9) 0.002 | 4062 (19.7)<br>1274 (6.2) | 1185 (22.8)<br>348 (6.7) | 0.076 | 1126 (22.7) 1114 (22.9) 0.006<br>337 (6.6) 329 (6.6) 0.006 | 4672.0 (23.0)<br>1417.6 (7.0) | 1183.0(22.8) 0.005<br>348.0(6.7) 0.011 | 9227 (18.4) 592 (24.0)<br>2554 (5.1) 100 (5.8) | 0.361<br>0.029<br>0.156 | 586 (24.7) 569 (23.7) 0.021<br>92 (5.4) 94 (5.6) 0.005<br>0.061 | 1696.1 (14.3) 591.0 (14.0) 0.007<br>2711.7 (5.6) 100.0 (5.8) 0.005 |
| White: n (%)<br>Asian: n (%)<br>Black: n (%) | | | | | | | | | Ħ | | | | 37384 (74.3) 1389 (79.5)<br>2632 (5.2) 74 (4.3)<br>5428 (20.8) 147 (8.5) | | 1341 (79.3) 1247 (79.7)<br>63 (1.7) 72 (4.3)<br>140 (8.3) 144 (8.5) | 28310.2 (79.8) 1387.0 (79.9)<br>2053.2 (4.3) 74.0 (4.3)<br>4075.4 (E.5) 147.0 (E.5)<br>1010.8 (2.1) 27.0 (2.3) |
| Hispanic: n (%)<br>Unknown/Missina/Other: n (%)<br>Dual status for medicare: n (%) | | | | | | | | | | | | | 2019 (4.1) 37 (2.1)<br>2794 (5.6) 92 (5.3)<br>13368 (26.7) 447 (25.7) | 0.021 | 34 (2.0) 37 (2.2)<br>112 (6.6) 50 (5.3)<br>444 (26.3) 438 (25.9) 0.008 | 1010.8 (2.1) 37.0 (2.1)<br>2574.3 (5.4) 92.0 (5.3)<br>12243.8 (25.5) 447.0 (25.7) 0.005 |

| Covariates | Source |
|---|---|
| Region | If region not available, from State, https://www2.census.gov/geo/pdfs/maps-data/maps/reference/us_regdiv.pdf |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://hcup-us.ahrq.gov/datainnovations/ICD- |
| Drug abuse or dependence | 10CaseStudyonOpioid-RelatedIPStays042417.pdf, https://stacks.cdc.gov/view/cdc/59394, https://pubmed.ncbi.nlm.nih.gov/34134872/ |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, |
| Alcohol abuse or dependence | https://espace.curtin.edu.au/bitstream/handle/20.500.11937/34117/19233_downloaded_stream_325.pdf?isAllowed=y&sequence=2 |
| Underweight or normal weight | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Overweight | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Obese | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Severe Obese | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Unspecified obesity | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| | Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic- |
| | packages/browse?at=refs%2Fheads%2Fcder_mpl2p_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic- |
| | packages/browse?at=refs%2Fheads%2Fcder_sir_wp002, https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| Smoking | https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/ |
| Diabetic retinopathy | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Diabetic neuropathy | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Diabetic nephropathy | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| | https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, https://www.health.mil/Reference- |
| | Center/Publications/2016/03/01/Diabetes-Mellitus, http://www.icd9data.com/2014/Volume1/240-279/249-259/250/default.htm, |
| Diabetes with unspecified complication | https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11- |
| Diabetes with other ophthalmic manifestations | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion |
| | Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, |
| | https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus, http://www.icd9data.com/2014/Volume1/240- |
| Diabetes with peripheral circulatory disorders | 279/249-259/250/default.htm, https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11- |
| Diabetic foot + Lower extremity amputation | Investigator review of codes based on: (modified codes) https://pubmed.ncbi.nlm.nih.gov/36102675/ |
| Skin infections | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ , ICD9 to ICD10 conversion |
| For add a destruction | Investigator review of codes based on: the paper then used ICD9/ICD10 website to expand it, |
| Erectile dysfunction | https://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-N53/N52-, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/ |
| Hypoglycemia | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| | Investigator review of codes based on: |
| | Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| | DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/, https://pubmed.ncbi.nlm.nih.gov/38262528/ |
| Hyperglycemia, DKA, HONK | HONK: https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnovation/DEF/DKA.pdf |

Hypertension

Hyperlipidemia

Atrial fibrillation
Acute MI
Old MI
Coronary atherosclerosis
History of CABG/PTCA
Previous cardiac procedure
Cerebrovascular procedure
Ischemic stroke
PVD diagnosis or surgery
CKD stage 3-4

Other cardiac dysrhythmia

Cardiomyopathy

Valve disorders COPD

Asthma

Obstructive sleep apnea Pneumonia CKD 1-2 Acute renal disease (AKI)

Nephrotic syndrome

Hypertensive nephropathy

Other renal conditions

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4910677/

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

 $Modified\ codes\ based\ on\ inclusion\ criteria,\ here\ we\ implement\ any\ care\ setting,\ any\ diagnosis\ position$ 

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://www.health.ny.gov/health care/medicaid/redesign/dsrip/vbp library/docs/arrblk.pdf,

https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology1.pdf, ICD9 to ICD10 conversion

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

https://pubmed.ncbi.nlm.nih.gov/38440888/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp009

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW algorithm (any care setting, any diagnosis position)

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

 $Investigator\ review\ of\ codes\ based\ on:\ https://nccd.cdc.gov/ckd/Methods.aspx? Qnum=Q637,\ https://www.cms.gov/icd10m/FY2024-properties and the properties of\ codes\ based\ on:\ https://nccd.cdc.gov/ckd/Methods.aspx? Qnum=Q637,\ https://www.cms.gov/icd10m/FY2024-properties and the properties of\ codes\ based\ on:\ https://nccd.cdc.gov/ckd/Methods.aspx? Qnum=Q637,\ https://www.cms.gov/icd10m/FY2024-properties and the properties of\ codes\ based\ on:\ https://nccd.cdc.gov/ckd/Methods.aspx? Qnum=Q637,\ https://www.cms.gov/icd10m/FY2024-properties and the properties of\ codes\ based\ on:\ https://nccd.cdc.gov/ckd/Methods.aspx? Qnum=Q637,\ https://www.cms.gov/icd10m/FY2024-properties and the properties an$ 

nprmversion41.0-fullcode-cms/fullcode\_cms/P2401.html Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637,

https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e29ab67-7a7d-4621-9af3-

81bd071bbc67/mmc1.pdf, https://www.icd10data.com/ICD10CM/Codes/I00-I99

Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637,

https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion

Liver disease Hypothyroidism Osteoarthritis **Fractures** Falls Osteoporosis Depression Anxiety Sleep disorder Dementia Delirium COVID Number of antidiabetic drugs ACE + ARBs Thiazide Beta blockers Calcium channel blockers Loop diuretics Other diuretics Nitrates HF drugs (Digoxin + Entresto + Ivabadrine) Anti-arrhythmics

COPD/asthma meds

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder sir wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, Modified algorightm from https://pubmed.ncbi.nlm.nih.gov/34256144/, Modified CCW algorithm Modified CCW algorithm Modified CCW algorithm https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder mpl2p wp009 https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp010 https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, CCW Algorithms https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-and-diagnostic-codes-3014779 https://pubmed.ncbi.nlm.nih.gov/35043165/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder mpl2p wp015 https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/ https://pubmed.ncbi.nlm.nih.gov/34913208/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/ Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5256065/, https://www.drugs.com/drug-class/antidiabetic-agents.html, https://www.ncbi.nlm.nih.gov/books/NBK279141/ Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using class I and class II as class 2 is beta blockers and class 4 is calcium channel blockers)

Investigator review of codes based on: https://www.copdfoundation.org/Learn-More/I-am-a-Person-with-COPD/Treatments-

Medications.aspx, https://getasthmahelp.org/medications-list.aspx

Statins

Other lipid-lowering drugs Antiplatelet agents

Oral anticoagulants NSAIDs

Oral corticosteroids
Bisphosphonates

Opioids

Anti-depressants
Gabapentnoids

Benzodiazepines Anxiolytics/hypnotics

Dementia meds

Office visits

**Endocrinologist visit** 

Cardiologist visits

Internal medicine/family medicine visits

Electrocardiograms

Echocardio
HbA1c tests received
Glucose tests ordered
Lipid tests ordered
Creatinine tests ordered

Investigator review of codes based on: https://www.drugs.com, https://www.heart.org/en/health-topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-medications

Investigator review of codes based on: https://www.drugs.com, https://www.heart.org/en/health-topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-medications

Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK537062/

Investigator review of codes based on: https://www.drugs.com, https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559

Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK547742/

Investigator review of codes based on: https://www.arugs.com, https://www.aaaai.org/tools-for-the-public/drug-guide/oral-

corticosteroid-medications

Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK470248/

Investigator review of codes based on: https://www.drugs.com,

C%20hydrocodone%2C

Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK538182/

GABAPENTIN, PREGABALIN

Investigator review of codes based on: https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-06/Benzodiazepenes-

2020.pdf, https://www.ncbi.nlm.nih.gov/books/NBK470159/

Investigator review of codes based on: https://www.drugs.com

Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/,

https://go.drugbank.com/drugs/DB00382

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document-pfs-payment-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document-pfs-payment-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document-office-outpatient-evaluation-and-management-visit-code-g2211.pdf, https://www.cms.gov/files/document-office-g2211.pdf, https://www.cms.gov/files/d

management-em-visits-fact-sheet.pdf

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Certification/Medicare Provider Sup Enroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-and-downloads/taxonomy.pdf, https://www.pdf, https://ww

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Certification/Medicare Provider Sup Enroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-and-downloads/taxonomy.pdf, https://www.pdf, https://ww

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf

Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-and-

Investigator review of codes based on: https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleId=57326, https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/, https://www.aapc.com/codes/coding-newsletters/my-cardiology-

coding-alert/cpt-answer-5-common-ecg-coding-questions-175952-article

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/,

https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleid=56625&ver=27&, https://www.medicalbillgurus.com/echocardiogram-cpt-code/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/

Investigator review of codes based on: https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleid=59040&ver=4,

https://static.cigna.com/assets/chcp/pdf/coveragePolicies/medical/mm 0300 coveragepositioncriteria bone mineral density measur

Bone mineral density test ement.pd

Basic or comprehensive metabolic blood chem test

Telemedicine

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder sir wp002, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleid=56448&ver=16&bc=0, http://www.icd9data.com/2012/Volume1/V01-V91/V70-

Mammogram V82/V76/default.htm

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder sir wp002, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V72/default.htm,

Pap smear http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

PSA packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002 packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002 packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-coverage-

Investigator review of codes, Flu vaccine/Pnemococcal vaccine database/view/article.aspx?articleId=54767&DocID=A54767

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/, https://www.cms.gov/newsroom/fact-

sheets/medicare-telemedicine-health-care-provider-fact-sheet, https://www.aafp.org/family-physician/practice-and-career/getting-

paid/coding/coding-telehealth-audio-virtual-digital-visits.html

Stable Angina Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://www.cms.gov/medicare-medicaid-coordination/medicare-and-medicaid-

DUAL status for medicare coordination/medicare-medicaid-coordination-office/downloads/mmco dualeligibledefinition.pdf

ED visit (Medicare) Revenue center codes: 0450, 0451, 0452, 0456, 0459, 0981; Place of service: 23

ED visit (Optum) Place of service: 23

Service sub-category codes: 10120, 10220, 10320, 10420, 10520, 12220, 20120, 20220, 21120, 21220, 22120, 22320, 30120, 30220,

ED visit (Marketscan) 30320, 30420, 30520, 30620, 31120, 31220, 31320, 31420, 31520, 31620; Place of service: 23

Hernia (negative control) https://pmc.ncbi.nlm.nih.gov/articles/PMC11320168/#note-ZOI240844-1-s

Lumbar radiculopathy (negative control) https://pmc.ncbi.nlm.nih.gov/articles/PMC11320168/#note-ZOI240844-1-s

https://pubmed.ncbi.nlm.nih.gov/32828874/, https://pubmed.ncbi.nlm.nih.gov/29433851/, https://pubmed.ncbi.nlm.nih.gov/29075781/, https://pubmed.ncbi.nlm.nih.gov/34935591/ and

Cataract surgery (negative control) https://pubmed.ncbi.nlm.nih.gov/23993357/ and department ICD-9 to ICD-10 conversion


PATIENT DOCUMENTED AS TOBACCO USER AND RECEIVED TOBACCO
CESSATION INTERVENTION (MUST INCLUDE AT LEAST ONE OF THE FOLLOWING:
ADVICE GIVEN TO QUIT SMOKING OR TOBACCO USE, COUNSELING ON THE
BENEFITS OF QUITTING SMOKING OR TOBACCO USE, ASSISTANCE WITH OR
REFERRAL TO EXTERNAL SMOKING OR TOBACCO USE, SASISTANCE WITH OR
REPERAL TO EXTERNAL SMOKING OR TOBACCO USE, ASSISTANCE WITH OR
REPORCEAMS, OR CLIBERNT ENROLL MENT IN SMOKING OR TOBACCO USE.


TYPE 1 DIABETES MELLITUS WITH PROLIFERATIVE DIABETIC RETINOPATHY


DILATION OF RIGHT COMMON CAROTID ARTERY, BIFURCATION, WITH THREE


UNSPECIFIED CHRONIC BRONCHITIS

COPD

J42

DX


UNSPECIFIED DISPLACED FRACTURE OF SURGICAL NECK OF UNSPECIFIED


-PART FRACTURE OF SURGICAL NECK OF RIGHT HUMERUS, SUBSEQUENT


SALTER-HARRIS TYPE IV PHYSEAL FRACTURE OF LOWER END OF RADIUS,


DISPLACED FRACTURE (AVULSION) OF LATERAL EPICONDYLE OF RIGHT


NONDISPLACED FRACTURE (AVULSION) OF LATERAL EPICONDYLE OF RIGHT


DISPLACED FRACTURE (AVULSION) OF MEDIAL EPICONDYLE OF RIGHT


NONDISPLACED FRACTURE OF OLECRANON PROCESS WITHOUT


DISPLACED FRACTURE OF OLECRANON PROCESS WITH INTRAARTICULAR


OTHER FRACTURE OF UPPER END OF LEFT RADIUS, SUBSEQUENT ENCOUNTER


DISPLACED COMMINUTED FRACTURE OF SHAFT OF ULNA, RIGHT ARM,


NONDISPLACED COMMINUTED FRACTURE OF SHAFT OF ULNA, RIGHT ARM,


UNSPECIFIED FRACTURE OF SHAFT OF RIGHT RADIUS, SUBSEQUENT


NONDISPLACED TRANSVERSE FRACTURE OF SHAFT OF LEFT RADIUS,


DISPLACED SPIRAL FRACTURE OF SHAFT OF RADIUS, LEFT ARM, SUBSEQUENT


DISPLACED COMMINUTED FRACTURE OF SHAFT OF RADIUS, UNSPECIFIED


DISPLACED SEGMENTAL FRACTURE OF SHAFT OF RADIUS, RIGHT ARM,


NONDISPLACED SEGMENTAL FRACTURE OF SHAFT OF RADIUS, RIGHT ARM,


DISPLACED FRACTURE OF UNSPECIFIED RADIAL STYLOID PROCESS,


OTHER EXTRAARTICULAR FRACTURE OF LOWER END OF LEFT RADIUS,


OTHER INTRAARTICULAR FRACTURE OF LOWER END OF LEFT RADIUS,


NONDISPLACED FRACTURE OF UNSPECIFIED ULNA STYLOID PROCESS,


SALTER-HARRIS TYPE I PHYSEAL FRACTURE OF LOWER END OF ULNA, RIGHT


SALTER-HARRIS TYPE IV PHYSEAL FRACTURE OF LOWER END OF ULNA, RIGHT


SALTER-HARRIS TYPE IV PHYSEAL FRACTURE OF LOWER END OF ULNA,


SALTER-HARRIS TYPE I PHYSEAL FRACTURE OF UPPER END OF RADIUS,


SALTER-HARRIS TYPE III PHYSEAL FRACTURE OF UPPER END OF RADIUS, RIGHT


SALTER-HARRIS TYPE III PHYSEAL FRACTURE OF UPPER END OF RADIUS,


SALTER-HARRIS TYPE IV PHYSEAL FRACTURE OF UPPER END OF RADIUS, LEFT


SALTER-HARRIS TYPE II PHYSEAL FRACTURE OF LOWER END OF RADIUS, LEFT


SALTER-HARRIS TYPE I PHYSEAL FRACTURE OF LOWER END OF LEFT FEMUR-


SALTER-HARRIS TYPE III PHYSEAL FRACTURE OF LOWER END OF LEFT FEMUR,


UNSPECIFIED FRACTURE OF HEAD OF RIGHT FEMUR, SUBSEQUENT


DISPLACED ARTICULAR FRACTURE OF HEAD OF UNSPECIFIED FEMUR,


NONDISPLACED ARTICULAR FRACTURE OF HEAD OF UNSPECIFIED FEMUR,


OTHER FRACTURE OF HEAD AND NECK OF LEFT FEMUR, SUBSEQUENT


DISPLACED FRACTURE OF LESSER TROCHANTER OF LEFT FEMUR, SUBSEQUENT


DISPLACED FRACTURE OF LESSER TROCHANTER OF UNSPECIFIED FEMUR,


NONDISPLACED INTERTROCHANTERIC FRACTURE OF UNSPECIFIED FEMUR,


DISPLACED SUBTROCHANTERIC FRACTURE OF UNSPECIFIED FEMUR,


NONDISPLACED SUBTROCHANTERIC FRACTURE OF RIGHT FEMUR,


NONDISPLACED SUBTROCHANTERIC FRACTURE OF UNSPECIFIED FEMUR,


DISPLACED TRANSVERSE FRACTURE OF SHAFT OF LEFT FEMUR, SUBSEQUENT


NONDISPLACED TRANSVERSE FRACTURE OF SHAFT OF LEFT FEMUR,


NONDISPLACED OBLIQUE FRACTURE OF SHAFT OF LEFT FEMUR, SUBSEQUENT


DISPLACED COMMINUTED FRACTURE OF SHAFT OF LEFT FEMUR, SUBSEQUENT


NONDISPLACED COMMINUTED FRACTURE OF SHAFT OF RIGHT FEMUR,


NONDISPLACED COMMINUTED FRACTURE OF SHAFT OF LEFT FEMUR,


NONDISPLACED SEGMENTAL FRACTURE OF SHAFT OF LEFT FEMUR,


UNSPECIFIED FRACTURE OF LOWER END OF UNSPECIFIED FEMUR,


DISPLACED UNSPECIFIED CONDYLE FRACTURE OF LOWER END OF RIGHT


DISPLACED UNSPECIFIED CONDYLE FRACTURE OF LOWER END OF


DISPLACED FRACTURE OF LATERAL CONDYLE OF LEFT FEMUR, SUBSEQUENT


NONDISPLACED FRACTURE OF MEDIAL CONDYLE OF RIGHT FEMUR,


DISPLACED FRACTURE OF LOWER EPIPHYSIS (SEPARATION) OF UNSPECIFIED


NONDISPLACED FRACTURE OF LOWER EPIPHYSIS (SEPARATION) OF LEFT


DISPLACED SUPRACONDYLAR FRACTURE WITHOUT INTRACONDYLAR


DISPLACED SUPRACONDYLAR FRACTURE WITHOUT INTRACONDYLAR


NONDISPLACED SUPRACONDYLAR FRACTURE WITHOUT INTRACONDYLAR


NONDISPLACED SUPRACONDYLAR FRACTURE WITHOUT INTRACONDYLAR


NONDISPLACED SUPRACONDYLAR FRACTURE WITHOUT INTRACONDYLAR


DISPLACED SUPRACONDYLAR FRACTURE WITH INTRACONDYLAR EXTENSION


| MUR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INE HEALING TURE WITH INTRACONDYLAR |
|---|
| MUR, SUBSEQUENT ENCOUNTER FOR<br>ING<br>TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR<br>INE HEALING |
| MUR, SUBSEQUENT ENCOUNTER FOR<br>ING<br>TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR<br>INE HEALING |
| ING<br>TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR<br>INE HEALING |
| TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR<br>INE HEALING |
| MUR, SUBSEQUENT ENCOUNTER FOR<br>INE HEALING |
| INE HEALING |
| MUR, SUBSEQUENT ENCOUNTER FOR |
| /ITH ROUTINE HEALING |
| TURE WITH INTRACONDYLAR |
| MUR, SUBSEQUENT ENCOUNTER FOR |
| ING |
| TURE WITH INTRACONDYLAR |
| MUR, SUBSEQUENT ENCOUNTER FOR |
| YED HEALING |
| TURE WITH INTRACONDYLAR |
| MUR, SUBSEQUENT ENCOUNTER FOR |
| /ITH DELAYED HEALING |
| TURE WITH INTRACONDYLAR |
| MUR, SUBSEQUENT ENCOUNTER FOR |
| THE WITH INTERCONDULAR |
| TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR |
| JNION |
| TURE WITH INTRACONDYLAR |
| MUR, SUBSEQUENT ENCOUNTER FOR |
| /ITH NONUNION |
| TURE WITH INTRACONDYLAR |
| MUR, SUBSEQUENT ENCOUNTER FOR |
| mon, sobsequent encountent on |
| , |
| TURE WITH INTRACONDYLAR |
| , |
| TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR<br>INION |
| TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR<br>INION<br>TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR<br>MUR, SUBSEQUENT ENCOUNTER FOR<br>INION |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR JINION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR JITH MALUNION |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR JINION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR //TH MALUNION TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR JINION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR JITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING ING SUBSEQUENT ENCOUNTER FOR INE HEALING |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR I/ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING IUR, SUBSEQUENT ENCOUNTER FOR INE HEALING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR INE HEALING |
| TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR INION TURE WITH INTRACONDYLAR MUR, SUBSEQUENT ENCOUNTER FOR ITH MALUNION TURE WITH INTRACONDYLAR MUR, SEQUELA TURE WITH INTRACONDYLAR UR TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR CLOSED TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, INITIAL ENCOUNTER FOR OPEN TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING TURE WITH INTRACONDYLAR UR, SUBSEQUENT ENCOUNTER FOR ING ING SUBSEQUENT ENCOUNTER FOR INE HEALING |

NONDISPLACED SUPRACONDYLAR FRACTURE WITH INTRACONDYLAR


NONDISPLACED SUPRACONDYLAR FRACTURE WITH INTRACONDYLAR


NONDISPLACED SUPRACONDYLAR FRACTURE WITH INTRACONDYLAR


UNSTABLE BURST FRACTURE OF T5-T6 VERTEBRA, SUBSEQUENT ENCOUNTER


WEDGE COMPRESSION FRACTURE OF T7-T8 VERTEBRA, INITIAL ENCOUNTER


DAPAGLIFLOZIN


IRBESARTAN/HYDROCHLOROT


Emergency Room

FACE WITH THE PATIENT AND/OR FAMILY.

OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF A NEW PATIENT, WHICH REQUIRES THESE 3 KEY COMPONENTS: A PROBLEM FOCUSED HISTORY; A PROBLEM FOCUSED EXAMINATION; STRAIGHTFORWARD MEDICAL DECISION MAKING. COUNSELING AND/OR COORDINATION OF CARE WITH OTHER PHYSICIANS, OTHER QUALIFIED HEALTH CARE PROFESSIONALS, OR AGENCIES ARE PROVIDED CONSISTENT WITH THE NATURE OF THE PROBLEM(S) AND THE PATIENT'S AND/OR FAMILY'S NEEDS. USUALLY, THE PRESENTING PROBLEM(S) ARE SELF LIMITED OR MINOR. TYPICALLY, 10 MINUTES ARE SPENT FACE-TO-


| | | Provider category |
|---|---|---|
| Endocrinologist visit | 1824 | code |
| | | Provider category |
| Endocrinologist visit | 1959 | code<br>Provider category |
| Endocrinologist visit | 2860 | code |
| | | Provider category |
| Endocrinologist visit | 3589 | code |
| Endocrinologist visit | 5775 | Provider category<br>code |
| - | | Provider category |
| Endocrinologist visit | 5853 | code |
| Endocrinologist visit | 207RE0101X | NUCC Taxonomy<br>Code 1 |
| S . | | NUCC Taxonomy |
| Endocrinologist visit | 207RE0101X | Code 2 |
| Cardiologist visit | 0400 | Provider category<br>code |
| | | Provider category |
| Cardiologist visit | 0401 | code |
| Cardiologist visit | 0402 | Provider category<br>code |
| | | Provider category |
| Cardiologist visit | 0403 | code |
| Cardiologist visit | 0404 | Provider category<br>code |
| | | Provider category |
| Cardiologist visit | 0405 | code |
| Cardiologist visit | 0407 | Provider category<br>code |
| | | Provider category |
| Cardiologist visit | 0408 | code |
| Cardiologist visit | 0409 | Provider category code |
| Car are registrist | 0.03 | Provider category |
| Cardiologist visit | 0410 | code |
| Cardiologist visit | 0411 | Provider category<br>code |
| Car aronograf visit | 0411 | Provider category |
| Cardiologist visit | 0412 | code |
| Cardiologist visit | 0416 | Provider category<br>code |
| Car are registrist | 0.120 | Provider category |
| Cardiologist visit | 1108 | code |
| Cardiologist visit | 1123 | Provider category<br>code |
| Car are registrist | 1123 | Provider category |
| Cardiologist visit | 1135 | code |
| Cardiologist visit | 1162 | Provider category<br>code |
| Car aronograf visit | 1102 | Provider category |
| Cardiologist visit | 1212 | code |
| Cardiologist visit | 1582 | Provider category<br>code |
| Car are registrist | 1302 | Provider category |
| Cardiologist visit | 1629 | code |
| Cardiologist visit | 1728 | Provider category<br>code |
| and the state of t | | Provider category |
| Cardiologist visit | 1856 | code |
| Cardiologist visit | 1947 | Provider category<br>code |
| | <del></del> | |

| Cardiologist visit | 2653 | Provider category code |
|---|---|---|
| Cardiologist visit | 2810 | Provider category code |
| Cardiologist visit | 3073 | Provider category code |
| Cardiologist visit | 3137 | Provider category code |
| Cardiologist visit | 3249 | Provider category code |
| Cardiologist visit | 3534 | Provider category code |
| Cardiologist visit | 4113 | Provider category code |
| Cardiologist visit | 4163 | Provider category code |
| Cardiologist visit | 4622 | Provider category code |
| Cardiologist visit | 4644 | Provider category code |
| Cardiologist visit | 5726 | Provider category code |
| Cardiologist visit | 5742 | Provider category code |
| Cardiologist visit | 5761 | Provider category code |
| Cardiologist visit | 5771 | Provider category code |
| Cardiologist visit | 6593 | Provider category code |
| Cardiologist visit | 6616 | Provider category code |
| Cardiologist visit | 6887 | Provider category code |
| Cardiologist visit | 7034 | Provider category code |
| Cardiologist visit | 7749 | Provider category code |
| Cardiologist visit | 207RC0000X | NUCC Taxonomy<br>Code 1<br>NUCC Taxonomy |
| Cardiologist visit | 207RC0000X | Code 2 |
| Internal medicine/family medicine visit | 0334 | Provider category<br>code<br>Provider category |
| Internal medicine/family medicine visit | 0335 | code<br>Provider category |
| Internal medicine/family medicine visit | 0336 | code Provider category |
| Internal medicine/family medicine visit | 0337 | code<br>Provider category |
| Internal medicine/family medicine visit | 0338 | code<br>Provider category |
| Internal medicine/family medicine visit | 0339 | code Provider category |
| Internal medicine/family medicine visit | 0340 | code<br>Provider category |
| Internal medicine/family medicine visit | 0341 | code<br>Provider category |
| Internal medicine/family medicine visit | 0342 | code<br>Provider category |
| Internal medicine/family medicine visit | 1133 | code |

| | | Provider category |
|------------------------------------------|------|---------------------------|
| Internal medicine/family medicine visit | 1419 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 1673 | code |
| Internal medicine/family medicine visit | 1607 | Provider category code |
| Internal medicine/family medicine visit | 1097 | Provider category |
| Internal medicine/family medicine visit | 1860 | code |
| _ | | Provider category |
| Internal medicine/family medicine visit | 1864 | code |
| Internal medicine/family medicine visit | 2050 | Provider category code |
| , | | Provider category |
| Internal medicine/family medicine visit | 2280 | code |
| Internal medicine/family medicine visit | 2302 | Provider category |
| Internal medicine/family medicine visit | 2302 | code<br>Provider category |
| Internal medicine/family medicine visit | 2313 | code |
| _ | | Provider category |
| Internal medicine/family medicine visit | 2314 | Code |
| Internal medicine/family medicine visit | 2373 | Provider category code |
| , | | Provider category |
| Internal medicine/family medicine visit | 2610 | code |
| Internal medicine/family medicine visit | 2042 | Provider category code |
| internal medicine/lamily medicine visit | 2042 | Provider category |
| Internal medicine/family medicine visit | 3268 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 3/55 | code<br>Provider category |
| Internal medicine/family medicine visit | 4641 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 4876 | code |
| Internal medicine/family medicine visit | 5724 | Provider category code |
| internal medicine, family medicine visit | 3724 | Provider category |
| Internal medicine/family medicine visit | 5736 | code |
| lakana laa disia Maasilaa adisia adisia | 5020 | Provider category |
| Internal medicine/family medicine visit | 5829 | code<br>Provider category |
| Internal medicine/family medicine visit | 5991 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 5998 | code |
| Internal medicine/family medicine visit | 0308 | Provider category<br>code |
| , | | Provider category |
| Internal medicine/family medicine visit | 0311 | code |
| Internal medicine /family medicine visit | 0212 | Provider category |
| Internal medicine/family medicine visit | 0312 | code<br>Provider category |
| Internal medicine/family medicine visit | 0313 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 0314 | code |
| Internal medicine/family medicine visit | 0316 | Provider category code |
| | - | Provider category |
| Internal medicine/family medicine visit | 0317 | code |
| Internal medicine/family medicine visit | 0318 | Provider category<br>code |
| memai medicine/ianiny medicine visit | 0310 | Provider category |
| Internal medicine/family medicine visit | 0319 | code |

| | | Provider category |
|------------------------------------------|------|---------------------------|
| Internal medicine/family medicine visit | 0326 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 0327 | code |
| Internal medicine/family medicine visit | 0220 | Provider category code |
| internal medicine/lamily medicine visit | 0329 | Provider category |
| Internal medicine/family medicine visit | 0330 | code |
| _ | | Provider category |
| Internal medicine/family medicine visit | 0331 | code |
| Internal medicine/family medicine visit | 0332 | Provider category code |
| , | | Provider category |
| Internal medicine/family medicine visit | 0333 | code |
| Internal medicine/family medicine visit | 1046 | Provider category |
| Internal medicine/family medicine visit | 1046 | code<br>Provider category |
| Internal medicine/family medicine visit | 1113 | code |
| _ | | Provider category |
| Internal medicine/family medicine visit | 1127 | Code |
| Internal medicine/family medicine visit | 1643 | Provider category code |
| , | | Provider category |
| Internal medicine/family medicine visit | 1646 | code |
| Internal medicine/family medicine visit | 1694 | Provider category code |
| internal medicine/lamily medicine visit | 1694 | Provider category |
| Internal medicine/family medicine visit | 1721 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 1/85 | code<br>Provider category |
| Internal medicine/family medicine visit | 1832 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 1865 | code |
| Internal medicine/family medicine visit | 1927 | Provider category code |
| internal medicine, family medicine visit | 1327 | Provider category |
| Internal medicine/family medicine visit | 2068 | code |
| lakana laa disia Maasilaa adisia adisia | 2100 | Provider category |
| Internal medicine/family medicine visit | 2189 | code<br>Provider category |
| Internal medicine/family medicine visit | 2219 | code |
| | | Provider category |
| Internal medicine/family medicine visit | 2233 | code |
| Internal medicine/family medicine visit | 2286 | Provider category<br>code |
| , | | Provider category |
| Internal medicine/family medicine visit | 2340 | code |
| Internal medicine /family medicine visit | 2254 | Provider category |
| Internal medicine/family medicine visit | 2354 | code<br>Provider category |
| Internal medicine/family medicine visit | 2378 | code |
| _ | | Provider category |
| Internal medicine/family medicine visit | 2403 | code |
| Internal medicine/family medicine visit | 2574 | Provider category<br>code |
| | | Provider category |
| Internal medicine/family medicine visit | 2614 | code |
| Internal medicine/family medicine visit | 2615 | Provider category<br>code |
| memai medicine/ianiny medicine visit | 2013 | Provider category |
| Internal medicine/family medicine visit | 2628 | code |

| | | Provider category |
|---|---|---|
| Internal medicine/family medicine visit | 2644 | code |
| Internal medicine/family medicine visit | 2790 | Provider category code |
| Internal medicine/family medicine visit | 2835 | Provider category code |
| Internal medicine/family medicine visit | 2978 | Provider category code |
| Internal medicine/family medicine visit | 2996 | Provider category code |
| Internal medicine/family medicine visit | 3122 | Provider category code |
| Internal medicine/family medicine visit | 3777 | Provider category code |
| Internal medicine/family medicine visit | 3787 | Provider category code |
| Internal medicine/family medicine visit | 4362 | Provider category<br>code |
| Internal medicine/family medicine visit | 4645 | Provider category<br>code<br>Provider category |
| Internal medicine/family medicine visit | 4648 | code Provider category |
| Internal medicine/family medicine visit | 5063 | code Provider category |
| Internal medicine/family medicine visit | 5683 | code Provider category |
| Internal medicine/family medicine visit | 5696 | code Provider category |
| Internal medicine/family medicine visit | 5706 | code Provider category |
| Internal medicine/family medicine visit | 5732 | code Provider category |
| Internal medicine/family medicine visit | 5774 | code Provider category |
| Internal medicine/family medicine visit | 5781 | code<br>Provider category |
| Internal medicine/family medicine visit | 5994 | code Provider category |
| Internal medicine/family medicine visit | 6000 | code<br>Provider category |
| Internal medicine/family medicine visit | 7017 | code<br>Provider category |
| Internal medicine/family medicine visit | 7592 | code<br>Provider category |
| Internal medicine/family medicine visit | 7777 | code<br>Provider category |
| Internal medicine/family medicine visit | 7792 | code<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207Q00000X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QA0000X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QH0002X | Code 1 |


| COMPUTER-AIDED DETECTION (COMPUTER ALGORITHM ANALYSIS OF DIGITAL |
|---------------------------------------------------------------------|
| IMAGE DATA FOR LESION DETECTION) WITH FURTHER PHYSICIAN REVIEW FOR |
| INTERPRETATION, WITH OR WITHOUT DIGITIZATION OF FILM RADIOGRAPHIC |
| IMAGES; SCREENING MAMMOGRAPHY (LIST SEPARATELY IN ADDITION TO |
| CODE FOR PRIMARY PROCEDURE) / COMPUTER-AIDED DETECTION (COMPUTER |
| ALGORITHM ANALYSIS OF DIGITAL IMAGE DATA FOR LESION DETECTION) WITH |
| FURTHER REVIEW FOR INTERPRETATION, WITH OR WITHOUT DIGITIZATION OF |
| FILM RADIOGRAPHIC IMAGES; SCREENING MAMMOGRAPHY (LIST SEPARATELY |


G0144 - SCREENING CYTOPATHOLOGY, CERVICAL OR VAGINAL (ANY REPORTING SYSTEM), COLLECTED IN PRESERVATIVE FLUID, AUTOMATED THIN LAYER PREPARATION, WITH SCREENING BY AUTOMATED SYSTEM, UNDER PHYSICIAN SUPERVISION

PSA test 84152 PX CPT/HCPCS PROSTATE SPECIFIC ANTIGEN (PSA); COMPLEXED (DIRECT MEASUREMENT)


G0145 - SCREENING CYTOPATHOLOGY, CERVICAL OR VAGINAL (ANY REPORTING SYSTEM), COLLECTED IN PRESERVATIVE FLUID, AUTOMATED THIN LAYER PREPARATION, WITH SCREENING BY AUTOMATED SYSTEM AND MANUAL RESCREENING UNDER PHYSICIAN SUPERVISION

P3000 - SCREENING PAPANICOLAOU SMEAR, CERVICAL OR VAGINAL, UP TO THREE SMEARS, BY TECHNICIAN UNDER PHYSICIAN SUPERVISION

P3001 - SCREENING PAPANICOLAOU SMEAR, CERVICAL OR VAGINAL, UP TO THREE SMEARS, REQUIRING INTERPRETATION BY PHYSICIAN

Q0091 - SCREENING PAPANICOLAOU SMEAR; OBTAINING, PREPARING AND CONVEYANCE OF CERVICAL OR VAGINAL SMEAR TO LABORATORY


Telemedicine

99215

PX

CPT/HCPCS

OF TOTAL TIME IS SPENT ON THE DATE OF THE ENCOUNTER.

G8

